Emulation of effects of injectable semaglutide on cardiovascular outcomes in individuals with type 2 diabetes: SUSTAIN6 trial

NCT06659744

23<sup>rd</sup> April 2025

# 1. Title Page

| Title | Emulation of effects of injectable semaglutide on cardiovascular outcomes in individuals with type 2 diabetes: SUSTAIN6 trial (NCT01720446) |
|---|---|
| Research question & Objectives | The SUSTAIN6 trial aims to evaluate the cardiovascular safety of Injectable Semaglutide |
| | versus placebo in individuals with type 2 diabetes. |
| Protocol version | Version 4 |
| Last update date | 23st April 2025 |
| Contributors | Primary investigator contact information: |
| | Dr. Shirley Wang |
| | Swang1@bwh.harvard.edu |
| | Contributor names: |
| | Shirley Wang, Sushama Kattinakere Sreedhara, Elyse DiCesare |
| | Sushama implemented the study design in the Aetion Evidence Platform. S/he is not |
| | responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: <text></text> |
| | Identifier: <text></text> |
| Sponsor | Organization: Food and Drug Administration |
| | Contact: Dianne Paraoan |
| | dianne.paraoan@fda.hhs.gov |
| Conflict of interest | Dr. Wang has consulted for Veracity Healthcare Analytics, Exponent Inc, and MITRE and FFRDC for Centers for Medicare and Medicaid for unrelated work. |

# Table of contents

| 1. Ti | itle Page | 1 |
|---|---|---|
| 2. A | Nbstract | 3 |
| 3. A | Amendments and updates | 3 |
| 4. R | Rationale and background | 5 |
| | Research question and objectives | |
| | Table 1 Primary and secondary research questions and objective | |
| 6. R | Research methods | |
| | 6.1. Study design | |
| | 6.2. Study design diagram | |
| | 6.3. Setting | |
| | 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | |
| | 6.3.2 Context and rationale for study inclusion criteria: | |
| | 6.3.3 Context and rationale for study exclusion criteria | |
| | 6.4. Variables | |
| | 6.4.1 Context and rationale for exposure(s) of interest | |
| | 6.4.2 Context and rationale for outcome(s) of interest | |
| | 6.4.3 Context and rationale for follow up | |
| | Table 2. Operational Definitions of Follow Up | |
| | 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) | |
| | Table 3. Operational Definitions of Covariates | |
| | 6.5. Data analysis | |
| | Table 4. Primary, secondary, and subgroup analysis specification | |
| | Table 5. Sensitivity analyses – rationale, strengths and limitations | |
| | 6.6. Data sources | |
| | 7.6.1 Context and rationale for data sources | |
| | Table 6. Metadata about data sources and software | |
| | 6.7. Data management | |
| | 6.8. Quality control | |
| | 6.9. Study size and feasibility | |
| 7. Li | imitation of the methods | 32 |
| | Protection of human subjects | |
| | References | |
| | Appendices | |
| | 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | |
| | 2 Code algorithms | |
| | 3 Flowchart for cohort assembly | |
| | 4 1st feasibility assessment | |
| | 5 2nd feasibility assessment | |
| | 6 Balance Assessment - PS Distribution and C-Statistic | 34 |
| | 7 Balance Assessment - Table 1 | 34 |

#### 2. Abstract

This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as possible in healthcare insurance claims data, the SUSTAIN6 trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be emulated in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SUSTAIN6 trial, is a non-inferiority trial to evaluate the effects of injectable semaglutide versus placebo in terms of cardiovascular safety (CV death, nonfatal MI, or nonfatal stroke) in patients with type 2 diabetes.

The database study designed to emulate SUSTAIN6 trial will be a new-user active comparative study, where we compare the effect of injectable semaglutide versus sitagliptin on MACE outcome among patients with T2DM. Sitagliptin was selected to act as an active-comparator proxy for placebo. Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being of similar cost.

The study will use three data sources: Optum Clinformatics, Merative Marketscan, and Medicare.

Optum: Study period between 5th Dec 2017 – 29th February 2024 Marketscan: Study period between 5th Dec 2017 - 31st Dec 2022 Medicare: Study period between 5th Dec 2017 – 31st Dec 2020

# 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 19 <sup>th</sup> Aug 2024 | 2 | 6.4, 6.5, Table 2-4,<br>appendices 5-8 | Inclusion Exclusion Criteria: Adding TIRZEPATIDE to the list of other GLP1, Stroke definition to include only Ischemic stroke Outcome: Stroke definition to include only Ischemic stroke | Better algorithms for exclusion criteria and outcome |

| | | | Added covariates for PS adjustment | To operationally define covariates and adjust for confounding |
|---|---|---|---|---|
| | | | Power and feasibility (balance checks) post PS matching added in appendices 5, 6 and table 1 | Pre-planned data check |
| | | | Changed primary analysis from PS fine-stratification weights to 1:1 PS matching | Power calculation indicates that there will be sufficient power with 1:1 matching |
| | | | Added planned sensitivity analyses | To pre-specify sensitivity analyses |
| 16 <sup>th</sup> December<br>2024 | 2.1 | Appendices | Added the FDA protocol review dates for first and second feasibility | The protocol review dates by the FDA were not documented in the previous version. |
| 10 <sup>th</sup> March<br>2025 | 3 | Appendices | Covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were corrected. | Errors in the implementation of covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were identified. |
| 17 <sup>th</sup> April 2025 | 5 | Negative control outcomes | Added Hernia and Lumbar radiculopathy | Given the ongoing discussion around semaglutide and its potential association with non-arteritic anterior ischemic optic neuropathy (NAION) as a negative control outcome, we wanted to include alternative negative control outcomes. |

# 4. Rationale and background

The purpose of this protocol is to describe the emulation of the SUSTAIN6 trial (NCT01720446). Market availability of Injectable Semaglutide began on 5th December 2017.¹ The trial enrolled 3,297 participants between February and December 2013. The trial design is event-driven to collect 122 events, which assumes an annual 1.98% event rate in both arms over 2.1 years, which would result in 90% power, to reject a 1.8 hazard ratio at a significance level of 0.05 to assess non-inferiority.²,³

# 5. Research question and objectives

#### Table 1 Primary and secondary research questions and objective

### A. Primary research question and objective

| Objective: | To evaluate the effect of injectable semaglutide versus sitagliptin on MACE outcomes (CV death, nonfatal MI, or nonfatal stroke) in patients with diabetes and established or subclinical CV disease. |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will be superior to sitagliptin at preventing MACE |
| Population (mention key inclusion-exclusion criteria): | The study population included patients with Type 2 Diabetes (Type2DM) who had not been treated with antihyperglycemic agents or had been treated with no more than two oral antihyperglycemic agents, with or without NPH or long-acting insulin, >=50 years with established cardiovascular disease OR >=60 years with subclinical cardiovascular disease. Patients were excluded if they had type1/gestational diabetes, prior use of GLP1 or pramlintide or DPP4-inhibitors or insulin other than basal or pre-mixed insulin, acute decompensation of glycemic control, history of pancreatitis, recent acute coronary or cerebrovascular events, class IV chronic heart failure, personal or family history of multiple endocrine neoplasia or medullary thyroid carcinoma, end stage liver disease, prior organ transplant, cancer, pregnancy, substance abuse, proliferative retinopathy/maculopathy requiring acute treatment. |
| Exposure: | Injectable Semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Major adverse cardiac event (MACE), including myocardial infarction, stroke, and all cause death |
| Time (when follow up begins and ends): | One day after cohort entry date until the first of outcome, disenrollment, end of study period, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the |

| | arms, start of any other GLP1 agonists (including oral Semaglutide), Other DPP4 or Pramlintide, Nursing home admission |
|---|---|
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from inpatient hospitalizations and/or death. |
| Main measure of effect: | Hazard ratio |

# B. Secondary research question 1 and objective

| Objective: | To evaluate the effect of injectable semaglutide versus sitagliptin on negative control outcomes, including A. cataract surgery, B. hernia and C. lumbar radiculopathy |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will not have a different effect than sitagliptin |
| Population (mention key inclusion-exclusion criteria): | The study population included patients with Type 2 Diabetes (Type2DM) who had not been treated with antihyperglycemic agents or had been treated with no more than two oral antihyperglycemic agents, with or without NPH or long-acting insulin, >=50 years with established cardiovascular disease OR >=60 years with subclinical cardiovascular disease. Patients were excluded if they had type1/gestational diabetes, prior use of GLP1 or pramlintide or DPP4-inhibitors or insulin other than basal or pre-mixed insulin, acute decompensation of glycemic control, history of pancreatitis, recent acute coronary or cerebrovascular events, class IV chronic heart failure, personal or family history of multiple endocrine neoplasia or medullary thyroid carcinoma, end stage liver disease, prior organ transplant, cancer, pregnancy, substance abuse, proliferative retinopathy/maculopathy requiring acute treatment. In addition, patients were excluded for baseline hernia or lumbar radiculopathy when the negative outcome was hernia or lumbar radiculopathy respectively. |
| Exposure: | Injectable semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Separate analyses were run for cataract surgery, hernia, and lumbar radiculopathy |
| Time (when follow up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, death, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide) |

| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from outpatient procedure codes. |
|---|---|
| Main measure of effect: | Hazard ratio |

#### 6. Research methods

# 6.1. Study design

Research design (e.g. cohort, case-control, etc.): New user active comparator cohort study

Rationale for study design choice: A new user active comparator cohort study is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group.<sup>4,5</sup> While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score (PS).

#### 6.2. Study design diagram



#### 6.3. Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to treatment Injectable Semaglutide versus Sitagliptin in the clinical trial design. See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

#### 6.3.2 Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.4. Variables

#### 6.4.1 Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, Injectable Semaglutide versus Sitagliptin. See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

### Algorithm to define duration of exposure effect:

Assuming the effect of pill lasts for 30 days after the days' supply, we allow 30 days gap between the dispensation (grace period) and also add 30 days at the end of days' supply of dispensation (exposure risk window).

### 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined to emulate the primary outcome for the trial of MACE. In the trial, this was a combination of myocardial infarction, stroke, and cardiovascular death. In our emulation, due to inability to capture cause of death, our modified MACE outcome was measured as inpatient myocardial infarction, inpatient stroke, and all-cause mortality. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead status up until 2016. Medicare includes information from the inpatient discharged dead status, NDI cause of death, and social security death master file. The positive predictive value for the myocardial infarction outcome algorithm using ICD-9 codes was observed to be 88.4% and 94% in validation studies.<sup>6,7</sup> The PPV for the ischemic stroke outcome algorithm was 88% and 95% in validation studies using ICD9

codes.<sup>6,8</sup> The ICD9 code algorithms were mapped to ICD10 codes and reviewed by a clinician, but the performance of the mapped codes was not further validated.

Secondary outcomes from the trial that will be evaluated include:

- 1. Myocardial infarction
- 2. Stroke
- 3. All cause Death

Control outcomes of interest include:

- 1. Cataract surgery. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 2. Hernia. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 3. Lumbar radiculopathy. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.

#### 6.4.3 Context and rationale for follow up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants.

Table 2. Operational Definitions of Follow Up

| Follow up start | Day 1 | |
|---|---|---|
| Follow up end <sup>1</sup> | Select all that apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | Part of the outcome |
| End of observation in data | Yes | Date of disenrollment |
| Day X following index date<br>(specify day) | Yes | Day 365 |
| End of study period (specify date) | Yes | Dates for different databases (Optum: 29th Feb 2024, Marketscan Dec 31st 2022, Medicare Dec 31st 2020) |
| End of exposure (specify operational details, | Yes | 30 days grace window and 30 days risk window |

| e.g. stockpiling algorithm, grace period) | | |
|---|---|---|
| Date of add to/switch from exposure (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Censor upon starting any other GLP1 agonists, including Oral Semaglutide, Other DPP4 inhibitors or Pramlintide, Nursing home admission |

<sup>&</sup>lt;sup>1</sup> Follow up ends at the first occurrence of any of the selected criteria that end follow up.

## 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders do to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

Table 3. Operational Definitions of Covariates

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment<br>window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Age | Cohort entry year - year of birth, (last observed value in the baseline) | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | n/a |
| Gender | Male, Female<br>(last observed<br>value in the<br>baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | n/a |
| Region | Northeast, Midwest/North central, South, West (last observed value in the baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Year of Cohort<br>Entry | 2019 (Sept-Dec),<br>2020 (Jan-March),<br>2020 (April-June),<br>2020 (July-Sept),<br>2020 (Oct-Dec), | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |


| Characteristic | Conceptual definitions | Type of<br>variable | Assessment window | Care<br>Settings¹ | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| SU-2nd gen | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Metformin | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Thiazolidinedione<br>s | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| SGLT-2i | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Alpha-<br>glucosidase<br>inhibitors | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| ACEs/ARBs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Thiazides | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Beta-blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Calcium channel<br>blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Loop diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Other diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Nitrates | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hear failure<br>medications<br>(Digoxin +<br>Entresto +<br>Ivabradine) | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-arrhythmics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| COPD/asthma medications | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Statins | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of<br>variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Other lipid-<br>lowering drugs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Antiplatelet agents | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral<br>anticoagulants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| NSAIDs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral<br>corticosteroids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Bisphosphonates | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Opioids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-depressants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure:<br>Injectable<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual<br>definitions | Type of variable | Assessment window | Care<br>Settings¹ | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Gabapentinoids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Benzodiazepines | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anxiolytics/hypno tics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Medications for dementia | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Combined comorbidity score | Comorbidity score ranging from -2 to 26 | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | | Gagne, Joshua J<br>et al. <sup>9,10</sup> |
| Frailty score | | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | | Kim et al. <sup>11</sup> |
| Unique generic<br>medicines | | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Unique brand medicines | | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure:<br>Injectable<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings¹ | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Hospitalizations<br>[-90, 0] | | Binary | [-90, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hospitalizations<br>[-180, 0] | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| ED visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Office visits | | Continuous | [-180, 0] | OP | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Endocrinologist<br>visit | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Cardiologist visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Internal<br>medicine/family<br>medicine visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Electrocardiogra<br>ms | | Binary | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Echocardiograms | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| HbA1c tests received | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Glucose tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Lipid tests<br>ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Creatinine tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Bone mineral density test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Basic or<br>comprehensive<br>metabolic blood<br>chem test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Mammogram | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual definitions | Type of variable | Assessment window | Care<br>Settings¹ | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Pap smear | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| PSA | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flu vaccine/<br>Pneumococcal<br>vaccine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Telemedicine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Injectable Semaglutide Reference: Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

 $<sup>^{1}</sup>$ IP = inpatient, OP = outpatient, ED = emergency department, OT = other,  $^{n}$ /a = not applicable

# 6.5. Data analysis

#### 6.5.1 Context and rationale for analysis plan

The study will use a propensity score (PS) 1:1 nearest neighbor matching with a caliper of 0.01 on the propensity score scale. The PS will be estimated as the probability of initiating injectable semaglutide versus sitagliptin given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate distributional covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for injectable semaglutide versus Sitagliptin inhibitor on MACE outcome in the matched population using a Cox proportional hazards model.

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup> Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

# Table 4. Primary, secondary, and subgroup analysis specification

# A. Primary analysis

| Hypothesis: | Injectable Semaglutide might decrease risk of MACE outcome compared to Sitagliptin in those with diabetes and |
|---|---|
| | established or subclinical CV disease |
| Exposure contrast: | Injectable Semaglutide vs Sitagliptin |
| Outcome: | MACE |
| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| O and a series of a discrete and an other de- | |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

# B. Secondary Analysis 1

| Hypothesis: | Injectable semaglutide has no effect on risk of negative control outcomes compared to sitagliptin. Negative control outcomes include: A. cataract surgery, B. hernia, C. lumbar radiculopathy |
|---|---|
| Exposure contrast: | Injectable semaglutide vs sitagliptin |
| Outcome: | Separate analyses were run for each negative control outcome, including cataract surgery, hernia and lumbar |
| | radiculopathy |
| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |

| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
|---|---|
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

Table 5. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Re-weighted population distribution | We will re-weight the population distribution of the pooled database study cohorts to reflect that of the RCT if that information is made public prior to publication of our results. | We will learn about potential effect modification due to different distributions of key characteristics such as age/sex in the RCT versus the database study. | The population distributions will be more aligned. | The measurement of these population characteristics may be measured differently in the RCT vs database study, with different levels of specificity and sensitivity. |
| Negative control<br>outcomes, including<br>cataract surgery,<br>hernia, lumbar<br>radiculopathy | We evaluate negative control outcomes of cataract surgery, hernia, and lumbar radiculopathy, where no causal effect is expected from semaglutide or sitagliptin | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of<br>the interpretation of the primary<br>analysis by evaluating the<br>potential magnitude of<br>unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| PS-adjustment<br>method | Instead of 1:1 PS matching, we will use PS fine stratification weights. The analytic cohort will be asymmetrically trimmed at 1% of the tails. The analytic cohort will be weighted to estimate the average effect in the treated (ATT). Each exposed patient will be assigned a weight = 1. | Use of fine-stratification<br>weights will have more power<br>than 1:1 matching | More power to estimate ATT | More complex to understand than simple 1:1 match, potentially less closely balanced |

Each comparator patient will be assigned a weight =  $\frac{\binom{Nexposed\ in\ strata\ i}{Ntotal\ exposed}}{\binom{Nunexposed\ in\ strata\ i}{Ntotal\ unexposed}}$ 

#### 6.6. Data sources

#### 7.6.1 Context and rationale for data sources

**Reason for selection:** The study will be conducted in 3 US health care claims databases: Optum Clinformatics (2017-Feb 2024), Merative Marketscan (2017-2022) and Medicare (a sample that includes all patients with diabetes or heart failure diagnosis, 2017-2020)

Strengths of data source(s): Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups. The death data is captured in the Medicare database from inpatient discharge status, and social security death master file. 12-14

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. Patients in Medicare may move in and out of fee-for-service plans. We are excluding person-time in health maintenance organization (HMO) plans due to concerns about the completeness of capture of diagnoses and procedures. This means that we require patients to be enrolled in Medicare parts AB and D during the baseline assessment window and censor patients if they switch to part C. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all cause death in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal.<sup>14</sup>

**Data source provenance/curation:** Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients. Information about Medicare data provenance and curation can be found on the ResDac website.<sup>15</sup>

#### Table 6. Metadata about data sources and software

| Data 1 | Data 2 | Data 3 |
|--------|--------|--------|

| Data Source(s): | Optum Clinformatics | Merative Marketscan | Medicare |
|---|---|---|---|
| Study Period: | 5 <sup>th</sup> Dec 2017-29 <sup>th</sup> Feb 2024 | 5 <sup>th</sup> Dec 2017-31 <sup>st</sup> Dec 2022 | 5 <sup>th</sup> Dec 2017-31 <sup>st</sup> Dec 2020 |
| Eligible Cohort Entry Period: | 5 <sup>th</sup> Dec 2017-29 <sup>th</sup> Feb 2024 | 5 <sup>th</sup> Dec 2017-31 <sup>st</sup> Dec 2022 | 5 <sup>th</sup> Dec 2017-31 <sup>st</sup> Dec 2020 |
| Data Version (or date of last update): | April 2024 | Mortality Cut Set A<br>Received 2024-03-01 | DUA 59286_Received 2023-<br>10-17 |
| Data sampling/extraction criteria: | n/a | n/a | Patients with a diabetes or heart failure diagnosis |
| Type(s) of data: | Administrative healthcare claims | Administrative healthcare claims | Administrative healthcare claims |
| Data linkage: | n/a | n/a | Linkage to National Death<br>Index |
| Conversion to CDM*: | n/a | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) |

<sup>\*</sup>CDM = Common Data Model

#### 6.7. Data management

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

<u>Archiving</u>: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This

event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

Backups: Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots.\_AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances. This backup approach allows elimination of EC2 instances when access to CMS data files is no longer needed. Use of temporary instances will allow highest security control to be applied regarding for whom and when CMS data files are accessible.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

#### 6.8. Quality control

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by both MGB and FDA team members. Team members will review code lists to ensure fidelity to intended algorithms.

# 6.9. Study size and feasibility

First feasibility assessment: Details of power calculations after applying eligibility criteria and matching on ages, sex and comorbidity score are available in appendix 4.

Second feasibility assessment: Details of power calculations after matching or weighting on all predefined propensity score variables are available in appendix 5..

Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7.

# 7. Limitation of the methods

As we are using secondary data and the data were not collected for research, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce

confounding by unmeasured factors. One measurement difference is for the primary outcome, where for the RCT, MACE was defined as stroke, myocardial infarction, and cardiovascular death, whereas in our database study, it is defined as stroke, myocardial infarction, and all cause death.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid which is not guaranteed.

Although we plan to emulate the important features of each RCT as closely as possible in healthcare claims, there may be some elements of RCT design that are not emulable with a database study, which means that the study generating RWE and the RCT will address slightly different clinical questions. For example, in routine clinical practice, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

# 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

#### 9. References

- 1. Novo Nordisk Receives FDA Approval of OZEMPIC® (semaglutide) Injection For the Treatment of Adults with Type 2 Diabetes. <a href="https://www.prnewswire.com/news-releases/novo-nordisk-receives-fda-approval-of-ozempic-semaglutide-injection-for-the-treatment-of-adults-with-type-2-diabetes-300567052.html#:~:text=OZEMPIC%C2%AE%20(semaglutide)%20injection%200.5%20mg%20or%201%20mg%20was,adults%20with%20type%202%20diabetes. PR Newswire.
- 2. ClinicalTrials.gov. Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes (SUSTAIN™ 6). National Institutes of Health. Accessed April 30, 2024. <a href="https://www.clinicaltrials.gov/study/NCT01720446">https://www.clinicaltrials.gov/study/NCT01720446</a>
- 3. Marso SP, Bain SC, Consoli A, et al. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. *N Engl J Med*. Nov 10 2016;375(19):1834-1844. doi:10.1056/NEJMoa1607141
- 4. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* Aug 2010;19(8):858-68. doi:10.1002/pds.1926
- 5. Ray WA. Evaluating medication effects outside of clinical trials: new-user designs. Am J Epidemiol. Nov 1 2003;158(9):915-20. doi:10.1093/aje/kwg231
- 6. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiology and drug safety*. Jun 2010;19(6):596-603. doi:10.1002/pds.1924
- 7. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J.* Jul 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 8. Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. *Stroke; a journal of cerebral circulation*. Oct 2002;33(10):2465-70. doi:10.1161/01.str.0000032240.28636.bd
- 9. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. Jul 2011;64(7):749-59. doi:10.1016/j.jclinepi.2010.10.004
- 10. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. Dec 2017;55(12):1046-1051. doi:10.1097/mlr.0000000000000824

- 11. Kim D, Schneeweiss S, Glynn R, Lipsitz L, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *Journals of Gerontology: Medical Sciences*. 2017;73:980-987. doi:10.1093/gerona/glx229
- 12. Jarosek S. Death Information in the Research Identifiable Medicare Data. Accessed June 17, 2024. <a href="https://resdac.org/articles/death-information-research-identifiable-medicare-data">https://resdac.org/articles/death-information-research-identifiable-medicare-data</a>
- 13. Hill ME, Rosenwaike I. The Social Security Administration's Death Master File: The Completeness of Death Reporting at Older Ages. *Social Security Bulletin*. 2002;64(1):45-51.
- 14. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *Journal of the American Heart Association*. May 3 2017;6(5)doi:10.1161/jaha.116.004966
- 15. Research Data Assistance Center (ResDAC). <a href="https://resdac.org/">https://resdac.org/</a>. Centers for Medicare & Medicaid Services (CMS).

# 10. Appendices

See accompanying excel file.

- 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1

## **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate algorithm sources
| | SUSTAIN 6 trial definitions | (Optum) | (Medicare) | (MarketScan) | Notes/Questions | Color coding |
|---|---|---|---|---|---|---|
| reatment assignment (tim<br>0, index date | | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-<br>exclusion criteria) | Non-randomized initiation of treatment A vs B (first eligible entry to study population) | Non-randomized initiation of treatment A vs B (first eligible entry to study population) | | |
| Ефовиг | Semaglutide (once-weekly in drug naïve subjects - monotherapy) Two experimental arms: (1.0mg and 0.5mg) | Code type:NDC, generic name Care setting:N/A Diagnosis position:N/A Weshout withow(1:80 - 1) Incident with respect to:semaglutide and sitagliptin in any dose or formulation Assessment window:N/A Source of algorithmidrug names linked to NDC Measurement characteristics//A | Code typen.NDC, generic name Care setting, NY, NA Diagnosia position:N, NA Washout window(:180, -1, 1) Incident with respect to:semaglutide and sitagliptin in any dose or formulation Assessment window:N/A Source of algorithmicing names linked to NDC Measurement characteristics:V/A | Code typex.NDC. generic name Care setting Ny. Ny. A Diagnosis position:Ny. A Washout withow(1:48). 3.1 Incident with respect to:semaglutide and sitagliptin in any dose or formulation Assessment window(Ny.A Source of algorithmidray names linked to NDC Measurement chearacteristicas(y/A | We defined Semaglutide using NDC codes for drug brand name Ozempic, route of administration injectable, with doses up to 1mg | Good proxy definition |
| Comparate | on Placebo | Code type: NDC Cane setting: NIA Diagnosis position: NIA Weshout Window: 1.80,1 Incident with respect tosemaglutide and sitagliptin in any dose or formulation Assessement window: NIA Source of algorithmicing names linked to NDC Measurement holaracteristics: | Code type: NDC Care setting: N/A Diagnoels poetton: N/A Washout windows; 1:80, -1] Incloent with respect to:semaglutide and sitagliptin in any dose or formulation Assessment windows: N/A Source of algorithmicing names linked to NDC Measurement characteristics: | Code type: NDC Care setting: N/A Diagnosis position: N/A Weshout window; 1:80, -1] Incident with respect to:semaglutide and sitagliptin in any dose or formulation Assessment window; N/A Source of algorithm:drug names linked to NDC Measurement characteristics: | We used sitagliptin as an active comparator proxy for placebo. We allowed sitagliptin alone or in combination pills with metformin only. | Moderate proxy definition |
| Primary Outcom | MACE, Defined as Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke | Lode type:DX Care setting: inpatient Diagnosis position:Primary for Stroke, Any for MI Washout window: Washout window: Measurement characteristics:PV for MI using ICD9 codes was 88.4% and 94.6%. Inline. Inlin | Code type:DX Caro setting: Inpatient Dilagnosip position:Primary for Stroke, Any for MI Washout window: Source of algorithm:ProMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94% [https://pubmed.ncbi.nlm.nih.gov/20140892/ and https://pubmed.ncbi.nlm.nih.gov/15215798/] PPV for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.nlm.nih.gov/12047393] BPV for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.nlm.nih.gov/20140892/] Bath of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | Code type:DX Care setting Inpatient Diagnosis position:Primary for Stroke, Any for MI Washout Window: Source of algorithm:PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94% [https://pubmed.ncbi.mim.in.gov/20140892/ and https://pubmed.ncbi.mim.in.gov/15215798/] PPV for Ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.mim.in.gov/20140892/] BPV for Ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.mim.in.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | Optum death includes information from the inpatient discharged dead status, social security death master file, and death caster sources. MarketScan includes information from the inpatient discharged dead status up until 2016. Medicare includes information from the inpatient discharged dead status, NDI cause of death, and social security death master file. | Poorly measured in database but not c |
| Palla | Day description days | One day after date of initiation of treatment A vs B | One day after date of initiation of treatment A vs B | One day after date of initiation of treatment A vs B | | for the analysis Poorly measured and important for the |
| rollow up sta | rl Randomization date | Earliest of: Outcome, end of data/study period, 109 weeks, | Earliest of: Outcome, end of data/study period, 109 weeks, | Earliest of: Outcome, end of data/study period, 109 weeks, | | analysis |
| Follow up en | 109) | discontinuation (30 days grace window and risk-window),<br>switch within or between GLP1 and DPP4 class or add<br>pramlintide, disenrollment, nursing home stay | discontinuation (30 days grace window and risk-window), switch<br>within or between GLP1 and DPP4 class or add pramlintide,<br>disenrollment, nursing home stay | discontinuation (30 days grace window and risk-window), switch<br>within or between GLP1 and DPP4 class or add pramlintide,<br>disenrollment, nursing home stay | | |
| Causal estimar | Modified intention-to-treat | On-treatment | On-treatment | On-treatment | | |
| Effect estimation inclusion criteri | | | | | | |
| | 1. Type 2 DM | Applied before/after selection of index datasefore Assessment window:[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicst/A | Applied before/after selection of index date/efore Assessment window:[±380, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm::PROMISE team Measurement characteristics:1//A | Applied before/after selection of Index date/efore Assessment windown(±180, 0) Code typetD, Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:IV/A | | |
| : | HbA1c above or equal to 7.0% at screening | Can't measure in claims | Can't measure in claims | Can't measure in claims | | |
| | Anti-diabetic drug naïve, or treated with one or two oral antidiabetic drug (OADs), or treated with unean Neutral Protamin Hagedorn (NPH) insulin or long-acting insulin analogue or pre-mixed insulin, both types of insulin either alone or in combination with one or two OADs | Applied before/after selection of Index dat@efore Assessment window:[-180, 0] Code type:NDC Care setting: r/o Diagnosis position:r/a Source of algorithm:PROMISE team Measurement characteristics:r/A | Applied before/after selection of index det@efore Assessment window:[-180, 0] Code type:NDC Care setting: n/a Diagnosis poetition:n/a Source of algorithm::PROMISE team Measurement characteristics:IV/A | Applied before/after selection of Index date/afore Assessment windows[:180, 0] Code type:NDC Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristios:N/A | We are implementing this by scoring each class of<br>antidiabetic medications as 1. Insulin long acting<br>and/or mixed is scored and all other oral antidiabetic<br>medications including combinations are scored as 1<br>if patients have score of more than 3 then we exclude<br>them. | |
| 4a or 4 | b | , | , | , | | |
| 4 | Age above or equal to 50 years at screening and clinical evidence of cardiovascular disease (specified below). Established CVD as one of the following: | Applied before/after selection of Index dateefore Assessment windows[0, 0] Code typen;/a Care setting: n/a Diagnosis position:n/a Source of algorithmen;/a Measurement characteristics:N/A | Applied before/after selection of index dates fore<br>Assessment window:[0, 0]<br>Code type:n/9<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:n/a<br>Measurement characteristics:N/A | Applied before/after selection of Index dataserier Assessment Windows(D, 0) Code typesn/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics:N/A | | |
| 4a. | 1 prior myocardial infarction | Applied before/after selection of index dat@efore<br>Assessment window.[-180, 0]<br>Code types.[V]<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithms:PROMISE team<br>Measurement characteristics:IV/A | Applied before/after selection of index dat@efore<br>Assessment window:[-180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics:IV/A | Applied before/after selection of index datelefore Assessment window:[-180, 0] Code byec:D/ Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:IV/A | | |
| <b>4</b> a: | 2 prior stroke or prior transient ischemic attack | Applied before/efter selection of index dateefore Assessment window:[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithms:PROMISE team Measurement characteristics:N/A | Applied before/after selection of index datelefore Assessment window:[-180, 0] Code type:[DA Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:!\/A | Applied before/after selection of Index dates/ore Assessment windows[-180, 0] Code byectD, Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement chearacteristics:N/A | | |

| <b>4e3</b> p | orior coronary, carotid or peripheral arterial revascularization | Applied before/after selection of index date/efore<br>Assessment window:[-180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team, investigator review of<br>codes<br>Measurement characteristics:N/A | Applied before/after selection of index datelefore Assessment window:[±180, 0] Code type:(1) Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team, Investigator review of codes Measurement characteristics:(N/A | Applied before/after selection of Index dat@efore Assessment window:[180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team, Investigator review of codes Measurement characteristics:N/A | |
|---|---|---|---|---|---|
| | more than 50% stenosis on anglography or imaging of coronary, carotid or lower<br>extremities arteries | Applied before/ after selection of Index datélefore Assessment window(=180,0) Code type:PX Care setting: Any Diagnosia position:Any Source of algorithm:PROMISE team Measurement characteristics:N/A | Applied before/efter selection of Index datelefore Assessment window:[-180, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:N/A | Applied before/after selection of Index datelefore Assessment windows [-180, 0] Code type:PX Cere setting: Any Diagnosia position:Any Source of algorithm:PROMISE team Measurement characteristics:N/A | Pert of this is captured in the above inclusion criteria. We also added peripheral vascular disease and coronary artery disease codes to be inclusive |
| | nistory of symptomatic coronary heart disease documented by e.g. positive exercise stress test or any cardiac imaging or unstable angina with ECG changes | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| 4a6 | asymptomatic cardiac ischemia documented by positive nuclear imaging test or<br>exercise test or stress echo or any cardiac imaging | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | chronic heart failure New York Heart Association (NYHA) class II-III | Applied before/after asketton of Index datelefore Assessment windows[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithmsPROMISE team Measurement characteristics:N/A | Applied before/after selection of Index dates fore Assessment window; [180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement oharacteristics:ti/A | Applied before/after selection of Index dat@efore Assessment windows(=180, 0) Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:N/A | We defined by using heart failure codes (patients with<br>type 4 heart failure are excluded so hopefully that wi<br>help with capturing patients with milder heart failur or<br>this class) |
| 4a8 <sup>C</sup> | per MDRD | Applied before/after selection of Index datélefore Assessment window;[-180, 0] Code type:(X) Care setting: Any Diagnosis position: Any Source of algorithms*PROMISE team Measurement characteristics:(X)A | Applied before/after selection of index dat@efore Assessment windows.[180,0] Code type:() Care setting: Any Diagnosis position:Any Source of algorithms:PROMISE team Measurement ohareotoristics:ti/A | Applied before/after selection of Index det&efore Assessment windows[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithms*PROMISE team Measurement characteristics:N/A | We defined it by CKD 3-4 |
| 4b | Aged 60 years or older with subclinical evidence of cardiovascular disease (specified below). Subclinical cardiovascular risk factors as one of the following: | Applied before/ after selection of Index datelefore Assessment windows.[0, 0] Code type:://a Care setting: //a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics:N/A | Applied before/after selection of Index datelefore Assessment window:[0, 0] Code type:://a Care setting: n/a Diagnosts postition:n/a Source of algorithm:n/a Measurement oharacteristics:N/A | Applied before/after selection of Index dat@efore Assessment window:[0, 0] Code type:n/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics:N/A | |
| | oersistent microalbuminuria (30–299 mg/g) or proteinuria | Applied before/after selection of Index datalefore Assessment Windows[-180, 0] Code type:DX Care setting Any Diagnosis position:Any Source of algorithms/PROMISE team Measurement of haracteristicsst/A | Applied before/efter selection of index dat@efore<br>Assessment window:[180,0]<br>Oode type:DX.<br>Oare setting: Apy<br>Diagnosis poetition:Any<br>Source of algorithms:PAOMISE team<br>Measurement characteristics:(VA | Applied before/after selection of Index detectore Assessment windows(=180, 0) Code type(DX Care setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement cheracterisations//A | We defined it using the diagnosis code for conditions where proteinuria is present (conditions like nephrots syndrome) or conditions defining proteinuria (exampli isolated proteinuria, bence jones proteinuria) |
| 4b2 1 | hypertension and left ventricular hypertrophy by electrocardiogram or imaging<br>eft ventricular systolic or diastolic dysfunction by imaging | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | |
| | ankle/brachial index less than 0.9 | Applied before/after selection of Index date/efore Assessment window:[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of align/thm/dirvestigator review of codes Measurement characteristics:IV/A | Applied before/after selection of index datelefore Assessment window; 180, 0] Code type:(X) Care setting: Any Diagnosis position:Any Source of algorithm:Investigator review of codes Measurement characteristics:(V) A | Applied before/after selection of Index det&efore Assessment window:[±80, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of significant selections of codes Measurement characteristics!\/A | We defined it using the diagnosis code for<br>atherosclerosis of native arteries of extremities with<br>intermittent claudication |
| | Type 1 diabetes mellitus, Secondary diabetes, Gestational diabetes | Applied before/after selection of Index datelefore<br>Assessment window:[-180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithms:PROMISE team<br>Measurement hareacteristics:V/A | Applied before/after selection of index date/efore<br>Assessment window:[-180, 0]<br>Code tyee:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithms:RADE<br>Measurement characteristics:\/A | Applied before/after selection of Index databefore Assessment window:[±80, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:SRADE Measurement characteristics!/A | Secondary diabetes, Gestational diabetes are the 2 additional criteria added |
| | Use of glucagon-like peptide-1 (GLP-1) receptor agonist (exenatide, liraglutide, or pramilintide within 90 days prior to screening | Applied before/after selection of Index det&efore Assessment window:[-120, 0] Code type:\times Code type:\times Code type:\times Code selecting: 1/8 Source of algorithmsPROMISE team Measurement of haracteristicstVA | Applied before/after selection of index datélefore Assessment window: [180, 0] Code type:\(\text{IDC}\) Care setting: \(\text{IPC}\) Diagnosis position:\(\text{IPC}\) Source of algorithm:\(\text{IPC}\) Measurement of heroctristics\(\text{IPC}\) Measurement of heroctristics\(\text{IPC}\) | Applied before/after selection of Index det&efore Assessment withdow:[180,0] Code typex/IDC Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement cheracterisdics/t/A | we are doing 180 days look back |
| | Use of any dipeptidyl peptidase 4 (DPP-IV) inhibitor within 30 days prior to<br>screening | Applied before/after selection of Index datelefore Assessment windows[-130, 0] Code type:NDC Care setting: n/a Diagnosis position:n/a Source of algorithms*PROMISE team Messurement haracteristicsty/A | Applied beforsy/after selection of Index date/afore Assessment window:[-180, 0] Code type:\NDC Care setting: r/\u00e3 Diagnosis poetition:n/a Source of algorithm:\u00e4POMISE team Measurement characteristics:\u00e4/\u00e4 | Applied before/after selection of index dat@efore Assessment windows:[=80, 0] Code type:NDC Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:V/A | we are doing 180 days look back |
| | | Applied before/after selection of Index date/efore<br>Assessment Window; 90, 0)<br>Code type:Generic<br>Care setting: n/a<br>Diagnosip position:n/a<br>Source of algorithme?#ROMISE team<br>Measurement characteristicts/A | Applied before/after selection of index datelefore<br>Assessment windows[-95, 0]<br>Code types:ceneric<br>Care setting: r/s<br>Diagnosis position:r/a<br>Source of algorithms:PROMISE team<br>Measurement characteristics:t//A | Applied before/after selection of Index dat@efore<br>Assessment window;[=0,0,0]<br>Code type:Generic<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:PROMISE team<br>Measurement characteristicasy/A | |

| Acute decompensation of glycaemic control requiring immediate intensification of <b>5</b> treatment to prevent acute complications of diabetes (eg diabetes ketoacidosis) within 90 days prior to screening | Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:N/A | Applied before/after selection of index dat@efore Assessment window:[-90, 0] Code type:DX Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:t//A | Applied before/after selection of index datelefore Assessment window:[=0,0] Code type:DX Core setting: r/a Diagnosis position:n/a Source of algorithmizmoMisE team Measurement characteristics:V/A | We defined it by diagnosis of diabetes ketoacdiosis (DKA) OR Hyper osmolar hypergreemic non-ketotic syndrome (HONK) |
|---|---|---|---|---|
| 6 History of chronic pancreatitis or idiopathic acute pancreatitis | Applied before/after selection of Index dat@efore Assessment window:[180, 0] Code type:DX Care setting: n/s Diagnosis position:n/s Source of algorithms/ROMISE team Measurement characteristics:t/A | Applied before/after selection of Index dataserore Assessment window(=180, 0) Code type:DX Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:t/A | Applied before/after selection of Index datasefore Assessment Mindows[-180, 0] Code type:DX Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:V/A | |
| 7 Acute coronary or cerebro-vascular event within 90 days prior to randomisation | Applied before/after selection of index dat@efore Assessment window:[90, 0] Code type:DX Care setting: Inpatient Disgnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:V/A | Applied before/after selection of index dat@efore Assessment window; [90, 0] Code type: DX Care setting in patient Disgnosts position: Any Source of algorithm:PROMISE team Measurement characteristics: V/A | Applied before/after selection of Index date@fore Assessment windox(=0,0,0) Code type:DX Care setting Inpatient Diagnosis position:Arry Source of algorithm:PROMISE team Measurement characteristics:V/A | We defined this using diagnosis codes for acute MI, tia, unstable angina, stable angina in inpatient setting |
| 9 Chronic heart failure New York Heart Association (NYHA) class IV | Can't measure in claims Applied before After selection of Index dat@efore Assessment Windows[-180, 0] Code type:DX, PX Care setting: IP, Any Diagnosis position:Any Source of algorithms/PROMISE team Measurement characteristicst//A | Can't measure in claims Applied before/after selection of Index dat@efore Assessment windows:[180, 0] Code type:DX, PX Care setting: IP, Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:1/A | Can't measure in claims Applied before after selection of Index datelefore Assessment windows:[180, 0] Code type:DX, PX Care setting: IP, Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:(/A | We defined this as heat failure codes in inpatient setting with oxygen use code on the same day |
| 10 Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma | Applied before/after selection of index detelefore Assessment windowr. 180. 0 Code type:DX Core setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicst//A | Applied before/after selection of index detelerore Assessment window(-180, 0) Code type:DX Core setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicst//A | Applied before/after selection of Index databefore Assessment window(-1.150, 0) Code type:(3) Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:(/A | |
| 11. Personal history of non-familial medullary thyroid carcinoma | Applied before/after selection of index dat@efore Assessment Windows [-180, 0] Code types DA Care setting: Any Diagnosis position:Any Source of algorithmichyestigator review of codes Measurement characteristics:t/A | Applied before/after selection of index dat@efore Assessment windows [-180, 0] Code type:DA Care setting: Any Diagnosis position:Any Source of algorithminvestigator review of codes Measurement characteristics:V/A | Applied before/after selection of index dat@efore Assessment windows [-180, 0] Code types DA Care setting: Any Diagnosis position:Any Source of algorithms/investigator review of codes Measurement characteristics:V/A | Assessment window may not capture cancer in distant past |
| 13 Chronic hemodialysis or chronic peritoneal dialysis | Can't measure in claims Applied before/after selection of Index det@efore Assessment windows[-60, 0] Code type:DX, PX Core setting: Inpatient Diagnosis position:Any Source of algorithms:PROMISE team Measurement characteristics:V/A | Can't measure in claims Applied before/after selection of index datasefore Assessment windows[-80, 0] Code type:DX, PX Core setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:t/A | Can't measure in claims Applied before/after selection of index datasefore Assessment windows[-80, 0] Code typecIX, PX Core setting in pagient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:(/A | We defined using CKD5/ESRD/Dialysis/Renal transplant code |
| | Applied before/after selection of Index date: Before<br>Assessment window:[-180, 0] | Applied before/after selection of Index date: Before<br>Assessment window:[-180, 0] | Applied before/after selection of Index date: Before<br>Assessment window:[-180, 0] | |
| | Code type:DX, PX, RX Care setting, 4ny Diagnosis position:Any Source of algorithm Inters/pubmed-ncb:nlm.nih.gov/22674685/ and Intrps//pubmed.ncb:nlm.nih.gov/34256144/ Measurement characteristics// | Code type DV, PX, RX Care setting: Any Diagnosis position: Any Source of algorithm: https://pubmed.ncb.inlm.nih.gov/22674685/ and https://pubmed.ncb.inlm.nih.gov/34256144/ Measurement characteristics/// | Assessment without per (1-50, t) Gode (spect), PX, RX Care setting: Any Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristics//A | According to<br>https://pubmed.ncbl.nlm.nih.gov/22674685/, ESLD in<br>claims can be defined using Orrohosis +<br>Decompensation event.<br>We used the LOS9/COI codes from the above study<br>and https://pubmed.ncbl.nlm.nih.gov/34256144/, to<br>define the codes required for Orrhosis and<br>Decompensation events |
| End-stage liver disease, defined as the presence of acute or chronic liver disease that and recent history of one or more of the following: ascites, encephalopathy, variceal bleeding, billrukin ≥ 2.0 mg/d, albumin level ≤ 3.5 g/d, protrombin time ≥4 seconds prolonged, international normalized ratio ≥1.7 or prior liver transplant of the properties of th | Code type:DX, PX, RX Care setting. Any Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674695/ and https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristicst//A Applied before/after selection of Index dat@efore Assessment windowe(-180, 0) Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicsti/A | Code type:DX, PX, RX Care setting. Any Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nim.nih.gov/22674685/ and https://pubmed.ncbi.nim.nih.gov/34256144/ Measurement characteristicst//A Applied before/after selection of Index dat@efore Assessment windows[-180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicsti//A | Code type:DX. PX. RX Care setting: Armany Diagnosis position: Any Source of algorithm: https://pubmed.ncbi.nim.nih.gov/34256144/ Measurement characteristics://A Applied before/after selection of Index datesfore Assessment windows:[180, 0] Code type:DX. PX Care setting: Inpatient Diagnosis position: Any Source of algorithm:PROMISE team Measurement characteristics:V/A | https://pubmed.ncbi.nlm.nih.gov/22674685/, ESLD in claims can be defined using Cirrohosis + Decompensation event. We used the ICD9/ICD10 codes from the above study and https://pubmed.ncbi.nlm.nih.gov/34256144/, to define the codes required for Cirrhosis and |
| End-stage liver disease, defined as the presence of acute or chronic liver disease and cecent history of one or more of the following: ascites, encephalopate, varience bleeding, billuriah = 2.0 mg/d, albumin level < 3.5 g/d, protrombin time ≥4 seconds prolonged, international normalized ratio ≥1.7 or prior liver transplant 15 A prior solid organ transplant or awaiting solid organ transplant 16 Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer) | Code type:DX, PX, RX Care setting: Ay Diagnosis position:Any Source of aligorithm: https://pubmed.ncbi.nlm.nin.gov/22674685/ and https://pubmed.ncbi.nlm.nin.gov/24256144/ Measurement characteristics:V/A Applied before/after selection of index deteefore Assessment window:[-180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of aligorithm:PRPOMISE team | Code type:DX, PX, RX Care setting:Ay Diagnosis position:Ayy Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/24256144/ Measurement characteristics:V/A Applied beforey after selection of index detectore Assessment window:[-180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Ayy Source of algorithm:PROMISE team | Code type:DX, PX, RX Care setting: Ay Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nlm.nin.gov/22674685/ and https://pubmed.ncbi.nlm.nin.gov/34256144/ Measurement characteristics:4/A Applied beforey after aslocition of Index datasefore Assessment windows(-180, 0) Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team | https://pubmed.ncbi.nlm.nih.gov/22674685/, ESI.D in claims can be defined using (fronteind using dirondein dusing dirondein dusing dirondein designed in the above study and https://pubmed.ncbi.nlm.nih.gov/34256144/, to define the codes required for Crirhosis and Decompensation events Assessment window may not capture transplant in |
| End-stage liver disease, defined as the presence of acute or chronic liver disease and cecent history of one or more of the following: ascites, encephalopate, varience bleeding, billuriah = 2.0 mg/d, albumin level < 3.5 g/d, protrombin time ≥4 seconds prolonged, international normalized ratio ≥1.7 or prior liver transplant 15 A prior solid organ transplant or awaiting solid organ transplant 16 Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer) | Code type:DX, PX, RX Care setting:Ay Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nlm.nin.gov/22674685/ and https://pubmed.ncbi.nlm.nin.gov/34256144/ Measurement characteristics/t/A Applied before/after selection of index dataefore Assessment window:[-180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PRONISE team Measurement characteristics/t/A Applied before/after selection of index dataefore Assessment window:[-1825, 0] Code type:DX Care setting:Any Diagnosis position:Any Source of algorithm:PRONISE team Measurement window:[-1825, 0] Code type:DX Care setting:Any Diagnosis position:Any Source of algorithm:PRONISE team | Code type:DX, PX, RX Care setting:Ay Diagnosis position:Ayy Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/24256144/ Measurement charactaristics/ti/A Applied before/after selection of index datesfore Assessment window:[-180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PRONISE team Measurement charactaristics/ti/A Applied before/after selection of index datesfore Assessment window:[-1825, 0] Code type:DX Care setting:Any Diagnosis position:Any Diagnosis position:Any Source of algorithm:PRONISE team | Code type:DX. PX. RX Care setting: Apy Diagnosis position: Any Diagnosis position: Any Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristicst//A Applied before/after selection of Index datasefore Assessment windows:[180, 0] Code type:DX. PX Care setting: Inpatient Diagnosis position: Any Source of algorithm:PRONISE team Measurement characteristicst//A Applied before/after selection of Index datasefore Assessment windows:[1825, 0] Code type:DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm:PRONISE team | https://pubmed.ncbi.nlm.nih.gov/22674685/, ESI.D in claims can be defined using (fronteind using dirondein dusing dirondein dusing dirondein designed in the above study and https://pubmed.ncbi.nlm.nih.gov/34256144/, to define the codes required for Crirhosis and Decompensation events Assessment window may not capture transplant in |
| End-stage liver disease, defined as the presence of acute or chronic liver disease and and recent history of one or more of the following: ascites, encephalopate, surfaced bleeding, billrubin 2-20, mg/d, albumin level 3-5, g/d, prothrombin time 2-4 seconds prolonged, international normalized ratio 2-1.7 or prior liver transplant. A prior solid organ transplant or awaiting solid organ transplant. Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer) Any acute condition or exacerbation of chronic condition that would in the investigator's opinion interfere with the initial trial visit schedule and procedures. Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using an adequate contraceptive method (adequate contraceptive method (adequate contraceptive method (adequate contraceptive method (adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) | Code type:DX, PX, RX Care setting: Ay Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nlm.nih.gov/22674685/ and https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristicst//A Applied before/after selection of index dat@efore Assessment window:[-180, 0] Code type:DX, PX Care setting: inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristicst//A Applied before/after selection of index dat@efore Assessment window:[-1825, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement of are of algorithm:PROMISE team Measurement of algorithm:PROMISE team | Code type:DX, PX, RX Care setting:Ay Diagnosis position:Ayy Source of algorithm: https://pubmed.ncbi.nim.nih.gov/22674685/ and https://pubmed.ncbi.nim.nih.gov/34256144/ Measurement characteristics/1/A Applied before/after selection of Index dat@efore Assessment window:[180, 0] Code type:DX, PX Care setting: Inpatient Diagnosis position:Ayy Source of algorithm:PROMISE team Measurement characteristics/1/A Applied before/after selection of Index dat@efore Assessment window:[1825, 0] Code type:DX Care setting:Ayy Diagnosis position:Ayy Source of algorithm:PROMISE team Measurement of arrival and any of the property of t | Code type:DX. PX. RX Care setting:Arry Diagnosis position:Any Source of algorithm: https://pubmed.ncbi.nim.nih.gov/34256144/ Measurement characteristics:V/A Applied before/after selection of Index datesfore Assessment window:[-180, 0] Code type:DX. PX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement window:[-180, 0] Code type:DX. Applied before/after selection of Index datesfore Assessment window:[-180, 0] Code type:DX Care setting:Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement window:[-1825, 0] Code type:DX Care setting:Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:V/A | https://pubmed.ncbi.nlm.nih.gov/22674685/, ESI.D in claims can be defined using (fronteind using dirondein dusing dirondein dusing dirondein designed in the above study and https://pubmed.ncbi.nlm.nih.gov/34256144/, to define the codes required for Crirhosis and Decompensation events Assessment window may not capture transplant in |

| 20 | Known use of non-prescribed narcotics or illicit drugs | Assessment window:[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:search of clinical code lists | Applied before/after selection of index dat@efore Assessment windows:[-180, 0] Code type::/X Care setting: Any Diagnosis position::Any Source of algorithms:search of clinical code lists Measurement characteristics:\( / X | Applied before/after selection of index dat@efore Assessment windows[-180, 0] Code types() Code types() Diagnosis position:Any Source of algorithms:search of clinical code lists Measurement characteristics()/A | We are defining it as drug dependence or abuse disorders |
|---|---|---|---|---|---|
| | Previous participation in this trial. | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| 22 | Simultaneous participation in any other clinical trial of an investigational agent. Participation in a clinical trial with investigational stent(s) is allowed | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| 23 | Receipt of any investigational medicinal product within 30 days prior to screening (Visit 1) or according to local requirements, if longer | | Can't measure in claims | Can't measure in claims | |
| 24 | Any other factor likely to limit protocol compliance or reporting of adverse event at the discretion of the investigator | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| 25 | Proliferative retinopathy/maculopathy requiring acute treatment | Assessment window:[-90, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm::LAD-2 | Applied before/after selection of Index det@efore Assessment windows[-90, 0] Code type.PX Care setting. Any Diagnosis poetton: Any Source of algorithm: LEAD-2 Measurement characteristics!\/\/A | | Additional criteria from PIONEER6, we defined it by either Anti-VEGFi injections or Photocoagulation |
| 26 | Age OR Gender Missing | Assessment window:[-180, 0] Code type:n/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a | Applied before/after selection of index detelerore Assessment windows [180, 0] Code type.n/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a Measurement obseratoristics:n/a | Applied before/after selection of index deteerore Assessment windows [-180, 0] Code type://a Core setting: //a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics://a | Additional criteria |
| 27 | Nursinghome | Assessment windowr.[-180, 0] Code typeDischarge Status Code, CPT/HCPCS Procedure Code, Provider Category Code Care setting: Any Diagnosis position: Any Source of algorithm:PROMISE team | Applied before/after selection of Index dat@efore<br>Assessment windows[180, 0]<br>Code type:Discharge Status Code, CPT/HCPCS Procedure Code,<br>Provider Category Code<br>Care setting:Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics:1/a | Applied before/after selection of Index datelerore Assessment windowr[-180, 0] Ood e type/Patient Discharge Status Code, CPT/HCPCS Procedure Code Care setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement characteristics: | Additional criteria |


| Antidiabetic medication score (sum of component 1-8, eac |
|---|
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, each |
| component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac component scored as 1) |
| Antidiabetic medication score (sum of component 1-8, eac |
| component scored as 1) |


BYPASS LEFT EXTERNAL ILIAC ARTERY TO BILATERAL FEMORAL ARTERIES WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC


| Peripheral Vascular Disease (PVD) or PVD 5047Q3D5 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALLUMINAL DEVICE, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047Q3D2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047Q3E2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047Q3E7 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047Q3F2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 5047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALLUMINAL DEVICES, PERCUTANEOUS APPROACH | |
|---|---|
| Peripheral Vascular Disease (PVD) or PVD 1047Q3E6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROPRIATE PART ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 1047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 1047Q3F2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PRIDE TO THE PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PRID TO THE PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PRID TO THE PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PRID TO THE PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PRID TO THE PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PROPROSE PROACH PART INTRALUMINAL DEVICES, PERCUTANEOUS PROACH PART INTRALUMINAL DEVI | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 104703EZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBLAL ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 104703F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBLAL ARTERY, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APP Peripheral Vascular Disease (PVD) or PVD 104703F2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBLAL ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APP | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD : 047Q3F2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | ROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 047Q3F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD : 047Q3F2 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q3FZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | |
| | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047Q3GZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROAC | |
| Peripheral Vascular Disease (PVD) or PVD \$047Q326 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, PERCUTANEOUS APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047Q3ZZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, PERCUTANEOUS APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q446 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANE | OUS ENDOSCOPIC APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q44Z PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOP | PIC APPROACH Established CVD component |
| DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERC | |
| Peripheral Vascular Disease (PVD) or PVD 50470456 PX ICD-10 APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD: 047Q452 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALLUMINAL DEVICES, PERCUTANEOUS END | |
| DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER | |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q466 PX ICD-10 APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 5 047Q46Z PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS EN | DOSCOPIC APPROACH Established CVD component |
| DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEV | ICES, PERCUTANEOUS |
| Peripheral Vascular Disease (PVD) or PVD 5047Q476 PX ICD-10 ENDOSCOPIC APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q47Z PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTAN | NEOUS ENDOSCOPIC APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD: 047Q4D6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBLAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOP | |
| Peripheral vascular insesse (PVD) or PVD 547Q4D2 PX (ICD-10 DILATION OF LET ANTERIOR TIBIAL ARTERY WITH INTRACUMINAL DEVICE, PERCUTANDUS SERVOSCOPIC PAPPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047Q4E6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS ENDI | |
| Peripheral Vascular Disease (PVD) or PVD \$047Q4EZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPRO | DACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047Q4F6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS END | DOSCOPIC APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q4FZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPR | ROACH Established CVD component |
| ., | |
| Peripheral Vascular Disease (PVD) or PVD 1047Q4G6 PX ICD-10 DILATION OF LEFT ANTERIOR TIBLAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTAN | IEOUS ENDOSCOPIC APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 5047Q4GZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBILAL ARTERY WITH FOUR OR MORE INTRALLUMINAL DEVICES, PROCURATED SHODSCO | |
| | • |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q426 PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047Q4ZZ PX ICD-10 DILATION OF LEFT ANTERIOR TIBIAL ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R046 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN AP | PROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R04Z PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R056 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OP | PEN APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R05Z PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 10478056 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING DIVINES, DEVICES, OR | |
| Peripheral Vascular Disease (PVD) or PVD \$047R06Z PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH | |
| Peripheral Vascular Disease (PVD) or PVD \$ 047R076 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL D | |
| Peripheral Vascular Disease (PVD) or PVD \$047R07Z PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN A | APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R0D6 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 5 047R0DZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH INTRALUMINAL DEVICE, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047R0E6 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R0EZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$ 047R0FZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R0G6 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN AI | PPROACH Established CVD component |
| | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD \$047R0GZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH | |
| | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 047R026 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH | Established CVD component Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R0Z6 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R0ZZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH | Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R0Z6 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R0ZZ PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA | Established CVD component ANEOUS APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R026 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PROPRIED TO DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROA | Established CVD component ANEOUS APPROACH Established CVD component ACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R026 Pripheral Vascular Disease (PVD) or PVD 1047R027 Pripheral Vascular Disease (PVD) or PVD 1047R027 Pripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PRIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PE | Established CVD component ANEOUS APPROACH Established CVD component ESTABLISHED CVD component ESTABLISHED CVD component ERCUTANEOUS APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PROFESSOR (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION DEVICES DEVICE | Established CVD component ANEOUS APPROACH Established CVD component ACH Established CVD component ERCUTANEOUS APPROACH Established CVD component PPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R345 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 | Established CVD component ANEOUS APPROACH Established CVD component Established CVD component ERCUTANEOUS APPROACH Established CVD component ESTABLISHED CVD component ESTABLISHED CVD component ESTABLISHED CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PROFESSOR (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION DEVICES DEVICE | Established CVD component ANEOUS APPROACH Established CVD component Established CVD component ERCUTANEOUS APPROACH Established CVD component ESTABLISHED CVD component ESTABLISHED CVD component ESTABLISHED CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R345 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 | Established CVD component ANEOUS APPROACH Established CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 047R026 Pripheral Vascular Disease (PVD) or PVD : 047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD : 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TORUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD : 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TORUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL Vascular Disease (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL Vascular Disease (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PINEL VASCULAR DISEASE (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTATION, WITH FORCE OR MORE DR | ANEOUS APPROACH Established CVD component ACH Established CVD component ERCUTANEOUS APPROACH Established CVD component APPROACH Established CVD component ERECUTANEOUS APPROACH Established CVD component ERECUTANEOUS APPROACH Established CVD component EVCES, PERCUTANEOUS |
| Peripheral Vascular Disease (PVD) or PVD 1047R026 Pripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DAVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DAVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DAVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DAVICES, PERCUTANE | ANEOUS APPROACH Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R022 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R022 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PE Peripheral Vascular Disease (PVD) or PVD 1047R352 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PE Peripheral Vascular Disease (PVD) or PVD 1047R352 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PE Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PE Peripheral Vascular Disease (PVD) or PVD 1047R362 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PE PERIPHERAL Vascular Disease (PVD) or PVD 1047R362 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT P | Established CVD component ANEOUS APPROACH Established CVD component ESTABLISHED CVD component EVICES, PERCUTANEOUS ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 047R026 Pripheral Vascular Disease (PVD) or PVD : 047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD : 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD : 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TIRED ENDUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Peripheral Vascular Disease (PVD) or PVD : 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER Peripheral Vascular Disease (PVD) or PVD : 047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPPHERAL VASCULAR DISEASE (PVD) or PVD : 047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PROPRICTION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PROPRIED OF PVD : 047R3765 | Established CVD component ANEOUS APPROACH Established CVD component ESTABLISHE CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R345 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R306 PX ICD-10 DILATION OF RIGHT POSTERIO | ANEOUS APPROACH Established CVD component ANEOUS APPROACH Established CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R325 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PROPRIED VASCULAR | Established CVD component ANEOUS APPROACH EStablished CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL Vascular Disease (PVD) or PVD 1047R362 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTR | ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 1047R325 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PERIPHERAL VASCULAR DISEASE (PVD) OR PVD 1047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUT PROPRIED VASCULAR | ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER PERIPHERAL Vascular Disease (PVD) or PVD 1047R362 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PER DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTR | ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD: 047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R3306 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R3366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY | ANEOUS APPROACH ANEOUS APPROACH ACH ACH BESTABIISHED CVD component ESTABIISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD : 0.478025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD : 0.478027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD : 0.478342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD : 0.478356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478367 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478302 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD : 0.478302 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVI | ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R367 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL | Established CVD component ANDOUS APPROACH Established CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD: 047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, DEVA APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R367 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FURD OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PERIPHERAL Vascular Disease (PVD) or PVD: 047R3102 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PCP PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R316 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PCP PICH | Established CVD component ANEOUS APPROACH Established CVD component ERCUTANEOUS APPROACH Established CVD component ERCUTANEOUS APPROACH Established CVD component ESTABLISHED CVD cVD c |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA Peripheral Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R367 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROA PERIPHERAL Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL | Established CVD component ANDOUS APPROACH Established CVD component ESTABLISHED CVD component |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DEPENDENT VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PROPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGH | ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 5047R026 Pripheral Vascular Disease (PVD) or PVD 5047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 5047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PROPERTY OF PVD 5047R347 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH P | ANEOUS APPROACH ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 1047R025 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 1047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, OPEN APPROACH PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R355 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL Vascular Disease (PVD) or PVD 1047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A Peripheral Vascular Disease (PVD) or PVD 1047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS A DEPENDENT VASCULAR DISEASE (PVD) or PVD 1047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PROPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 1047R316 PX ICD-10 DILATION OF RIGH | ANEOUS APPROACH ANEOUS APPROACH ANEOUS APPROACH ACH ACH ACH ACH ACH ACH ACH |
| Peripheral Vascular Disease (PVD) or PVD 5047R026 Pripheral Vascular Disease (PVD) or PVD 5047R027 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD 5047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA PROPERTY OF PVD 5047R347 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Peripheral Vascular Disease (PVD) or PVD 5047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R377 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R376 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD 5047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH P | Established CVD component ANEOUS APPROACH ESTablished CVD component Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD: 047R325 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R342 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROAPPEORAL Peripheral Vascular Disease (PVD) or PVD: 047R352 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROAPPEORAL Peripheral Vascular Disease (PVD) or PVD: 047R352 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R352 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEase (PVD) or PVD: 047R3727 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEase (PVD) or PVD: 047R365 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH TIME DILATION DEVICES, PERCUTANEOUS APPROACH PERIPHERAL VASCULAR DISEASE (PVD) or PVD | Established CVD component ANEOUS APPROACH ESTablished CVD component Established CVD component |
| Peripheral Vascular Disease (PVD) or PVD: 047R0Z5 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, OPEN APPROACH Peripheral Vascular Disease (PVD) or PVD: 047R346 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R347 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA Peripheral Vascular Disease (PVD) or PVD: 047R356 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTA PERIPHERAL VASCULAR DISEASE (PVD) or PVD: 047R366 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS Peripheral Vascular Disease (PVD) or PVD: 047R367 PX ICD-10 DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS PERPORACH PERPORA | ANEOUS APPROACH Established CVD component |


TYPE 1 DIABETES MELLITUS WITH SEVERE NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT


DIABETES MELLITUS DUE TO UNDERLYING CONDITION WITH PROLIFERATIVE DIABETIC RETINOPATHY


DRUG OR CHEMICAL INDUCED DIABETES MELLITUS WITH PROLIFERATIVE DIABETIC RETINOPATHY


Acute coronary/cerebro-vascular event


Acute coronary/cerebro-vascular event


Acute coronary/cerebro-vascular event

Acute coronary/cerebro-vascular event


ATHEROSCLEROSIS OF NATIVE CORONARY ARTERY OF TRANSPLANTED HEART WITH ANGINA PECTORIS Acute coronary/cerebro-vascular event


ICD-10

BREAKDOWN (MECHANICAL) OF VASCULAR DIALYSIS CATHETER, INITIAL ENCOUNTER

DX

CKD stage 5, End-stage renal disease, dialysis or renal transplant T82.41XA


DX

ICD-10

HEPATIC SCLEROSIS

Decompensation event) component

Cirrhosis

K74.1

PROLONGED NURSING FACILITY EVALUATION AND MANAGEMENT SERVICE(S) BEYOND THE TOTAL TIME FOR THE PRIMARY SERVICE (WHEN THE PRIMARY SERVICE HAS BEEN SELECTED USING TIME ON THE DATE OF THE PRIMARY SERVICE); EACH ADDITIONAL 15 MINUTES BY THE PHYSICIAN OR


End stage liver disease (Cirrhosis + Decompensation event) component


PERIPHERAL T-CELL LYMPHOMA, NOT ELSEWHERE CLASSIFIED, LYMPH NODES OF HEAD, FACE, AND


| Pregnancy O16.3 DX ICD-10 UNSP Pregnancy O16.4 DX ICD-10 UNSP Pregnancy O16.5 DX ICD-10 UNSP Pregnancy O16.9 DX ICD-10 UNSP | PECIFIED MATERNAL HYPERTENSION, SECOND TRIMESTER PECIFIED MATERNAL HYPERTENSION. THIRD TRIMESTER |
|---|---|
| Pregnancy O16.4 DX ICD-10 UNSP Pregnancy O16.5 DX ICD-10 UNSP Pregnancy O16.9 DX ICD-10 UNSP | |
| Pregnancy O16.5 DX ICD-10 UNSP Pregnancy O16.9 DX ICD-10 UNSP | PECIFIED MATERNAL HYPERTENSION, COMPLICATING CHILDBIRTH |
| Pregnancy O16.9 DX ICD-10 UNSP | ECIFIED MATERIAL HYPERTENSION, COMPLICATING CHILDBIRTH |
| | PECIFIED MATERNAL HYPERTENSION, UNSPECIFIED TRIMESTER |
| | ORRHAGE IN EARLY PREGNANCY |
| · · | ATENED ABORTION |
| · · | R HEMORRHAGE IN EARLY PREGNANCY |
| | ORRHAGE IN EARLY PREGNANCY, UNSPECIFIED |
| · · | SSIVE VOMITING IN PREGNANCY |
| · · | HYPEREMESIS GRAVIDARUM |
| | REMESIS GRAVIDARUM WITH METABOLIC DISTURBANCE |
| | VOMITING OF PREGNANCY |
| | R VOMITING COMPLICATING PREGNANCY |
| · · | TING OF PREGNANCY, UNSPECIFIED |
| · · | OUS COMPLICATIONS AND HEMORRHOIDS IN PREGNANCY |
| · · | COSE VEINS OF LOWER EXTREMITY IN PREGNANCY |
| | COSE VEINS OF LOWER EXTREMITY IN PREGNANCY, UNSPECIFIED TRIMESTER |
| | COSE VEINS OF LOWER EXTREMITY IN PREGNANCY, FIRST TRIMESTER |
| | COSE VEINS OF LOWER EXTREMITY IN PREGNANCY, SECOND TRIMESTER |
| | COSE VEINS OF LOWER EXTREMITY IN PREGNANCY, THIRD TRIMESTER |
| | TAL VARICES IN PREGNANCY |
| | TAL VARICES IN PREGNANCY, UNSPECIFIED TRIMESTER |
| Pregnancy 022.11 DX ICD-10 GENIT | TAL VARICES IN PREGNANCY, FIRST TRIMESTER |
| Pregnancy 022.12 DX ICD-10 GENIT | TAL VARICES IN PREGNANCY, SECOND TRIMESTER |
| Pregnancy 022.13 DX ICD-10 GENIT | TAL VARICES IN PREGNANCY, THIRD TRIMESTER |
| Pregnancy O22.2 DX ICD-10 SUPE | RFICIAL THROMBOPHLEBITIS IN PREGNANCY |
| Pregnancy O22.20 DX ICD-10 SUPE | RFICIAL THROMBOPHLEBITIS IN PREGNANCY, UNSPECIFIED TRIMESTER |
| Pregnancy O22.21 DX ICD-10 SUPE | RFICIAL THROMBOPHLEBITIS IN PREGNANCY, FIRST TRIMESTER |
| Pregnancy O22.22 DX ICD-10 SUPE | RFICIAL THROMBOPHLEBITIS IN PREGNANCY, SECOND TRIMESTER |
| Pregnancy O22.23 DX ICD-10 SUPE | RFICIAL THROMBOPHLEBITIS IN PREGNANCY, THIRD TRIMESTER |
| Pregnancy O22.3 DX ICD-10 DEEP | PHLEBOTHROMBOSIS IN PREGNANCY |
| Pregnancy 022.30 DX ICD-10 DEEP | PHLEBOTHROMBOSIS IN PREGNANCY, UNSPECIFIED TRIMESTER |
| Pregnancy 022.31 DX ICD-10 DEEP | PHLEBOTHROMBOSIS IN PREGNANCY, FIRST TRIMESTER |
| | PHLEBOTHROMBOSIS IN PREGNANCY, SECOND TRIMESTER |
| | PHLEBOTHROMBOSIS IN PREGNANCY, THIRD TRIMESTER |
| | DRRHOIDS IN PREGNANCY |
| | DRRHOIDS IN PREGNANCY, UNSPECIFIED TRIMESTER |
| | DRRHOIDS IN PREGNANCY, FIRST TRIMESTER |
| | DRRHOIDS IN PREGNANCY, SECOND TRIMESTER |
| | DRRHOIDS IN PREGNANCY, THIRD TRIMESTER |
| | BRAL VENOUS THROMBOSIS IN PREGNANCY |
| | BRAL VENOUS THROMBOSIS IN PREGNANCY, UNSPECIFIED TRIMESTER |
| | BRAL VENOUS THROMBOSIS IN PREGNANCY, FIRST TRIMESTER |
| · · | BRAL VENOUS THROMBOSIS IN PREGNANCY, SECOND TRIMESTER |
| | BRAI VENOUS THROMBOSIS IN PREGNANCY, THIRD TRIMESTER |
| | R VENOUS COMPLICATIONS IN PREGNANCY |
| | R VENOUS COMPLICATIONS IN PREGNANCY |
| | R VENOUS COMPLICATIONS IN PREGNANCY, FIRST TRIMESTER |
| · · | R VENOUS COMPLICATIONS IN PREGNANCY, SECOND TRIMESTER |
| · · | R VENOUS COMPLICATIONS IN PREGNANCY, THIRD TRIMESTER |
| | R VENOUS COMPLICATIONS IN PREGNANCY, UNSPECIFIED TRIMESTER |
| | OUS COMPLICATION IN PREGNANCY, UNSPECIFIED |
| | DUS COMPLICATION IN PREGNANCY, UNSPECIFIED, UNSPECIFIED TRIMESTER |
| | OUS COMPLICATION IN PREGNANCY, UNSPECIFIED, FIRST TRIMESTER |
| | OUS COMPLICATION IN PREGNANCY, UNSPECIFIED, SECOND TRIMESTER |
| | OUS COMPLICATION IN PREGNANCY, UNSPECIFIED, THIRD TRIMESTER |
| | CTIONS OF GENITOURINARY TRACT IN PREGNANCY |
| | CTIONS OF GENTOOKINAKY TRACT IN PREGNANCY |
| · · | CTIONS OF KIDNEY IN PREGNANCY, UNSPECIFIED TRIMESTER |
| | CTIONS OF KIDNEY IN PREGNANCY, UNSPECIFIED TRIVIESTER |
| | CTIONS OF KIDNEY IN PREGNANCY, SECOND TRIMESTER CTIONS OF KIDNEY IN PREGNANCY, THIRD TRIMESTER |
| Pregnancy O23.1 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY |
| | CTIONS OF BLADDER IN PREGNANCY, UNSPECIFIED TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, FIRST TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC | |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC Pregnancy O23.12 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC Pregnancy O23.12 DX ICD-10 INFEC Pregnancy O23.13 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER CTIONS OF BLADDER IN PREGNANCY, THIRD TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC Pregnancy O23.12 DX ICD-10 INFEC Pregnancy O23.13 DX ICD-10 INFEC Pregnancy O23.2 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER<br>CTIONS OF BLADDER IN PREGNANCY, THIRD TRIMESTER<br>CTIONS OF URETHRA IN PREGNANCY |
| Pregnancy 023.10 DX ICD-10 INFEC Pregnancy 023.11 DX ICD-10 INFEC Pregnancy 023.12 DX ICD-10 INFEC Pregnancy 023.13 DX ICD-10 INFEC Pregnancy 023.2 DX ICD-10 INFEC Pregnancy 023.20 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER CTIONS OF BLADDER IN PREGNANCY, THIRD TRIMESTER CTIONS OF URETHRAIN PREGNANCY CTIONS OF URETHRAIN PREGNANCY, UNSPECIFIED TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC Pregnancy O23.12 DX ICD-10 INFEC Pregnancy O23.13 DX ICD-10 INFEC Pregnancy O23.2 DX ICD-10 INFEC Pregnancy O23.20 DX ICD-10 INFEC Pregnancy O23.21 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER CTIONS OF BLADDER IN PREGNANCY, THIRD TRIMESTER CTIONS OF URETHRA IN PREGNANCY, UNSPECIFIED TRIMESTER CTIONS OF URETHRA IN PREGNANCY, UNSPECIFIED TRIMESTER CTIONS OF URETHRA IN PREGNANCY, FIRST TRIMESTER |
| Pregnancy O23.10 DX ICD-10 INFEC Pregnancy O23.11 DX ICD-10 INFEC Pregnancy O23.12 DX ICD-10 INFEC Pregnancy O23.13 DX ICD-10 INFEC Pregnancy O23.2 DX ICD-10 INFEC Pregnancy O23.20 DX ICD-10 INFEC Pregnancy O23.21 DX ICD-10 INFEC Pregnancy O23.22 DX ICD-10 INFEC | CTIONS OF BLADDER IN PREGNANCY, SECOND TRIMESTER CTIONS OF BLADDER IN PREGNANCY, THIRD TRIMESTER CTIONS OF URETHRAIN PREGNANCY CTIONS OF URETHRAIN PREGNANCY, UNSPECIFIED TRIMESTER |


CONTINUING PREGNANCY AFTER SPONTANEOUS ABORTION OF ONE FETUS OR MORE, FIRST


CONTINUING PREGNANCY AFTER ELECTIVE FETAL REDUCTION OF ONE FETUS OR MORE, SECOND


MATERNAL CARE FOR KNOWN OR SUSPECTED PLACENTAL INSUFFICIENCY, SECOND TRIMESTER,


MATERNAL CARE FOR OTHER KNOWN OR SUSPECTED POOR FETAL GROWTH, THIRD TRIMESTER,


DISEASES OF THE DIGESTIVE SYSTEM COMPLICATING PREGNANCY, CHILDBIRTH AND THE


Proliferative retinopathy or maculopathy


SUBSEQUENT NURSING FACILITY CARE, PER DAY, FOR THE EVALUATION AND MANAGEMENT OF A NEW OR ESTABLISHED PATIENT, WHICH REQUIRES AT LEAST TWO OF THESE THREE KEY COMPONENTS: A PROBLEM FOCUSED INTERVAL HISTORY; A PROBLEM FOCUSED EXAMINATION; MEDICAL DECISION


```
COLLIDANA DI TROCAS DI RETRINO CERRAL ARREY

COLLIDANA DEI TROCAS DI RETRINO CERRAL ARREY

COLLIDANA DEI TROCAS DI PARI ARRES CERRALA, ARREY

COLLIDANA DEI TROCAS DI PARI ARRES CERRALA, ARREY

COLLIDANA DEI TROCAS DI RETRINO ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI AR
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        CD-10

Rominian Stockes

Rominian Sto
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                            166.1
166.12
166.12
166.13
166.19
166.2
166.2
166.22
166.23
166.3
166.8
166.9
20
41
42
21
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                            MINISTRAY STRAW, WITH COSTRUCTION, WITHOUT GAMBERS

REALITION FERROR.
```

### Flowchart for Cohort Assembly

<u>Link to Aetion reports:</u>

<u>Date conducted:</u>

Semaglutide injection vs Sitagliptin

Marketscan-

https://bwh-dope.aetion.com/project/2322/cohort/59482/116371/comparative/basics

Optum-

https://bwh-dope.aetion.com/project/2321/cohort/59484/116373/comparative/basics

Medicare-

https://bwh-dope.aetion.com/project/2323/cohort/59486/116375/comparative/basics 8/2/24

| | • | Optum<br>(Dec 05, 2017 - Feb 29, 2024) | | Marketscan<br>(Dec 05, 2017 - December 31,<br>2022) | | Medicare<br>(Dec 05, 2017 - December 31, 2020) |
|---|---|---|---|---|---|---|
| | Less Excluded Patients | Remaining<br>Patients | Less Excluded Patients | Remaining<br>Patients | Less Excluded Patients | Remaining<br>Patients |
| Patients in dataset | | 93,159,383 | | 119,592,975 | | 28,874,258 |
| Patient with cohort entry criteria (Exposure: Semaglutide injection, Refrence: Sitaglitpin) | | | | | | |
| Date of dispensing is cohort entry date (CED, 0,0) | | 889000 | | 693822 | | 988554 |
| Excluded due to insufficient enrollment (30 day gap allowed) (-180, 0) | -134,394 (15%) | 754,606 | -72,103 (10%) | 621,719 | -246,334 (25%) | 742,220 |
| Exclude due to prior use of reference (-180, -1) | -247,070 (33%) | 507536 | -290,765 (47%) | 330954 | -527,137 (71%) | 215083 |
| Exclude due to prior use of reference (-180, -1) | -321,331 (63%) | 186205 | -219,094 (66%) | 111860 | -63,844 (30%) | 151239 |
| Excluded because patient qualified in >1 exposure category | -36 (<1%) | 186,169 | -38 (<1%) | 111,822 | -15 (<1%) | 151,224 |
| Excluded based on Inclusion: Type 2 DM (-180, 0) | -16,751 (9%) | 169,418 | -20,614 (18%) | 91,208 | -2,167 (1%) | 149,057 |
| Excluded based on Inclusion: Antidiabetic medication score | -2,282 (1%) | 167,136 | -1,367 (1%) | 89,841 | -1,510 (1%) | 147,547 |
| Excluded based on Inclusion: >=50 years with established CVD OR >=60 years with subclinical CVD (-180, 0) | | | | | | |
| Exclude if patient is between 50 and 60 years of age without established CVD | -11,310 (7%) | 155,826 | -20,091 (22%) | 69,750 | -0 (<1%) | 147,547 |
| Exclude if patient is greater than or equal to 60 years of age without established or subclinical CVD | -45,814 (29%) | 110,012 | -18,907 (27%) | 50,843 | -44,213 (30%) | 103,334 |
| Excluded based on Age (<=49 years) | -9,893 (9%) | 100,119 | -18,887 (37%) | 31,956 | -0 (<1%) | 103,334 |
| Excluded based on Exclusion: Use of Sitagliptin/Semaglutide [any formulations] (-180, -1) | -4,191 (4%) | 95,928 | -1,497 (5%) | 30,459 | -5,165 (5%) | 98,169 |
| Excluded based on Exclusion: Type 1 DM (-180, 0) | -1,463 (2%) | 94,465 | -565 (2%) | 29,894 | , , , | 96,084 |
| Excluded based on Exclusion: Gestational DM (-180, 0) | -0 (<1%) | 94,465 | -0 (<1%) | 29,894 | , , , | 96,084 |
| Excluded based on Exclusion: Secondary DM (-180, 0) | -987 (1%) | 93,478 | -332 (1%) | 29,562 | ` ' | 94,680 |
| Excluded based on Exclusion: Pramlintide, Other DPP4i/GLP1 (-180, 0) | -5,383 (6%) | 88,095 | -1,491 (5%) | 28,071 | -4,452 (5%) | 90,228 |
| Excluded based on Exclusion: Bolus (short acting insulin) (-90, 0) | -2,841 (3%) | 85,254 | -399 (1%) | 27,672 | -1,056 (1%) | 89,172 |
| Excluded based on Exclusion: HONK (-90, 0) | -192 (<1%) | 85,062 | -60 (<1%) | 27,612 | -256 (<1%) | 88,916 |
| Excluded based on Exclusion: Diabetic ketoacidosis (-90, 0) | -91 (<1%) | 84,971 | -36 (<1%) | 27,576 | -121 (<1%) | 88,795 |
| Excluded based on Exclusion: History of pancreatitis (-180, 0) | -163 (<1%) | 84,808 | -49 (<1%) | 27,527 | -239 (<1%) | 88,556 |
| Excluded based on Exclusion: Acute coronary/cerebrovascular event (-90, 0) | -921 (1%) | 83,887 | -554 (2%) | 26,973 | -1,589 (2%) | 86,967 |
| Excluded based on Exclusion:Heart failure class IV (-180, 0) | -171 (<1%) | 83,716 | -35 (<1%) | 26,938 | -0 (<1%) | 86,967 |
| Excluded based on Exclusion: History of MEN-2 (-180, 0) | -0 (<1%) | 83716 | -0 (<1%) | 26938 | -2 (<1%) | 86965 |
| Excluded based on Exclusion: Personal history of non-familial medullary thyroid carcinoma (-180, 0) | -65 (<1%) | 83651 | -20 (<1%) | 26918 | -94 (<1%) | 86871 |
| Excluded based on Exclusion: End-stage renal disease (-180, 0) | -501 (<1%) | 83150 | -163 (<1%) | 26755 | -781 (<1%) | 86090 |
| Excluded based on Exclusion: End stage liver disease (-180, 0) | -70 (<1%) | 83080 | -24 (<1%) | 26731 | -121 (<1%) | 85969 |
| Excluded based on Exclusion: Organ transplant (-180, 0) | -76 (<1%) | 83004 | -22 (<1%) | 26709 | -64 (<1%) | 85905 |
| Excluded based on Exclusion: Cancer (-1825, 0) | -3,862 (5%) | 79142 | -1,105 (4%) | 25604 | -6,235 (7%) | 79670 |
| Excluded based on Exclusion: Pregnancy (-180, 0) | -3 (<1%) | 79139 | -0 (<1%) | 25604 | ` ' | 79667 |
| Excluded based on Exclusion: Drug abuse or dependence (-180, 0) | -693 (<1%) | 78446 | -86 (<1%) | 25518 | | 79253 |
| Excluded based on Exclusion: Proliferative retinopathy or maculopathy (-90, 0) | -391 (<1%) | 78055 | -118 (<1%) | 25400 | ` ' | 78793 |
| Excluded based on Exclusion: Nursing home stay (-180, 0) | -479 (<1%) | 77576 | -91 (<1%) | 25309 | , , | 77487 |
| Excluded based on Exclusion: Missing Age (-180, 0) | -0 (<1%) | 77,576 | -0 (<1%) | 25,309 | - ' ' ' | 77,487 |
| Excluded based on Exclusion: Missing Gender (-180, 0) | -1 (<1%) | 77,575 | -0 (<1%) | 25,309 | | 77,487 |
| Patients in Exposure Group | | 38,980 | | 9,698 | | 12,773 |
| Patients in Referent Group | | 38,595 | | 15,611 | | 64,714 |
| Total patients | | 77,575 | | 25,309 | | 77,487 |

8/2/24

8/2/24

### Appendix 4. 1st Feasibility Assessment

- Table of Contents

  A. Patient characteristics by treatment group

  B. Summary Parameters of Study Population

  C. Median Follow up Time in Overall Study Population

  D. Reasons for Censoring in Overall Study Population

  E. Initial Power Assessment

  F. Aetion Report Links

  G. Review by Principal Investigator and FDA

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a 1.1 PS-matched comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

Optum: Study period between 5th Dec 2017 - 29th February 2024 Marketscan: Study period between 5th Dec 2017 - 31st Dec 2022 Medicare: Study period between 5th Dec 2017 - 31st Dec 2020

| UNMATCHED | | Optum | | | Truven | | | Medicare | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference-Sitagliptin | Exposure - Semagiutide inj | Difference | Reference-Sitagliptin | Exposure - Semaglutide inj | Difference | Reference-Sitagliptin | Exposure - Semagiutide inj | Difference |
| Number of patients | 38,548 | 38,871 | -(-,-) | 15,588 | 9,686 | - (-, -) | 64,645 | 12,751 | - (-, -) |
| Age | | | | | | | | | |
| mean (sd) | 73.40 (7.94) | 68.10 (7.78) | 5.31 (5.19, 5.42) | 67.77 (10.50) | 61.61 (7.72) | 6.16 (5.93, 6.38) | 75.55 (7.09) | 71.99 (5.28) | 3.56 (3.46, 3.67) |
| median [IQR] | 73.00 [68.00, 79.00] | 68.00 [63.00, 73.00] | - (-,-) | 66.00 [60.00, 76.00] | 61.00 [56.00, 65.00] | · (·, ·) | 75.00 [70.00, 80.00] | 71.00 [68.00, 75.00] | - (-, -) |
| Gender without unknown | | | | | | | | | |
| Male; n (%) | 18,789 (48.7%) | 18,584 (47.8%) | 0.9% (0.2%, 1.6%) | 9,157 (58.7%) | 5,544 (57.2%) | 1.5% (0.2%, 2.8%) | 31,747 (49.1%) | 6,753 (53.0%) | -3.9% (-4.8%, -2.9%) |
| Female; n (%) | 19,759 (51.3%) | 20,287 (52.2%) | -0.9% (-1.6%, -0.2%) | 6,431 (41.3%) | 4,142 (42.8%) | -1.5% (-2.8%, -0.2%) | 32,898 (50.9%) | 5,998 (47.0%) | 3.9% (2.9%, 4.8%) |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.77 (2.42) | 2.30 (2.18) | 0.48 (0.44, 0.51) | 1.99 (2.16) | 1.67 (1.87) | 0.32 (0.27, 0.37) | 2.06 (2.18) | 1.97 (2.00) | 0.09 (0.05, 0.13) |
| median (IQR) | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | -(-,-) | 2.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 2.00 [0.00, 3.00] | 2.00 [0.00, 3.00] | - (-, -) |

### B. Summary Parameters of Overall Study Population

| UNMATCHED | Optum | Truven | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in full<br>cohort | 77,575 | 25,309 | 77,487 |
| Number of patients dropped<br>as incomplete cases | 0 | 0 | 0 |
| Number of patients that did<br>not begin follow-up | 156 | 35 | 91 |
| Number of patients in<br>analytic cohort | 77,419 | 25,274 | 77,396 |
| Number of events | 1630 | 437 | 2443 |
| Number of person-years | 34,592.94 | 11,760.67 | 37,109.92 |
| Number of patients in group: Reference: Sitagliptin | 38,548 | 15,588 | 64,645 |
| Number of patients in<br>group: Exposure:<br>Semaglutide injection | 38,871 | 9,686 | 12,751 |
| Risk per 1,000 patients | 21.05 | 17.29 | 31.56 |
| Rate per 1,000 person-<br>years | 47.12 | 37.16 | 65.83 |

## C. Median Follow up Time in Overali Study Population

| Ī | UNMATCHED | Optum | Truven | Medicare |
|---|---|---|---|---|
| Ī | | | Median Follow-Up Time<br>(Days) [IQR] | Median Follow-Up Time<br>(Days) [IQR] |
| - | Overall Patient Population | 118 [62, 242] | 118 [58, 285] | 126 [68, 287] |

### D. Reasons for Censoring in Overall Study Population

| UNMATCHED | Optum | Truven | Medicare |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 1,630 (2.1%) | 437 (1.7%) | 2,442 (3.2%) |
| Start of an additional<br>exposure | 681 (0.9%) | 285 (1.1%) | 488 (0.6%) |
| End of index exposure | 42,288 (54.6%) | 12,153 (48.1%) | 38,415 (49.6%) |
| Maximum follow-up time | 11,485 (14.8%) | 4,756 (18.8%) | 14,045 (18.1%) |
| Specified date reached | 10,798 (13.9%) | 3,008 (11.9%) | 13,447 (17.4%) |
| End of patient enrollment | 5,793 (7.5%) | 3,441 (13.6%) | 3,102 (4.0%) |
| Extra censor: Medications<br>(Pramlintide/Other<br>DPP4i/GLP) + Nursing<br>home + Oral Sema began | 4,744 (6.1%) | 1,194 (4.7%) | 5,457 (7.1%) |

| Fine stratification | Optum | Truven | Medicare |
|---------------------|--------|--------|----------|
| Exposure | 38,871 | 9,686 | 12,751 |
| Reference | 34,693 | 14,029 | 58,181 |

| Matched number | Optum | Truven | Medicare |
|----------------|--------|--------|----------|
| Exposure | 18,531 | 9,163 | 12,751 |
| Reference | 18,531 | 9,163 | 12,751 |

The clinical trial was powered to find the absolute risk difference of 4%. Using the values of risk from the trial, we calculated the risk ratio and calculated the estimated power for a range of effect estimates from the lower to the upper 95% confidence limit of the HR observed in the RCT.

| Superiority Analysis (fine strati) | |
|------------------------------------|---------|
| Number of patients matched | |
| Reference | 106,903 |
| Exposed | 61,308 |
| Rick nor 1 000 nationts | 25.04 |

| Superiority Analysis (1:1) | |
|----------------------------|-------|
| Number of patients | |
| matched | |
| Reference | 40,44 |
| Exposed | 40,44 |
| Rick nor 1 000 nationts | 25.0 |

Desired HR from RCT = RR from RCT

| Desired HR from RCT | 0.74 |
|---------------------------|--------|
| Alpha (2-sided) | 0.05 |
| Number of events expected | 4212.5 |
| Power | 1.0 |

| Desired HR from RCT | 0.7 |
|------------------------------|-------|
| Alpha (2-sided) | 0.0 |
| Number of events<br>expected | 2025. |
| Power | 1. |

### F. Aetion Report Links

Aetion report link:

For Semaglutide vs Sitagliotin cohort

Octum
Step 1: https://bwh-dope.aetion.com/project/2321/rwrs/116793
Step 2: https://bwh-dope.aetion.com/project/23221/rwrs/116381
Markstacan
Step 1: https://bwh-dope.aetion.com/project/23221/rws/116380
Step 2: https://bwh-dope.aetion.com/project/23221/rws/116389
Madicare
Step 1: https://bwh-dope.aetion.com/project/23221/rws/116389
Step 2: https://bwh-dope.aetion.com/project/2323/rwrs/116792
Step 2: https://bwh-dope.aetion.com/project/2323/rwrs/116385

### G. Review by principal investigator and FDA

Stop analyses until feasibility and power are reviewed by primary investigators and FDA.

| First review by FDA | Date reviewed: | 30th Sept 2024 |
|---|---|---|
| Final review and approval<br>by FDA after comments<br>were addressed | Date reviewed: | 3rd October 2024 |

### Appendix 5. 2nd Feasibility Assessment

### Table of Contents

- A. Median Follow up Time by Treatment Group
- B. Reasons for Censoring by Treatment Group
- C. Final Power Assessment
- E. Review by Principal Investigator and FDA

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a 1:1 PS-matched comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

### A. Median Follow Up Time by Treatment Group (Step 1)

| UNMATCHED | Optum | Truven | Medicare |
|---|---|---|---|
| | | Median Follow-Up Time<br>(Days) [IQR] | Median Follow-Up<br>Time (Days) [IQR] |
| Overall Patient<br>Population | 118 [62, 242] | 118 [58, 285] | 126 [68, 287] |

### B. Summary Parameters of Overall Study Population (Step 1)

| UNMATCHED | Optum | Truven | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in<br>full cohort | 77,575 | 25,309 | 77,487 |
| Number of patients<br>dropped as incomplete<br>cases | 0 | 0 | 0 |
| Number of patients<br>that did not begin<br>follow-up | 156 | 35 | 91 |
| Number of patients in<br>analytic cohort | 77,419 | 25,274 77,396 | |
| Number of events | 1630 | 437 | 2443 |
| Number of person-<br>years | 34,592.94 | 11,760.67 | 37,109.92 |
| Number of patients in<br>group: Reference:<br>Sitagliptin | 38,548 | 15,588 | 64,645 |
| Number of patients in<br>group: Exposure:<br>Semaglutide injection | 38,871 | 9,686 | 12,751 |
| Risk per 1,000<br>patients | 21.05 | 17.29 | 31.56 |
| Rate per 1,000<br>person-years | 47.12 | 37.16 | 65.83 |

### C. Reasons for Censoring in Overall Study Population (Step 1)

| UNMATCHED | Optum | Truven Medica | |
|---|---|---|---|
| Overall | Value | Value | Value |
| Outcome | 1,630 (2.1%) | 437 (1.7%) | 2,442 (3.2%) |
| Start of an additional<br>exposure | 681 (0.9%) | 285 (1.1%) | 488 (0.6%) |
| End of index exposure | 42,288 (54.6%) | 12,153 (48.1%) | 38,415 (49.6%) |
| Maximum follow-up<br>time | 11,485 (14.8%) | 4,756 (18.8%) | 14,045 (18.1%) |
| Specified date<br>reached | 10,798 (13.9%) | 3,008 (11.9%) | 13,447 (17.4%) |
| End of patient<br>enrollment | 5,793 (7.5%) | 3,441 (13.6%) | 3,102 (4.0%) |
| Extra censor:<br>Medications<br>(Pramlintide/Other<br>DPP4i/GLP) +<br>Nursing home + Oral<br>Sema began | 4,744 (6.1%) | 1,194 (4.7%) | 5,457 (7.1%) |

### D. Final Power Assessment (Step 3)

The clinical trial was powered to find the absolute risk difference of 4%. Using the values of risk from the trial, we calculated the risk ratio and calculated the estimated power for a range of effect estimates from the lower to the upper 95% confidence limit of the HR observed in the RCT.

calculate\_ess <- function(weights) { sum(weights)^2 / sum(weights^2)}

ess\_treatment\_1 <- calculate\_ess(soul\_fs\$psweight[soul\_fs\$Treatment == 1))
ess\_treatment\_0 <- calculate\_ess(soul\_fs\$psweight[soul\_fs\$Treatment == 0])

OPTUM: ESS for Reference: 6306.44 ESS for Exposure: 38,883

MARKETSCAN-ESS for Reference: 2,991.91 ESS for Exposure: 9,666

MEDICARE-ESS for Reference: 12,990 ESS for Exposure: 12,745

Numbers below are based on the PS assessed based on all the covariates given in the Balance - Table 1 sheet

| Superiority A | Superiority Analysis (fine strati) |
|------------------------------|------------------------------------|
| Number of patients | |
| matched | |
| Reference | 22,288 |
| Exposed | 61,294 |
| Risk per 1,000 patients | 25.04 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events<br>expected | 2093.2 |
| Power | 1.0 |

| Superiority | Analysis (1:1) |
|---------------------|----------------|
| Number of patients | |
| matched | |
| Reference | 32,554 |
| Exposed | 32,554 |
| Risk per 1,000 | |
| patients | 25.04 |
| Desired HR from RCT | 0.83 |
| Alpha (2-sided) | 0.05 |
| Number of events | 1630.5 |
| expected | |
| Power | 1.0 |

### E. Aetion Report Links

Aetion report link:

For Semaglutide vs Sitagliptin cohort

Optum
Step 1: https://bwh-dope.aetion.com/project/2321/rwrs/116793
Step 3: https://bwh-dope.aetion.com/project/2321/rwrs/116933

Marketscan
Step 1: https://bwh-dope.aetion.com/project/2322/rwrs/116807
Step 3: https://bwh-dope.aetion.com/project/2322/rwrs/116930

Medicare
Step 1: https://bwh-dope.aetion.com/project/2323/rwrs/116792
Step 3: https://bwh-dope.aetion.com/project/2323/rwrs/116931

# F. Review by Principal Investigator and FDA

Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| First review by FDA | Date reviewed: | 30th Sept 2024 |
|---|---|---|
| Final review and<br>approval by FDA<br>after comments were<br>addressed | Date reviewed: | 3rd October 2024 |
| Reason for stopping ( | if required): | |



### fine-stratified cstats, Optum: 0.50033



Exposure

### fine-stratified cstats, Marketscan: 0.50023



| 0.00 | 0.25 | 0.50<br>Propensity Scor | * | 0.75 | 1.00 | |
|---|---|---|---|---|---|---|
| Summary, PS distribution, Unadjusted cohort | | | | | | |
| MARKETSCAN | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 2.58E-05 | 0.989 | 0.242 | 0.16 | 0.0573 | 0.372 |
| Exposure | 0.00646 | 0.998 | 0.611 | 0.655 | 0.431 | 0.816 |

| Summary, PS distribution, 1:1 cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN | Minimum Maximum N | | Mean | Median | 25th pct | 75th pct |
| Reference | 0.00644 | 0.989 | 0.469 | 0.468 | 0.302 | 0.627 |
| Exposure | 0.00646 | 0.992 | 0.47 | 0.47 | 0.302 | 0.63 |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.058 | 38 | 1 | 0.272 | 0.058 | 1.08 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

### fine-stratified cstats, Medicare: 0.50008



| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.00007 | 0.975 | 0.123 | 0.0676 | 0.0213 | 0.169 |
| Exposure | 0.0025 | 0.971 | 0.379 | 0.342 | 0.186 | 0.55 |

| Summary, PS distribution, 1:1 cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.0025 | 0.963 | 0.324 | 0.299 | 0.17 | 0.458 |
| Exposure | 0.0025 | 0.963 | 0.325 | 0.299 | 0.17 | 0.458 |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.065 | 33.3 | 1 | 0.397 | 0.065 | 1.24 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

| Option: Usedjusted orbert Variable Stagliptis-reference Senaptide-sepoure 156 diff Number of patients 18,512 18,512 | Optum: 1.1 matched cohort Optum: Fine stratification cohort Stagligitis reference Samuglatide exposure 2d diff Stagligitis reference Samuglatide exposure 15,000 11,510 11,510 11,510 | Marketscan: Unadjusted cohort Sitagliptin - reference Semagluide - exposure Std dill 15.541 9,600 | Marketscan: 1.3 matched cohort Stagliptin - reference Semajuside - exposure 518 017 5.534 | Marketscan: Fine stratification cohort Stagliptin -reference Semaguide -exposure 15,224 9,666 | Medicare: Unadjusted cohert Stagliptin-reference Semajutide expassee 9:6 017 64,451 12,746 | Medicare: 1:3 matched cohort Stagligiss -esterence Semajuside -exposure 11,070 11,070 | Medicare: Fine stratification cohort Situgiptin - reference Semaguistic - exposure 63,414 12,745 |
|---|---|---|---|---|---|---|---|
| | 71.06 (7.64) 70.92 (7.49) 0.010 E8.22 (7.34) (68.10 (7.78)<br>8179 (51.3) 1920 (51.5) 0.004 2005 (3.8.2.9) 100.05 (52.2)<br>1051 (10.44) 1661 (10.4) 1222 (10.44) 1232 (10.44) 1232 (10.44) | 0.002 (67.79 (10.50) (41.61 (7.72) 0.67<br>6402 (41.2) 4138 (42.7) 0.031<br>0.02 (0.32) 0.323 | 53.15 (8.67) | 61.53 (8.15) 61.62 (7.72) 0.011<br>6396.8 (42.0) 4132.0 (42.7) 0.015<br>0.046<br>2619.2 (37.2) 1644.0 (37.0) | 75.55 (7.00) 71.99 (5.28) 0.57<br>22784 (50.9) 5995 (87.0) 0.077<br>12888 (20.0) 1972 (55.5) | 72.35(5.63) 72.32(5.38) 0.005<br>5262(47.5) 5265(47.6) 0.001<br>0.016<br>1783 (6.1) 1747 (15.8) | 71.92 (5.50) 71.98 (5.27) 0.01<br>10275.8 (47.7) 5994.0 (47.0) 0.014<br>0.021<br>0403.8 (44.9) 1977.0 (15.5) |
| Midwes(North Central, n (N) 4000 (15.6) 7666 (19.7) 5604 (19.7) 5604 (19.7) 5604 (19.7) 5604 (19.7) 5604 (19.7) 5605 (19.7) 56 | 7822 (12.77) 2821 (12.77) 7435 (19.4) 7661.0 (18.77) 8901 (15.48) 8878 (5.77) 7201 (18.76) 737 (18.77) 7375 (14.1) 7390 (16.77) 7375 (14.1) 7390 (16.77) 7390 (16 | 4820 [21.0] 2085 [21.5]<br>6170 [28.7] 5182 [25.5]<br>912 [5.9] 768 [7.9]<br>0.11 | 1287 (23.2) 1220 (23.9)<br>2755 (40.8) 2777 (60.2)<br>404 (7.3) 366 (7.2)<br>0.048 | 1005.0 (10.7) 2085.0 (21.6)<br>8270.0 (55.0) 5169.0 (53.5)<br>1229.8 (8.1) 768.0 (7.9)<br>0.027 | 13166 (D.5) 2878 (D.6)<br>27627 (4.59) 6083 (47.7)<br>10742 (16.7) 1812 (8.2) 0.875<br>2551 (D.0.1) 1864 (7.0) | 2464 (22.3) 2469 (22.1)<br>5371 (46.7) 5254 (47.5)<br>1652 (4.6) 1653 (34.6) 0.021 | 14050.1 (22.2) 2878.0 (22.6)<br>10755.9 (46.5) 6082.0 (47.7)<br>9134.1 (14.4) 1812.0 (14.2) 0.016<br>4413.7 (27.50) 923.0 (27.0) |
| 1003 Dan Origin (N) | 144(9.1) (42) 8.9 (156.4(4.1) (23) 8.9 (156.4(4.1) (23) 8.9 (156.4(4.1) (23) 8.9 (16) 8.9 (16 | 1848 [2-3] 1278 [4-2]<br>776 [5-6] 459 [4-7]<br>609 [1-9] 1212 [4-7]<br>227 [4-7] 408 [4-7] | 1130 (0.2) 1123 (0.3)<br>211 (5.6) 315 (5.7)<br>256 (4.7) 256 (4.3)<br>108 (5.6) 282 (5.1) | 2288.0 (4.8) 1378.0 (4.3)<br>740.9 (4.9) 459.0 (4.7)<br>550.2 (2.7) 233.0 (3.4)<br>630.6 (4.1) 408.0 (4.2) | 22006 [24.1] 4924 [28.7]<br>674 [7.4] 592 [5.1]<br>5900 [6.1] 559 [2.2]<br>645 [6.9] 1695 [3.3] | 4476 (0.4) 4462 (0.3)<br>1442 (0.39) 1582 (4.3)<br>1286 (0.17) 1302 (11.8)<br>1441 (0.10) 1408 (0.27) | 26800.1 (29.1) 4934.0 (38.7)<br>9496.5 (15.0) 4922.0 (15.1)<br>7951.3 (12.5) 1596.0 (12.2)<br>8316.8 (13.1) (465.0 (13.3) |
| 2000 2007 (CCC) 0 (N) 2007 (CCC) 2 | \$41,147.21 \$45,07.27 \$450,07.27 \$451,07.27 \$ | 7789(43) 494(5.1)<br>2420(15.6) 1400(24.6)<br>1921(12.4) 1795(39.2) | ##7 (6.1) ##5 (5.4)<br>1390 (5.1) 1355 (54.5)<br>1465 (36.5) 1506 (27.2) | 786.5 (5.0) | 6079 (s.d) 1742 (s.d.7) | 14/0 (12.4) 14/5 (12.9) | 142.0(1.7) |
| Microbal abuses of dependence, pt (N) 464 (F, 2) 472 (1.2) 0.004 | 185 (3.7) 185 (2.2) 0.003 49.8 (4.1) 47.2 (0.2) 185 (2.7) 440 (2.1) 185 (2.7) 440 (2.1) 185 (2.7) 184 (0.1) 184 (0.1 | 0.505 | 50 (0.59) 47 (0.81) 0.006<br>68 (0.59) 40 (0.71) 0.016<br>122 (5.8) 123 (6.6) 0.009<br>603 (10.9) 609 (11.0) 0.003<br>927 (12.81) 977 (17.5) 0.019 | 126.0 (0.8) 74.0 (0.8) 0.007<br>18.4 (0.6) 65.0 (0.5) 0.016<br>849.3 (5.6) 517.0 (5.3) 0.01<br>1795.8 (11.8) 1178.0 (12.2) 0.012<br>3425.2 (22.5) 2395.0 (22.8) 0.032 | 277 (9.6) 52 (9.5) 0.011<br>2576 (4.9) 274 (3.4) 0.161<br>7251 (11.3) 1191 (9.3) 0.061<br>10566 (16.3) 3061 (9.4.2) 0.197<br>(215 (9.6) 2857 (2.27) 0.361 | 57 p.5] 54 p.5] 0.004<br>166 (1.5) 166 (1.5) 0.001<br>1001 (0.0) 1082 (0.8) 0.002<br>2590 (2.4) 2576 (23.2) 0.002<br>2510 (10.5) 2100 (10.5) 0.001 | 103.7 (0.5) (2.0)(0.5) (0.001<br>166.9 (1.4) (74.0 (1.4) (0.001<br>1059.2 (0.6) (199.0 (1.3) (0.007<br>15732.0 (24.8) 1081.0 (12.2) (0.015<br>14932.9 (22.8) 2897.0 (22.7) (0.001 |
| Unspecified obstity; n PG | 294 [EA.3] [EA.2 (EA.5) 0.006 200.5 (20.4 (20.5 (20.4 (20.4 (20.5 (20.4 | 0.015 2102 (21.5) 22.86 (23.6) 0.347<br>0.005 1489 (26.6) 91.2 (24.4) 0.005<br>0.023 1051 (6.8) 788 (6.1) 0.052<br>0.066 2228 (20.8) 2090 (21.6) 0.02<br>0.066 2228 (20.8) 2090 (21.6) 0.02 | 1015 (18.3) 1021 (18.4) 0.003<br>134 (9.7) 550 (9.9) 0.009<br>180 (9.3) 187 (7.0) 0.005<br>1107 (20.0) 1138 (20.6) 0.014<br>1107 (20.0) 0.014 | 3304.1 (31.7) 2221.0 (23.0) 0.331<br>1411.0 (9.1) 999.0 (9.4) 0.004<br>1206.1 (7.9) 785.0 (8.1) 0.007<br>3340.9 (7.1) 7084.0 (71.6) 0.009<br>1340.9 (71.9) 0.004.0 (71.6) 0.009 | 9755 [15.1] 2322 [25.5] 0.24<br>10538 [16.3] 2103 [16.5] 0.004<br>4362 [8.3] 1231 [9.5] 0.1<br>12466 [19.7] 2322 [25.3] 0.124<br>12466 [19.7] 2322 [25.3] 0.125 | 2622 (23.7) 2605 (23.5) 0.004<br>1805 (77.1) 1862 (16.6) 0.012<br>275 (8.8) 166 (8.7) 0.001<br>2625 (23.7) 2636 (23.7) 0.001<br>2625 (23.7) 2636 (23.7) 0.001 | 16601.1 (26.2) 1252.0(25.5) 0.015<br>10846.2 (17.1) 2100.0 (16.5) 0.016<br>1008.0(0.5) 1211.0(3.3) 0.001<br>16277.9 (25.4) 1222.0(25.3) 0.008<br>16277.9 (25.4) 1222.0(25.3) 0.008 |
| Disbetes with unspecified constitution on PS 1007(10.8) 0.018(0.90.9) 0.028 | 224(16.7) 234(16.7) 0.001 1245.7(21.5) 1114.0(20.3) 1245.7(21.5) 1114.0(20.3) 1246.7(21.5) 1114.0(20.3) 1246.7(21.5) 12 | 0.055 1511(10.4) 1221(12.4) 0.051<br>0.002 255(1.6) 148(1.5) 0.009<br>0.001 1692(10.9) 118(11.5) 0.001<br>0.005 22(2.1) 205(2.1) 0.004<br>0.005 4856(3) 45516(7) 0.016 | 860[11.9] (455 (27.0) 0.003<br>75 [1.4] 75 (1.4) 0.001<br>581 (10.5) (403 (10.8) 0.012<br>118(7.4) 114(7.1) 0.005<br>180(8.5) 155 [8.4] 0.004 | 7110.8 (71.9) 1218.0 (12.6) 0.007<br>229.1 (1.6) 148.0 (1.5) 0.003<br>1787.2 (1.17) 114.0 (11.5) 0.007<br>468.8 (2.7) 203.0 (2.1) 0.038<br>1900.7 6.0 6.3 (2.1) 0.038 | 6782[7.4] 1195 g.4] 0.071<br>678 [1.5] 216 [1.7] 0.014<br>565 g.8] 1266 [0.2] 0.05<br>1220 [1.7] 229 [1.9] 0.01<br>236 g.8 g.9 0.01 0.01 | 999 (8-0) 1001 (8-0) 0.001<br>189 (1-7) 179 (1-6) 0.007<br>1072 (8-7) 1000 (8-6) 0.004<br>183 (1-7) 193 (1-7) 0.007<br>681 (6-7) 673 (6-7) 0.005 | \$004.1(0.6) \$1195.0(3.4) \$0.000 \$1020.0(1.6) \$125.0(1.7) \$0.004 \$126.0(1.7) \$0.004 \$126.0(1.0) \$1266.0(1.0.2) \$0.007 \$1201.7(1.6) \$1206.0(1.0.2) \$0.007 \$1201.7(1.6) \$1205.0(1.0.2) \$0.001 |
| Execution dynAmerization (IN) 942.0.41 1209 (1.4) 0.055 ingraphysemist, (PM) 7712 (PM) 7712 (PM) 7712 (PM) 0.064 ingraphysemist, DAV, MONCon (PM) 15070 (42.1) 16600 (44.2) 0.034 ingraphysemist, DAV, MONCon (PM) 15110 (14.2) 5322 (EM) 0.021 ingraphysemistry (PM) 15110 (14.2) 5322 (EM) 0.001 ingraphysemistry (PM) 15110 (14.2) 3235 (27.4) 0.001 | 486 (3.0) 489 (3.1) 0.001 1206 (8.1) 1207 (9.4) 1206 (9.1) 1207 (9.4) 1206 (9.5) 1206 (9.5) 1206 (9.5) 1206 (9.5) 1206 (9.5) 1207 (9.5) 1208 (9 | 100 | 165 (3.0) 157 (2.8) 0.000<br>623 (12.4) 646 (1.3) 0.000<br>240 (44.8) 450 (45.0) 0.004<br>472 (85.5) 476 (86.1) 0.014<br>1373 (70.1) 4405 (70.6) 0.004 | 467.4 (2.1) 203.0 (2.1) 0.004<br>1985.9 (2.10) 1299.0 (21.3) 0.009<br>755.5 (190.6) 1299.0 (21.3) 0.009<br>1295.7 (190.6) 1299.0 (21.3) 0.024<br>12085.2 (86.0) 8242.0 (84.4) 0.024<br>12085.2 (86.0) 8242.0 (84.3) 0.01 | 542 [0.8] 156 [1.2] 0.028<br>506 (17.9) 1110 [0.3] 0.051<br>22657 [16.2] 5052 [66.7] 0.224<br>62746 [75.6] 9410 [74.1] 0.024<br>7286 [76.8] 10.023 | 129 (1.2) 126 (1.1) 0.003<br>100 10 (2) 100 10 100 (1.1) 0.003<br>100 10 (2) 100 100 (1.1) 0.009<br>100 (1.4) 100 100 (1.1) 0.009<br>101 (1.1) 0.000<br>101 (1.1) 0.000<br>101 (1.1) 0.000<br>101 (1.1) 0.000 | 762.3 (2.2) 156.0 (1.2) 0.002<br>1008.7 (9.5) 1189.0 (9.3) 0.005<br>12955.1 (46.3) 925.0 (46.7) 0.006<br>12955.2 (46.3) 925.0 (46.7) 0.000<br>12955.3 (50.0) 0.006<br>12955.5 (50.0) 0.006 |
| | 2298[144] 2257 [6.1.7] 0.007 1647 (61.7.7) 5641.0[14.5] 1877 (11.7.7) 1841.23 0.007 1847 (11.7.7) 1841.23 0.007 1800.4[2.3] 1841.23 0.007 1800.4[2.3] 1841.23 0.007 1800.4[2.3] 1841.23 0.007 1800.4[2.3] 1841.23 0.007 1800.4[2.3] 1841.23 0.007 1841.23 0.00 | 0.005 1029 [13.1] 1039 [10.7] 0.072<br>0.095 416 [2.7] 122 [3.3] 0.038<br>0.095 416 [2.7] 122 [3.3] 0.038<br>0.091 705 [4.5] 460 [4.8] 0.01<br>0.094 7708 [49.8] 1078 [52.5] 0.057<br>0.094 7708 [49.8] 1078 [52.5] 0.057 | 384 (10.4) 374 (10.4) 0.006<br>156 (2.8) 152 (2.7) 0.004<br>345 (4.4) 240 (4.5) 0.004<br>283 (51.6) 280 (50.7) 0.004 | 1494.6 (6.8) 1038.0 (10.7) 0.03<br>41.2.5 (2.7) 220.0 (2.3) 0.035<br>573 (4.5) 600.0 (4.8) 0.014<br>7503.4 (5.1.9) 5063.0 (5.4) 0.01 | 10831 (16.8) 1846 (14.5) 0.064<br>1467 (7.3) 321 (7.5) 0.014<br>4681 (7.3) 929 (7.3) 0.001<br>3319 (51.7) 6870 (5.8) 0.04 | 1580 (14.4) 1601 (14.5) 0.003<br>261 (2.4) 262 (2.4) 0.001<br>819 (7.4) 801 (7.2) 0.006<br>502 (9.15) 5.005 (9.13) 0.002 | 9270.9(14.6) 1842.0(14.5) 0.005<br>1550.7(2.4) 223.0(2.5) 0.009<br>4723.7(74) 223.0(2.5) 0.009<br>34348.6(53.9) 4660.0(53.9) 0.005 |
| | 0001 120 | 0.0000 10000 (7.00) | 127 (Fig. 8) 12.5 (Fig. 9) 12.5 (Fig. 9) | 1278-3 (8-9) (193-0 (27) (20-2) (193-0 (27) | 10000 (20-0) 12000 (21-0) 0.0021<br>022 (1.4) 2000 (2.5) 0.017<br>71 (0.1) 15 (0.1) 0.002<br>11055 (17.7) 1882 (14.8) 0.065<br>11882 (18.4) 2166 (17.6) 0.028 | 188 (1.7) 176 (1.6) 0.0004<br>189 (1.7) 176 (1.6) 0.0004<br>189 (1.7) 176 (1.6) 0.0001<br>189 (1.7) 169 (1.7) 0.0001<br>169 (1.7) 169 (1.7) 0.001<br>1992 (17.5) 1888 (17.1) 0.001 | 1035-1(127-4) 12800-0(17-4) 0.0001<br>1035-1(169) 0.00-0(1.6) 0.001<br>98.1(0.2) 15.0(0.1) 0.01<br>98.1(0.2) 15.0(0.1) 0.01<br>10987.1(17.3) 2166.0(17.0) 0.000 |
| (XXX Saga 3-4; (R) (R) (A12) ( | 5688[35.7] 5687[35.7] 0.001 17991.3[33.4] 12582.5[12.4] | 0.091 7781 (24.3) 2037 (21.0) 0.079 0.079 0.079 0.071 0. | 1212 (21.9) 1211 (21.9) 0.001<br>905 (16.4) 905 (16.4) 0.001<br>911 (7.8) 416 (7.9) 0.002<br>108 (2.0) 112 (2.0) 0.005<br>206 (12.8) 220 (13.0) 0.008 | 3244.7 (21.3) 2034.0 (21.0) 0.007<br>3400.2 (6.3) 1000.0 (16.4) 0.007<br>1246.6 (9.2) 790.0 (8.2) 0.001<br>1265.5 (1.8) 198.0 (2.0) 0.022<br>1918.9 (2.26) 1226.0 (12.7) 0.002 | 20512 (21.8) 4275 (24.3) 0.051<br>11178 (27.2) 1848 (24.5) 0.078<br>3922 (5.1) 769 (6.0) 0.002<br>2011 (21.3) 348 (2.7) 0.052<br>0782 (5.2) 1835 (4.4) 0.022 | 2718 (33.6) 14699 (23.4) 0.004<br>1660 (25.1) 1612 (14.8) 0.009<br>636 (5.8) 657 (5.9) 0.007<br>636 (5.6) 109 (2.8) 0.013<br>1652 (64.3) 1599 (14.4) 0.004 | 2121.1 (23.4) 4274.0[14.3] 0.018<br>9274.1[14.8] 1846.0[14.5] 0.008<br>1753.7(5.9) 769.0 (6.0) 0.009<br>1802.4(2.8) 348.0[2.7] 0.007<br>9165.5(14.5) 1834.0[14.4] 0.002 |
| Administracy (N) 2008 (6.1) 3644 (9.4) 0.096 Obstructive siles pagener (n (N) 5429 (4.1) 11356 (9.3) 0.318 Penamonic (N) 391 (6.1) 155 (1.0) 0.044 CKS (Sage 3-2) (N) 230 (9.2) 200 (7.2) 0.044 Acute resul disease (AN) (n (N) 295 (7.7) 1893 (4.9) 0.015 | 1215 (7.4) 1215 (7.4) 0.001 1266 (2.06.6) 3661.3 (9.6.4) 1317 (18.6) 1317 (18.6) 0.001 1317 (18.0) 1312 (19.8) 1314 (19.6) 0.004 1316 (1.1) 1312 (19.8) 1312 (19.8) 1312 (19.8) 1312 (19.8) 1312 (19.8) 1312 (19.8) 1314 (1.1) 1344 (1.1) | 100 | 20.5 | 1076.2 (7.1) 613.0 (6.3) 0.029<br>1232.3 (8.4) 2807.0 (29.0) 0.014<br>562.7 (2.7) 245.0 (2.6) 0.007<br>359.3 (2.4) 225.0 (2.3) 0.002<br>500.4 (2.9) 610.0 (4.2) 0.015 | 2444 [5-3] 251 [5-9] 0.024<br>6796 [10.5] 2320 [8.4) 0.224<br>2133 [4.9] 421 [2.3] 0.079<br>1466 [0.3] 283 [2.2] 0.004<br>6490 [7.9] 925 [6.9] 0.007 | TABLE TABL | |
| Negativatic syndromer, n (N) 0) 0, 0 7 0, 0 0, 004 | (6.0.4) \$1.0.01 0.004 \$2.0.0.0 7.6.0.0 \$1.0.0.0 | 0.004 3(0.0) 1(0.0) 0.007<br>0.044 2061 (13.3) 1045 (16.8) 0.076<br>0.061 8642 (54.4) 5649 (56.4) 0.079<br>0.097 1354 (8.7) 1569 (56.4) 0.03<br>0.099 2346 (15.1) 1556 (15.6) 0.013 | 10.1) 1(0.1) 0.019 501(0.0) 614(11.1) 0.006 1100(56.1) 1120(56.4) 0.006 511(7.3) 538(6.5) 0.009 121(15.0) 847(15.3) 0.008 | 1.8 (0.0) 1.0 (0.0) 0.013<br>1586.8 (0.04) 1043.0 (0.03) 0.012<br>1668.9 (0.05) 1643.0 (0.8.3) 0.026<br>1529.0 (0.00) 926.0 (0.5) 0.016<br>1529.0 (0.00) 926.0 (0.5) 0.016 | 11 (0.0) | 11070 (100.0) 11070 (100.0) 0.001<br>1522 (13.8) 1524 (13.8) 0.001<br>1346 (57.3) 1529 (57.6) 0.006<br>719 (6.5) 707 (6.4) 0.004<br>1848 (6.7) 1820 (16.5) 0.004 | 2.5 [0.0] 1.0 [0.0] 0.005<br>1885.5 (14.0) 1811.0 [14.2] 0.006<br>17940.7 [59.8] 7695.0 [60.4] 0.011<br>4365.9 (6.9) 841.0 [6.6] 0.011<br>107724.1 [6.8] 1.040.0 [16.9] 0.001 |
| DisseastFritt(n) | 364(22.8) 279(23.4) 0.011 3806.8(55.8) (883.0(53.3) 261(27) 0.000 (22.9(7) 55.10,4) 200(11) 551(2.2) 0.000 (22.7(2.3) 1.04.0(5.0) 279(4.5) 279(4.5) 0.001 1551.9(.0) 1557.9(.5) 1557.9(.5) 279(4.5) 279(4.5) 279(4.5) 0.000 (20.0(1.8) (20.0(1.8) 279.0(1.5) | 0.011 2451 [15.8] 15.72 [15.7] 0.002<br>0.019 210(1.4) 14 (1.0) 0.035<br>0.021 430(2.8) 15312.7] 0.072<br>0.097 248(2.2) 14512.5] 0.055<br>0.092 1529 [2.8] 110(12.0) 0.009 | \$12 (15.0) \$60 (15.5) 0.015<br>\$15 (19.9) \$4 (1.0) 0.006<br>\$106 (1.9) \$104 (1.9) 0.003<br>\$2 (1.7) \$7 (1.4) 0.009<br>\$44 (10.0) \$50 (10.0) 0.003 | 2425.7 (2.59) 1537.0 (25.7) 0.007<br>127.0 (0.8) 94.0 (1.0) 0.015<br>297.7 (2.0) 163.0 (1.7) 0.02<br>295.1 (1.3) 144.0 (1.5) 0.022<br>1711.2 (1.12) 1554.0 (1.19) 0.022 | 1231 (15.1) 2545 (20.0) 0.022<br>1041 (1.4) 156 (1.5) 0.004<br>221 (2.3) 15 (2.3) 0.012<br>227 (4.4) 456 (2.3) 0.041<br>608 (2.4) 1263 (0.7) 0.042 | 2179 (9.0.7) 2207 (10.9) 0.006<br>[42 (1.5) 165 (1.5) 0.002<br>20 (9.3) 11 (6.3) 0.002<br>20 (9.3) 425 (1.8) 0.002<br>109 (3.6) 425 (1.8) 0.002<br>1178 (9.6) 1154 (10.4) 0.006 | 12205.2 (20.9) 2545.0 (20.0) 0.021<br>927.6 (1.5) 196.0 (1.5) 0.006<br>174.8 (0.3) 15.0 (0.3) 0.001<br>2245.0 (2.7) 484.0 (1.8) 0.005<br>6922.3 (10.9) 1163.0 (10.7) 0.008 |
| Anoistr, n PS 447 (11.5) 630 (15.5) 0.111 | 2027 13.0 2110 13.2 0.007 1286.1 104.4 (605.0 15.5) (105.0 15.6) (105.0 15.5) (105.0 15.5) (105.0 15.5) (105.0 15.6) (10 | 0.024 1400 (2.0) 1150 (11.9) 0.004<br>0.031 2622 (16.9) 1811 (18.7) 0.048<br>0.011 769 (4.9) 159 (1.6) 0.114<br>0.002 266 (1.7) 15 (2.5) 0.114<br>0.002 160 (1.7) 15 (2.5) 0.114<br>0.004 165 (2.3) 160 (2.6) 0.115 | 581 (0.5) 562 (0.02) 0.011<br>571 (17.5) 578 (17.7) 0.003<br>507 (1.9) 116 (7.1) 0.012<br>42 (0.8) 42 (0.8) 0.001<br>22744.31 2.004.31 0.002 | 172.4.(1.1.3) 11.47.0(11.9) 0.017<br>2891.2 (19.0) 1807.0 (18.7) 0.008<br>251.7 (1.7) 158.0 (1.8) 0.001<br>80.6(9.5) 51.0 (9.5) 0.001<br>887.0 (5.8) 590.06.21 0.016 | 6657(7.2) 935 (7.3) 0.004<br>10219 (18.8) 2410 (18.9) 0.001<br>2992 (8.2) 344 (2.7) 0.17<br>1181 (1.8) 101 (0.8) 0.091<br>266 (9.4) 990.51 0.023 | 828 (7.5) 812 (7.3) 0.006<br>828 (7.5) 10.78 (18.8) 0.004<br>288 (3.1) 222 (2.9) 0.009<br>103 (0.9) 96 (0.9) 0.007<br>78 (0.7) 68 (0.6) 0.011 | 8667.1 (7.4) 925.0 (7.3) 0.001<br>1468.6 (19.7) 1400.0 (12.9) 0.019<br>1764.8 (2.8) 144.0 (2.7) 0.005<br>674.8 (0.7) 101.0 (9.8) 0.005<br>1774.0 (64) 79.0 (64) 0.003 |
| Number of antidiabetic drugs meso (of) 1.15 (0.81) 1.10 (0.87) 0.055 tesuffer, or (h) 660 (11.77) 5794 (0.75) Melgistrader, or (h) 127 (0.6) 228 (0.6) 0.044 (0.5) 4.6 (0.75) 0.051 (0.75) 0.051 (0.75) 0.051 (0.5) 4.6 (0.75) 0.051 (0.75) 0.051 (0.75) 0.051 | WILLIAM WILL | | | 1.24(0.86) 1.20(0.80) 0.028<br>4754.8(0.12) 2962.0(03.7) 0.011<br>74.5(0.5) 47.0(0.5) 0.001<br>3411.9(0.74) 2931.0(0.90) 0.036 | YEAR | | 1.27 (0.85) 1.27 (0.86) 0.001<br>26072.6 [41.1] 5291.0 [41.5] 0.008<br>786.6 [1.2] 153.0 [1.2] 0.004 |
| Methors: pt 10 2009 [6.3] 2009 [6.3] 2018 [6.1] 0.038 Methors: pt 10 0.038 Methors: pt 10 0.038 Methods: pt 10 0.038 Methods: pt 10 0.012 Methods: pt 10 0.012 Methods: pt 10 0.012 Methods: pt 10 0.038 Methods | 892 26-52 8892 55-77 0.000 71805 25-65 71805 26-65 1283 26-15 1285 26-65 1283 26-15 1285 26-65 1283 26-15 1285 26-65 1285 26-15 1285 | | REAR | 929.1.5 (61.0) 5850.0 (60.5) 0.01<br>788.2 (5.2) 427.0 (6.5) 0.021<br>4887.2 (8.2) 549.0 (24.4) 0.055<br>23.4 (0.2) 15.0 (6.2) 0.001 | 36204 (56.3) 7231 (57.4) 0.024<br>2643 (5.7) 811 (6.4) 0.021<br>4117 (6.4) 1032 (55.2) 0.364<br>229 (5.4) 28 (5.2) 0.028 | TABLE | 16788.1 (58.0) 7311.0 (57.4) 0.013<br>4177.4 (6.5) 813.0 (5.4) 0.005<br>9966 2 (5.7) (933.0 (15.2) 0.015<br>157.1 (6.2) 28.0 (0.2) 0.006 |
| 1786 | 1227/1962 1227/1963 0.000 1227/1963 12 | 0.0007 (2012) (2 | 1541 (27.9) 1558 (28.2) 0.005<br>1541 (27.9) 1558 (28.2) 0.006<br>1445 (56.8) 1192 (57.7) 0.017<br>1577 (10.3) 157 (21.7) 0.021<br>1048 (18.9) 1045 (18.9) 0.001 | 1205 - (1905 - 1) | 1800 (2.0.9) 1770 (9.6.) 0.054<br>1803 (2.0.9) 1770 (9.6.) 0.054<br>39945 (6.1.9) 2851 (61.6.) 0.011<br>24050 (27.3) 4388 (24.4) 0.054<br>16987 (6.4) 3652 (9.7) 0.051 | 0.0002 0 | 1877.7.9 (27.5.9) 1888.0 (17.7.7) 0.0000<br>1877.7.9 (27.5.) 1770.0 (27.6.5) 0.002<br>18815.7 (61.2.) 7855.0 (61.6.5) 0.003<br>12020.2 (24.6.) 4186.0 (24.4.4) 0.003<br>18286.4 (28.8.) 1652.0 (28.7) 0.004 |
| User Guerrico, n.p.j. 2007/17 4881(1.1.1) 0.124. Whenex, n.p.j. 2007/17 2007/17 4881(1.1.1) 0.124. Whenex, n.p.j. 3007/18 2007/18 2007 | 1499 143 1497 1 | 0.0014 1.000 [8.8] 1000 [3.1.4] 0.0005<br>0.001 1777 [11.1] 1009 [11.3] 0.005<br>0.007 562 [6.6] 417 [6.3] 0.005<br>0.001 460 [1.0] 275 [2.8] 0.007<br>0.001 3417 [22.0] 342 [25.0] 0.007 | 394 [10.2] 344 [10.2] 0.001<br>[991[0.3] 611 [1.10] 0.007<br>202[2.7] 215 [2.5] 0.011<br>[146[2.6] 147 [2.7] 0.001<br>[127 [23.1] 128 [23.1] 0.002 | 1792.4 (§1.4) 1097.0 (§1.4) 0.0001<br>1792.4 (§1.8) 1090.0 (§1.3) 0.016<br>130.4 (4.1) 417.0 (4.3) 0.000<br>1463.2 (2.4) 275.0 (2.8) 0.002<br>1793.2 (2.4) 275.0 (2.8) 0.002 | 1244 (U.S) | 1000 (0.99) 1100 (0.91) 0.3002<br>1392 (2.6) 1393 (12.6) 0.001<br>389 (3.5) 404 (3.6) 0.007<br>374 (3.4) 172 (3.4) 0.001<br>2992 (27.0) 3943 (36.6) 0.01 | \$137.5(1.8) \$159.0(12.9) 0.000<br>\$137.5(1.8) \$159.0(12.9) 0.001<br>\$228.4(1.6) \$469.0(1.7) 0.004<br>\$209.4(1.3) 426.0(1.3) 0.002<br>\$1706.0(1.8) \$406.0(1.7) 0.004 |
| Stating in (b) 2044 (79.1) 2009 (80.0) 0.021 Other typic-flowwring drugs in (b) 4138 (10.7) 5.239 (11.7) 0.002 Antigitatiet agent's in (b) 4009 (17.2) 0.756 (17.4) 0.006 Other stationage lasting in (b) 5122 (11.8) 5438 (14.5) 0.018 Other stationage lasting in (b) 5122 (11.8) 5438 (14.5) 0.018 Other stationage lasting in (b) 5122 (11.8) 5122 (11.8) 0.008 Other stationage lasting in (b) 5122 (11.8) 0.009 (11.8) Other stationage lasting in (b) 5122 (11.8) 0.009 (11.8) Other stationage lasting in (b) 5122 (11.8) 0.009 (11.8) Other stationage lasting in (b) 5122 (11.8) Other stationage lasting in (b) 5122 (11.8) Other stationage lasting in (b) 5122 (11.8) Other stationage lasting in (b) 5122 (11.8) Other stationage lasting in (b) Other sta | 1340 [85.1] 1776 [86.0] 0.805 11177 [81.2] 11076 [86.0] 0.805 11177 [81.2] 11076 [86.0] 0.805 11177 [81.2] 11076 [86.0] 0.805 11177 [81.2] 0.805 [81 | 0.021 1417 22.28 9421 25.48 0.071 0.001 0.00 | 4302 (77.8) 4332 (78.3) 0.011<br>900 (14.45) 297 (14.4) 0.006<br>1319 (23.8) 1322 (23.9) 0.001<br>646 (13.7) 657 (13.9) 0.006<br>9031 (18.6) 1041 (18.8) 0.005 | 1201.4(78.9) 7582.2(78.4) 0.011<br>2315.4(5.2) 1540.0(15.9) 0.02<br>1615.8(23.9) 2346.0(24.3) 0.009<br>1803.1(11.8) 1207.0(12.5) 0.02<br>2977.0(9.6) 1905.0(19.7) 0.004 | 50545 (78.4) 10327 (81.1) 0.667<br>7931 (12.2) 1885 (84.8) 0.072<br>12727 (10.7) 2565 (0.4) 0.015<br>11084 (17.2) 2000 (6.5) 0.019<br>11155 (17.4) 2351 (84.4) 0.028 | 8647(91.0) 8914 (80.5) 0.012<br>1556 (34.4) 1544 (14.3) 0.002<br>2351 (20.3) 2211 (20.0) 0.009<br>1778 (36.1) 1794 (36.2) 0.004<br>2005 (8.7) 2002 (18.6) 0.003 | \$1372.0 (81.5) 10336.0 (81.1) 0.002<br>9136.4 (14.4) 1815.0 (14.8) 0.011<br>12864.7 (30.3) 2594.0 (20.4) 0.002<br>1035.7 (16.3) 2090.0 (16.5) 0.004<br>12166.8 (19.3) 2351.0 (18.4) 0.019 |
| Onicerticosteratide, n (N) 4451 (12.9) CB37 (E.4.) 0.160 Inigerosphenistic, n (N) 1200 (2.1) 800 (2.1) 0.064 Opinide, n (N) 2318 (21.3) 986 (25.5) 0.064 Anti-degreeast, n (N) 15648 (27.7) 14458 (97.2) 0.201 Chapperisonic in (N) 7794 (02.2) 0.931 (5.9) 0.111 | 2146(12.5) 2147(23.7) 0.004 5246.9 (E.4) 6343.0 (E.6.) (1342.6) (1 | 0.001 2127 [13.8] 1465 [15.1] 0.039<br>0.006 225 [1.5] 75 [3.8] 0.009<br>0.03 2957 [19.0] 3004 [20.7] 0.042<br>0.049 3655 [23.5] 1127 [22.3] 0.197<br>0.049 272 [14.6] 1729 [18.1] 0.004 | 102 (14.5) 715 (14.2) 0.009 | 239.2 (5.7) 1462.0 (5.1) 0.016<br>116.7 (0.8) 75.0 (0.8) 0.006<br>1284.2 (0.16) 1099.0 (20.7) 0.022<br>5040.4 (0.11) 1116.0 (02.7) 0.029<br>1274.8 (18.0) 1744.0 (18.0) 0.002 | 5007 (14.0) 1726 (13.6) 0.01<br>1894 (2.9) 246 (1.9) 0.055<br>1435 (22.3) 3157 (24.8) 0.059<br>1817 (28.1) 4260 (24.4) 0.127<br>11791 (18.3) 200 (22.8) 0.111 | 1524 (0.3.8) 1518 (13.7) 0.0021<br>208 (1.9) 222 (2.0) 0.009<br>2621 (02.7) 1698 (04.4) 0.016<br>3720 (03.6) 3732 (03.7) 0.002<br>2425 (21.6) 2415 (21.8) 0.002 | \$789.8 (12.9) 1735.0 (13.6) 0.007<br>1275.2 (2.00) 246.0 (1.9) 0.006<br>16086.5 (25.4) 1357.0 (24.8) 0.014<br>22349.2 (25.2) 4290.0 (24.4) 0.017<br>16437.4 (23.1) 9090.0 (22.8) 0.007 |
| Beroxofiaepiser, c (S) | \$151.09.5 \$151.09.5 \$0.000 \$190.0 (2.08) \$1.210.0 (2.08) | 001 997 (92.9) 2094 (92.7) 0.042<br>0.046 501 (92.3) 1127 (22.3) 0.172<br>0.046 227 (14.4) 1746 (14.1) 0.064<br>1277 (14.4) 1746 (14.1) 0.064<br>0.001 1398 (4.) 1898 (7.) 0.044<br>0.046 278 (4.) 178 (6.) 0.066<br>0.047 (14.) 178 (6.) 0.066<br>0.041 189 (14.) 116 (14.) 0.064<br>0.044 118 (14.) 0.064<br>1.07 (14.) 0.064<br>1.07 | 355 [2.1] 457 [6.0] 0.005<br>356 [7.2] 401 [7.1] 0.005<br>[44 [1.2] 50 [1.1] 0.007<br>150 [1.97] 0.004 | 5000.4 (33.1) 3115.0 (32.2) 0.019<br>2734.6 (31.00) 1744.0 (31.0) 0.002<br>1515.2 (30.0) 95.0 (9.7) 0.009<br>1245.3 (9.7) 774.0 (8.0) 0.006<br>202.3 (2.1) 95.0 (9.9) 0.027<br>1.68 (1.87) 1.67 (3.87) 0.007 | 0945 [10.8] 1338 [10.5] 0.003<br>2894 [6.0] 227 [7.4] 0.052<br>2898 [6.4] 225 [7.4] 0.141<br>280 [6.4] 235 [7.4] 0.141 | 1332 (11.1) 1181 (10.7) 0.015<br>818 (7.4) 110 (7.3) 0.001<br>302 (2.7) 308 (2.8) 0.001<br>10 (2.7) 10 (2.8) 0.001 | 5795.9(10.7) 1238.0(10.5) 0.007<br>4748.8(7.5) 927.0(7.4) 0.005<br>1748.9(2.6) 125.0(2.6) 0.001<br>1549.9(2.6) 125.0(2.6) 0.001 |
| Farally score | 0.17 (0.65) | 0.065 0.17 (0.04) 0.16 (0.04) 0.175 | 0.16 (0.04) 0.16 (0.04) 0.015 | 0.16 (0.04) 0.16 (0.04) 0.005<br>12.21 (5.51) 12.12 (5.23) 0.017 | 0.20 (5.06) 0.20 (3.05) 0.081<br>11.32 (4.74) 12.20 (4.83) 0.204 | 0.20 (0.05) 0.39 (0.05) 0.015 | 0.20 (0.05) 0.20 (0.05) 0.021<br>12.38 (5.01) 12.30 (4.87) 0.018 |
| 11.75 (5.11) 12.75 (5.51) 0.185 | 100 pt 1 | 0.002 10.88 (6.81) 12.14 (5.25) 0.349<br>0.003 11.00 (6.91) 12.26 (5.34) 0.345<br>0.001 1190 (77) 400 (4.1) 0.323<br>0.001 190 (77) 400 (4.1) 0.323<br>0.004 (535 (9.2) 3566 (5.58) 0.024 | 11.37 (5.14) 11.52 (6.97) 0.029<br>11.49 (5.24) 11.64 (5.07) 0.029<br>265 (4.8) 272 (6.9) 0.005<br>127 (8.9) 0.005<br>127 (8.9) 0.005<br>128 (5.77) 1471 (6.6) 0.021 | 12.35 (5.63) 12.25 (5.32) 0.016<br>673.6 (4.4) 600.0 (4.1) 0.014<br>1507.0 (9.9) 917.0 (9.5) 0.014<br>1599.1 (26.3) 2501.0 (25.9) 0.009 | 11.32 (4.74) 12.30 (4.31) 0.204<br>11.42 (4.32) 12.44 (4.35) 0.205<br>(2209 (4) 154 (4.35) 0.205<br>(2209 (4) 154 (4.35) 0.327<br>(2417 (4.4) 12.77 (0.05) 0.347<br>15116 (25.7) 1502 (27.25) 0.333 | 12.08 (4.94) 12.05 (4.36) 0.006<br>12.22 (5.05) 12.19 (4.86) 0.007<br>148 (5.3) 469 (5.0) 0.024<br>1186 (0.04) 1122 (0.03) 0.007<br>124 (7.64) 2.066 (24.1) 0.027 | 12.53 (5.12) 12.44 (4.95) 0.018<br>1034.1 (6.8) 586.0 (4.6) 0.009<br>5590 (10.3) 1272.0 (10.0) 0.012<br>15328.6 (24.2) 1027.0 (23.8) 0.01 |
| Uniforwards | \$\frac{13\pi_122}{14\pi_122}\$\$ \$\frac{1}{3}\pi_1231\$\$ \$\frac{1}{3}\p | 0.059 | 5.59 (4.18) 5.65 (4.10) 0.012<br>966 (15.6) 860 (15.5) 0.002<br>2868 (50.7) 2822 (51.2) 0.009<br>4578 (4.5) 4697 (84.0) 0.02 | 6.07 (4.75) 6.02 (4.46) 0.000<br>3319.5 (31.8) 2125.0 (32.0) 0.004<br>8002.5 (53.0) 5152.0 (53.3) 0.007<br>12593.8 (82.7) 8005.0 (82.8) 0.002 | 6.54(7.57) 7.22(7.10) 0.002<br>782(72,2) 1.068(7.4) 0.389<br>715(72,2) 1.068(7.4) 0.389<br>715(72,66.5) 1.544(86.2) 0.064<br>54012(83.8) 1.0245(80.4) 0.069<br>1.02(7.31) 0.36(1.58) 0.063 | 7.14 (8.04) 7.05 (8.94) 0.011<br>2484 (9.24) 15.20 (2.31) 0.008<br>1378 (86.0) 15.00 (48.0) 0.002<br>1096 (81.3) 6095 (80.3) 0.011<br>2.80 (1.65) 0.66 (1.61) 0.014 | 7.34 (8.17) 7.22 (7.10) 0.015<br>16313.8 (25.7) 4486.0 (27.4) 0.037<br>30778.4 (86.2) 4144.0 (48.2) 0.001<br>51079.8 (80.5) 10344.0 (80.4) 0.004 |
| | 0.32 (0.51) 0.22 (0.52) 0.001 0.24 (0.52) 0.24 (0.60) | 0.028 1.31(2.96) 1.09(2.07) 0.066<br>0.002 0.58(2.14) 2.46(1.37) 0.068 | 1.10 (2.16) 1.10 (2.19) 0.001<br>0.46 (1.40) 0.46 (1.40) 0.003 | 1.08 (2.00) 1.09 (2.07) 0.003<br>0.45 (1.39) 0.46 (1.37) 0.007 | 0.32 (1.12) 0.27 (0.69) 0.049 | 0.28 (0.74) 0.27 (0.69) 0.01 | 0.88 (1.70) 0.86 (1.58) 0.015<br>0.28 (0.86) 0.27 (0.69) 0.008 |
| mean (ul) | 1.42 (0.12) | 0.054 1.39(1.12) 1.38(1.01) 0.381<br>0.049 0.45(1.42) 0.50(1.85) 0.031<br>0.001 0.85(0.94) 0.99(0.97) 0.139 | 1.34 (1.12) | 1.40(0.99) 1.38(1.01) 0.021<br>0.50(1.21) 0.50(1.85) 0.001<br>1.00(0.92) 0.88(0.96) 0.015 | 1.52 (1.37) 1.62 (1.27) 0.687<br>0.61 (2.27) 0.67 (2.82) 0.02<br>1.05 (1.21) 1.10 (1.14) 0.045 | 1.59 (1.72) | 1.65 (2.25) 1.63 (1.27) 0.013<br>0.65 (2.82) 0.67 (2.82) 0.007<br>1.12 (2.06) 1.10 (1.14) 0.014 |
| Creations set ordered | 1.45 2.45 | 0.005 0.006 0.008.331 0.008.231 0.002 0.005 0.005 1190.213 0.002 0.005 0 | 0.03 (0.22) 0.03 (0.24) 0.003<br>120(2.2) 123 (2.2) 0.004<br>6456 (01.2) 6454 (02.1) 0.002<br>583 (10.5) 500 (10.5) 0.002 | 0.02 (0.21) 0.02 (0.21) 0.018<br>316.4 (0.1) 223.0 (2.4) 0.022<br>12712.7 (0.82) 0017.0 (0.23) 0.015<br>176.9 (1.16) 1125.0 (11.6) 0.001 | TOTAL TOTA | 0.5 (0.33) 0.55 (0.31) 0.008<br>45 (4.2) 0.004.5) 0.015<br>45 (4.2) 0.004.5) 0.015<br>1235 (1.3) 1245 (11.2) 0.007<br>1235 (1.3) 1245 (11.2) 0.007<br>1145 (0.54) 1138 (0.54) 0.001 | 0.05 (0.31) 0.05 (0.31) 0.005<br>2010-2(6.6) 572.0 (6.5) 0.005<br>5726-6 (90.4) 11455.0 (90.5) 0.016<br>7412-2 (1.77) (446-5 (01.3) 0.011 |
| Pop smear; n (N) 2565 (E.S.) 2364 (ELS) 0.334 (ELS) 0.334 (ELS) 0.334 (ELS) 0.334 (ELS) 0.334 (ELS) 0.334 (ELS) 0.334 (ELS) 0.344 (ELS) 0. | 1855 (1.7) | 0.006 1186 [7.6] 1057 [10.6] 0.116<br>0.024 259 [16.7] 1741 [18.6] 0.036<br>0.022 745 [4.8] 772 [5.9] 0.05<br>0.001 1846 [22.3] 1854 [19.2] 0.079 | 346 (9.3) 338 (9.7) 0.005<br>3050 (9.6) 3041 (18.8) 0.004<br>287 (5.2) 290 (6.2) 0.002<br>296 (19.8) 111,120,11 0.008 | 1667.5 (11.0) 1054.0 (10.0) 0.000<br>2784.5 (18.3) 1728.0 (18.0) 0.000<br>866.7 (5.7) 572.0 (5.9) 0.01<br>3882.1 (18.9) 1850.0 (19.1) 0.004 | 555 (8.6) 1280 (8.6) 0.079<br>990 (14.7) 217 (9.70) 0.661<br>2844 (8.4) 703 (5.5) 0.051<br>2560 (9.8) 5279 (4.4) 0.031 | | 7155.0 (11.3) 1390.0 (11.0) 0.01<br>10666-3 (16.8) 2273.0 (17.0) 0.006<br>2574.6 (5.6) 703.0 (5.5) 0.006<br>2574.6 (5.6) 703.0 (5.5) 0.006 |
| Telemodicine n [%] 1439 (11.4) C556 (17.5) 0.555 Heart follow's Ph 1459 (11.4) C556 (17.5) 0.555 Heart follow's Ph 1570 (2.8) 0.575 (15.1) 0.056 History Ph 1570 (2.8) 0.057 (15.1) 0.056 History Ph 1570 (2.8) 0.057 (15.1) 0.057 (15.1) History Ph 1570 (2.8) History Ph 1570 | 2518 1518 2472 1515 0.008 4272 1(7.3) (550-0)(4.5) (472 1(7.3) (550-0)(4.5) (472 1(7.3) (550-0)(4.5) (472 1(7.3) (550-0)(4.5) (472 1(7.3) (550-0)(4.5) (472 1(7.3) (472)1(7.3) (472)1(7. | 0.011 4665 (27.2) (354 (19.2) 0.079 0.000 0.000 0.001 114 (57.2) 0.279 0.002 | 056 (19.8) 1112/0.1) 0.008<br>104 (19.7) 101 (18.3) 0.011<br>884 (17.8) 1007 (18.2) 0.011<br>179 (12.2) 185 (2.3) 0.001<br>179 (12.2) 185 (2.3) 0.001<br>179 (14.3) 115 (2.6) 0.012 | 266.1 (2.6) 166.0 (2.6) 0.001<br>266.1 (2.6) 2.6 (2.6) 0.001<br>264.1 (2.9) 1862.0 (9.3) 0.002<br>50.2 (2.3) 239 (2.3) 0.003<br>566.1 (2.6) 248.0 (2.6) 0.001 | 4479(5.9) 1907 (5.7) 0.279<br>15635 (24.3) 2963 (23.2) 0.224<br>2237 (24.5) 256 (24.5) 0.05<br>2655 (4.3) 596 (4.7) 0.03 | 196 (E.4) (1995.3) 0.022 (1918.40 (1995.3) 0.022 (1918.40 (1995.3) 0.022 (1918.40 (1995.3) 0.022 (1918.40 (1995.3) 0.022 (1918.40 (1995.3) 0.025 (1918 | 9803.0 (15.5) 1997.0 (15.7) 0.006<br>14868.9 (23.4) 2962.0 (23.2) 0.005<br>1695.5 (2.6) 22.60 (2.6) 0.003<br>3073.1 (4.8) 594.0 (4.7) 0.000 |
| White, e (K) #### (K) #### (K) #### (K) #### (K) ##### (K) ###### (K) ################################### | | | | | 49566 (76.5) 10742 (94.3) 0.229<br>2847 [4.4] 229 (1.3) 6040 (10.2) 55 (7.5) 2344 [4.4] 199 (1.4) 199 (1.4) 1227 [5.1] 199 (1.4) 199 (1.4) 1227 [5.1] 199 (1.4) | 2272 (0.3.8) 9250 (0.3.6) 0.002 / 223 (0.3.8) 9250 (0.3.6) 0.002 / 223 (0.3) 219 (2.0) 840 (7.6) 160 (7.6) 160 (7.9) 206 (1.9) 190 (1.7) 226 (1.9) 190 (1.7) 126 (4.8) (4.2) 640 (1.9) 190 (1.7) 126 (4.8) (4.2) 640 (1.9) 190 (1.7) 126 (4.8) (4.2) 640 (1.9) 190 (1.7) 126 (4.8) (4.2) 640 (1.9) 190 (1.7) 126 (4.8) (4.2) 640 (1.9) 190 (1.7) 126 (4.8) (4.2) 190 (1.7) 126 (4.8) (4.2) (4.2) (4. | 52526.3 (84.4) (0742.0 (84.3) (1141.1 (1.8) (250.0 (1.8) (141.1 (1.8) (250.0 (1.8) (141.1 (1.8) (1.9) |
| Uniform research (Control (N)) Out of datas for med care is (N) | | | | | 16896 (26.2) 2248 (37.6) 0.208 | 2000 (18.6) 2044 (18.5) 0.004 | 11364.4 (17.9) 921.0 (4.9) 0.008 |

| Covariates | Source |
|---|---|
| Region | If region not available, from State, https://www2.census.gov/geo/pdfs/maps-data/maps/reference/us_regdiv.pdf |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://hcup- |
| | us.ahrq.gov/datainnovations/ICD-10CaseStudyonOpioid-RelatedIPStays042417.pdf, |
| Drug abuse or dependence | https://stacks.cdc.gov/view/cdc/59394, https://pubmed.ncbi.nlm.nih.gov/34134872/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, |
| | https://espace.curtin.edu.au/bitstream/handle/20.500.11937/34117/19233_downloaded_stream_325.pdf?isAllo |
| Alcohol abuse or dependence | wed=y&sequence=2 |
| Underweight or normal weight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Overweight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Severe Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Unspecified obesity | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| | Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_mpl2p_wp015, |
| | https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_sir_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, |
| Smoking | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/ |
| 50 L 10 L 10 L 10 L | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| Diabetic retinopathy | https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Dishatia na una sastiu. | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| Diabetic neuropathy | https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Diabetic nephropathy | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| | https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference- |
| Disheta with was sifted as 10 mg | Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-279/249- |
| Diabetes with unspecified complication | 259/250/default.htm, https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetes with other ophthalmic manifestations | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion |
| | Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, |
| | https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus, |
| Disheter with peripheral size-ulate and dis-ulate- | http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm, |
| Diabetes with peripheral circulatory disorders | https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetic foot + Lower extremity amputation | Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/ |
| Skin infections | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion |
| | Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, |
| Fractile durfunction | https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-, |
| Erectile dysfunction | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/ |
| Hynoglycemia | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Hypoglycemia | IICCho://haniiiea:ucn:uiiii:liiii:80x/22042102/ |

Hyperglycemia, DKA, HONK

Hypertension

Hyperlipidemia

Atrial fibrillation
Acute MI
Old MI
Coronary atherosclerosis
History of CABG/PTCA
Previous cardiac procedure
Cerebrovascular procedure
Ischemic stroke
PVD diagnosis or surgery
CKD stage 3-4

Other cardiac dysrhythmia

Cardiomyopathy

Valve disorders COPD

Asthma

Obstructive sleep apnea

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/HONK: https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovation/DEF/DKA.pdf

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4910677/

algorithm (any care setting, any diagnosis position)

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

 $https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconcepts cardiology 1.pdf, ICD9\ to\ ICD10\ conversion$ 

 $Investigator\ review\ of\ codes\ based\ on:\ https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at=refs\%2Fheads\%2Fcder\_mpl2p\_wp015$ 

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp009 Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

Pneumonia Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/ CKD 1-2 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Acute renal disease (AKI) Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, Nephrotic syndrome https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode-cms/fullcode cms/P2401.html Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-Hypertensive nephropathy 9af3-81bd071bbc67/mmc1.pdf, https://www.icd10data.com/ICD10CM/Codes/I00-I99 Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637. https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion Other renal conditions https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinelanalytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, Modified algorightm from Liver disease https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm Modified CCW algorithm Hypothyroidism Osteoarthritis Modified CCW algorithm https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder mpl2p wp009 Fractures https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, Falls https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp010 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Osteoporosis packages/browse?at=refs%2Fheads%2Fcder sir wp002, CCW Algorithms Depression https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms https://pubmed.ncbi.nlm.nih.gov/35043165/ Anxiety Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-diagnostic-codes-Sleep disorder 3014779 https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Dementia packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015 Delirium https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/ COVID https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/ Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5256065/, https://www.drugs.com/drug-class/antidiabetic-Number of antidiabetic drugs agents.html, https://www.ncbi.nlm.nih.gov/books/NBK279141/ Investigator review of codes based on: https://www.drugs.com, ACE + ARBs https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Thiazide

Investigator review of codes based on: https://www.drugs.com, Beta blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Calcium channel blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Loop diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Other diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Nitrates https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ HF drugs (Digoxin + Entresto + Ivabadrine) Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is beta blockers and class 4 is Anti-arrhythmics calcium channel blockers) Investigator review of codes based on: https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-COPD/asthma meds COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medications-list.aspx Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-Statins topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-Other lipid-lowering drugs topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/ Antiplatelet agents Investigator review of codes based on: https://www.drugs.com, https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559 Oral anticoagulants Investigator review of codes based on: https://www.drugs.com, **NSAIDs** https://www.ncbi.nlm.nih.gov/books/NBK547742/ Investigator review of codes based on: https://www.drugs.com, https://www.aaaai.org/tools-for-the-public/drug-Oral corticosteroids guide/oral-corticosteroid-medications Investigator review of codes based on: https://www.drugs.com, **Bisphosphonates** https://www.ncbi.nlm.nih.gov/books/NBK470248/ Investigator review of codes based on: https://www.drugs.com, https://pubmed.ncbi.nlm.nih.gov/31643200/#:~:text=They%20can%20also%20be%20informally,%2C%20codeine Opioids %2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes based on: https://www.drugs.com, Anti-depressants https://www.ncbi.nlm.nih.gov/books/NBK538182/ Gabapentnoids GABAPENTIN, PREGABALIN Investigator review of codes based on: https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf, https://www.ncbi.nlm.nih.gov/books/NBK470159/ Benzodiazepines Investigator review of codes based on: https://www.drugs.com Anxiolytics/hypnotics Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/, https://go.drugbank.com/drugs/DB00382

Dementia meds

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visitcomplexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-Office visits officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-**Endocrinologist visit** enrollment-and-certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-Cardiologist visits enrollment-and-certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Internal medicine/family medicine visits Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleId=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-ecg-coding-Electrocardiograms questions-175952-article Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/, https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56625&ver=27&, https://www.medicalbillgurus.com/echocardiogram-cpt-Echocardio code/ HbA1c tests received Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Glucose tests ordered Lipid tests ordered Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Creatinine tests ordered Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=59040&ver=4, https://static.cigna.com/assets/chcp/pdf/coveragePolicies/medical/mm 0300 coveragepositioncriteria bone min Bone mineral density test eral density measurement.pdf Basic or comprehensive metabolic blood chem test Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56448&ver=16&bc=0, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm Mammogram Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-Pap smear V82/V72/default.htm, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-PSA packages/browse?at=refs%2Fheads%2Fcder sir wp002 Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy packages/browse?at=refs%2Fheads%2Fcder sir wp002 Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767

Investigator review of codes, Flu vaccine/Pnemococcal vaccine

Telemedicine
Heart failure
TIA
Ankle-brachial index<0.9
Microalbuminuria/proteinuria

DUAL status for medicare ED visit (Medicare) ED visit (Optum)

ED visit (Marketscan)
Hernia (negative control)
Lumbar radiculopathy (negative control)

Cataract surgery (negative control)

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/,

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-fact-sheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-telehealth-audio-virtual-digital-visits.html

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Investigator review of codes based on: https://www.cms.gov/medicare-medicaid-coordination/medicare-and-medicaid-coordination/medicare-medicaid-coordination/medicare-medicaid-coordination-gff Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service: 23

Place of service: 23

Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23

https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s

https://pubmed.ncbi.nlm.nih.gov/32828874/, https://pubmed.ncbi.nlm.nih.gov/29433851/, https://pubmed.ncbi.nlm.nih.gov/29075781/, https://pubmed.ncbi.nlm.nih.gov/34935591/ and https://pubmed.ncbi.nlm.nih.gov/23993357/ and department ICD-9 to ICD-10 conversion


| AT LEAST ONE OF THE FOLLOWING: | A CURRENT TOBACCO USER OUSER AND RECEIVED TOBACCO CESSATION INTERVENTION (MUST INCLUDE ADVICE GIVEN TO QUIT SMOKING OR TOBACCO USE, COUNSELING ON THE IN TOBACCO USE, ASSISTANCE WITH OR REFERRAL TO EXTERNAL SMOKING OR DGRAMS, OR CURRENT ENROLLMENT IN SMOKING OR TOBACCO USE |
|---|---|
| AT LEAST ONE OF THE FOLLOWING: | ADVICE GIVEN TO QUIT SMOKING OR TOBACCO USE, COUNSELING ON THE<br>OR TOBACCO USE, ASSISTANCE WITH OR REFERRAL TO EXTERNAL SMOKING OR |
| Diabetic retinopathy 379.23 DX 09 VITREOUS HEMORRHAGE | |
| Diabetic retinopathy 362 DX 09 DIABETIC RETINOPATHY | |
| Diabetic retinopathy 362.01 DX 09 BACKGROUND DIABETIC RETINOPAT | тнү |
| Diabetic retinopathy 362.02 DX 09 PROLIFERATIVE DIABETIC RETINOPA | ATHY |
| Diabetic retinopathy 362.03 DX 09 NONPROLIFERATIVE DIABETIC RETIN | NOPATHY NOS |
| Diabetic retinopathy 362.04 DX 09 MILD NONPROLIFERATIVE DIABETIC | CRETINOPATHY |
| Diabetic retinopathy 362.05 DX 09 MODERATE NONPROLIFERATIVE DIA | ABETIC RETINOPATHY |
| Diabetic retinopathy 362.06 DX 09 SEVERE NONPROLIFERATIVE DIABET | |
| Diabetic retinopathy 362.07 DX 09 DIABETIC MACULAR EDEMA | |
| Diabetic retinopathy E10.3 DX 10 TYPE 1 DIABETES MELLITUS WITH OF | PHTHALMIC COMPLICATIONS |
| ··· | INSPECIFIED DIABETIC RETINOPATHY |
| , , | INSPECIFIED DIABETIC RETINOPATHY WITH MACULAR EDEMA |
| , , | INSPECIFIED DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA |
| | MILD NONPROLIFERATIVE DIABETIC RETINOPATHY |
| | ALLD NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR EDEMA |
| | MILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR EDEMA, |
| Diabetic retinopathy E10.3212 DX 10 TYPE 1 DIABETES MELLITUS WITH M EYE | MILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR EDEMA, LEFT |
| Diabetic retinopathy E10.3213 DX 10 TYPE 1 DIABETES MELLITUS WITH M<br>BILATERAL | IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR EDEMA, |
| UNSPECIFIED EYE | IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR EDEMA, |
| | IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA |
| RIGHTEYE | IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA, |
| LEFT EYE | MILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA, |
| BILATERAL | IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA, IILD NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR EDEMA, |
| UNSPECIFIED EYE | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY |
| , , | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR |
| Diabetic retinipatity £10.531 DA 10 HTF2 DIABETES WIELTHOS WITH WI | NODERATE NONPROLIFERATIVE DIABETIC RETINOPATHT WITH WACCLAR |
| | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR |
| Diabetic retinopathy E10.3312 DX 10 TYPE 1 DIABETES MELLITUS WITH M EDEMA, LEFT EYE | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR |
| Diabetic retinopathy E10.3313 DX 10 TYPE 1 DIABETES MELLITUS WITH M EDEMA, BILATERAL | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR |
| Diabetic retinopathy E10.3319 DX 10 TYPE 1 DIABETES MELLITUS WITH M EDEMA, UNSPECIFIED EYE | 10DERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITH MACULAR |
| EDEMA | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR |
| EDEMA, RIGHT EYE | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR |
| EDEMA, LEFT EYE | MODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR |
| Diabetic retinopathy E10.3393 DX 10 TYPE 1 DIABETES MELLITUS WITH M EDEMA, BILATERAL | ODERATE NONPROLIFERATIVE DIABETIC RETINOPATHY WITHOUT MACULAR |


| Professic cardiac gronodum (CARS, PTCA, Sent) 271466 PX 10 DILATION DE CORONAM PATTERS, TWO ARTERES, MERIZACITION, WITH YOU DIREALUMINAL DEVICES, PERCUTANEOUS PROFESSION CARRIER STREET, SAME PARTIES, SAME PARTIES, SAME | Previous cardiac procedure (CABG, PTCA, Stent) | 02714DZ | PX | 10 | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH |
|---|---|---|---|---|---|
| Pervious cardius procedure (CAGG, PTC, Stert) O2714F7 PX 10 DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH THREE RITRICUMANAL DEVICES, PERCUTANEOUS BIOLOGOPIC APPROACH DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH THREE RITRICUMANAL DEVICES, PERCUTANEOUS BIOLOGOPIC APPROACH Previous cardius procedure (CAGG, PTC, Stert) O2714G6 PX 10 DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALLIMINAL DEVICES, PERCUTANEOUS BIOLOGOPIC APPROACH Previous cardius procedure (CAGG, PTC, Stert) Previous cardius procedure (CAGG, PTC, Stert) O2714T8 PX 10 DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH FADIOACTIVE INTRALLIMINAL DEVICES, PERCUTANEOUS BIOLOGOPIC APPROACH Previous cardius procedure (CAGG, PTC, Stert) Previous cardius procedure (CAGG, PTC, Stert) O2714T8 PX 10 DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH PRODOACTIVE INTRALLIMINAL DEVICE, PERCUTANEOUS BIOLOGOPIC APPROACH DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH PRODOACTIVE INTRALLIMINAL DEVICE, PERCUTANEOUS BIOLOGOPIC APPROACH DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH PRODOACTIVE INTRALLIMINAL DEVICE, PERCUTANEOUS BIOLOGOPIC APPROACH DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH PRODOACTIVE INTRALLIMINAL DEVICE, PERCUTANEOUS BIOLOGOPIC APPROACH Previous cardius procedure (CAGG, PTC, Stert) O2714T7 PX 10 DIACTORIO CORROMAN PATERT, TWO ARTERIES, BIFURCATION, WITH PATE DATE PATER P | Previous cardiac procedure (CABG, PTCA, Stent) | 02714E6 | PX | 10 | · |
| Perious cardius procedure (CABC, PTCA, Stent) 0271472 PX 10 DILATION OF ARTERIES WITH TIMES INTRALLMINAL DEVICES, PERCUTANEOUS Provious cardius procedure (CABC, PTCA, Stent) 0271462 PX 10 DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALLMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALLMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH ADDIOACTIVE INTRALLMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH ADDIOACTIVE INTRALLMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH PRevious cardius procedure (CABC, PTCA, Sent) 0271462 PX 10 DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH ADDIOACTIVE INTRALLMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH PRevious cardius procedure (CABC, PTCA, Sent) 0271462 PX 10 DILATION OF CORROBAN ARTERY, TWO ARTERIES, BIFURCATION, WITH ADDIOACTIVE INTRALLMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH PRevious cardius procedure (CABC, PTCA, Sent) 0271462 PX 10 DILATION OF CORROBAN ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG ELUTING INTRALLMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH PRevious cardius procedure (CABC, PTCA, Sent) 0271462 PX 10 DILATION OF CORROBAN ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO DRUG ELUTING INTRALLMINAL DEVICE, OF EN APPROACH DILATION OF CORROBAN ARTE | Previous cardiac procedure (CABG, PTCA, Stent) | 02714EZ | PX | 10 | · |
| Previous cardiac procedure (CAG, PTCA, Stent) 0771466 PX | Previous cardiac procedure (CABG, PTCA, Stent) | 02714F6 | PX | 10 | |
| PERCIVAREOUS BRODGOOR/ APPROACH | Previous cardiac procedure (CABG, PTCA, Stent) | 02714FZ | PX | 10 | · |
| Frevious cardiac procedure (CA86, PTCA, Stent) 0271415 PX 10 DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, PRECUTANEOUS SHOOSCOPIC APPROACH Previous cardiac procedure (CA86, PTCA, Stent) 0271422 PX 10 DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, PRECUTANEOUS SHOOSCOPIC APPROACH Previous cardiac procedure (CA86, PTCA, Stent) 0271422 PX 10 DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, PRECUTANEOUS SHOOSCOPIC APPROACH Previous cardiac procedure (CA86, PTCA, Stent) 0272042 PX 10 DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, PRECUTANEOUS SHOOSCOPIC APPROACH DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO DRUG-CEPT APPROACH DIATION OF CORONANY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO DRUG-CEPT APPROACH DIATION OF CORONANY ARTERY, THERE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH DIATION OF CORONANY ARTERY, THERE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH DIATION OF CORONANY ARTERY, THERE ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH DIATION OF CORONANY ARTERY, THERE ARTERIES, BIFURCATION, WITH THRED DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH DIATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THRED DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DIATI | Previous cardiac procedure (CABG, PTCA, Stent) | 02714G6 | PX | 10 | |
| Previous cardiac procedure (CABC, PTCA, Stent) 0714172 PX 10 DILATION OF CORONARY ATTERY, TWO AFFERIES, BIFURCATION, PERCUTANEOUS EMOSCOPIC APPROACH Previous cardiac procedure (CABC, PTCA, Stent) 0714272 PX 10 DILATION OF CORONARY ATTERY, TWO AFFERIES, BIFURCATION, PERCUTANEOUS EMOSCOPIC APPROACH Previous cardiac procedure (CABC, PTCA, Stent) 0714272 PX 10 DILATION OF CORONARY ATTERY, TWO AFFERIES, BIFURCATION, PERCUTANEOUS EMOSCOPIC APPROACH DILATION OF CORONARY ATTERY, TWO AFFERIES, PERCUTANEOUS EMOSCOPIC APPROACH OPEN APPROACH PREVIOUS cardiac procedure (CABC, PTCA, Stent) 0714072 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERIES, PERCUTANEOUS EMOSCOPIC APPROACH OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERIES, BIFURCATION, WITH TWO DEUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERIES, BIFURCATION, WITH TWO DEUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERIES, BIFURCATION, WITH TWO DEUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ARTERIES, BIFURCATION, WITH THRE | | | | | ENDOSCOPIC APPROACH |
| Previous cardiac procedure (CABC, PTCA, Stent) 0271425 PX 10 OILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH Previous cardiac procedure (CABC, PTCA, Stent) 0272042 PX 10 OILATION OF CORONARY ARTERY, TWO ARTERIES, PERCUTANEOUS ENDOSCOPIC APPROACH Previous cardiac procedure (CABC, PTCA, Stent) 0272042 PX 10 OILATION OF CORONARY ARTERY, TWO ARTERIES, PERCUTANEOUS ENDOSCOPIC APPROACH OPEN APPROACH PRevious cardiac procedure (CABC, PTCA, Stent) 0272056 PX 10 OILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALLMINAL DEVICE, OPEN APPROACH DEVICES, OPEN APPROACH D | | | | | PERCUTANEOUS ENDOSCOPIC APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 2714-82 PX 10 DILATION OF CORONARY ATTERY, THECA ATTERICS, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH PREVIOUS cardiac procedure (CABG, PTCA, Stent) 272042 PX 10 DILATION OF CORONARY ATTERY, THECA ATTERISES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH PREVIOUS cardiac procedure (CABG, PTCA, Stent) 272056 PX 10 DILATION OF CORONARY ATTERY, THEE ATTERISES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH PREVIOUS cardiac procedure (CABG, PTCA, Stent) 272066 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH PREVIOUS cardiac procedure (CABG, PTCA, Stent) 272066 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERISES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ATTERY, THREE ATTERISES WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH PREVIOUS cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERISES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERISES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 0272075 PX 10 DILATION OF CORONARY ATTERY, THREE ATTERIS, BIFURCATION, WITH THREI INTRALUMINAL DEVICES, OPEN APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 0272075 PX 10 DIL | | | | | ENDOSCOPIC APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 272046 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALLMINAL DEVICE, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 272052 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES WITH TWO DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES WITH THREE DRUG-ELUTING INTRALLMINAL DEVICES, OPEN APPROACH DILATION OF CORONANY ARTERY, THREE ARTERIES WITH THREAL DILATION DEVICES, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 277205 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES WITH INTRALLMINAL DEVICE, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 277205 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALLMINAL DEVICES, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 277205 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THROU INTRALLMINAL DEVICES, OPEN | | | | | |
| Previous cardiac procedure (CABG, PTCA, Stent) 027204Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027205Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027205Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027206Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207C PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207C PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207C PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207C PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207C PX 10 DILATION OF CORDNARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FINGE INTRALUMINAL DEVICES, OPEN APPROACH Previou | • | | | | |
| Previous cardiac procedure (CABG, PTCA, Stent) 272056 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272066 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272062 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH HOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH HOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH HOW INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272076 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272077 PX 10 DILATION OF CORONANY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APP | | | | | OPEN APPROACH |
| DEWICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027205Z PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES WITH TWO DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027206Z PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALLUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALLUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX 10 DILATION DE CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027200E PX | | | | | APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 272066 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272067 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREI INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH | | | | | DEVICES, OPEN APPROACH |
| DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027206Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE DRIUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027207Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720DZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720DZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720DZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720DZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720DZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONA | | | | | APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 272076 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH HOUR OR MORE DRUG-ELUTING INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALLUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALLUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THOUR OR MORE INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALLUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALLUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIO | | | | | DEVICES, OPEN APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 0272072 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720D2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICE, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATIO | | | | | APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720D6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720E6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 P | , , , , , | | | | INTRALUMINAL DEVICES, OPEN APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720EZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720EZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH PREvious cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH PREvious cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH PREvious cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH PREvious cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVious cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH D | | | | | OPEN APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720E5 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVious cardiac procedure (CABG, PTCA, Stent) 0272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, | | | | | |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720EZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720G6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720GZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720TZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PROVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH | • | | | | |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720F6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720F2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720G6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720G2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 0272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PRevious cardiac procedure (CABG, PTCA, Stent) 0272342 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIous cardiac procedure (CABG, PTCA, Stent) 0272342 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAL PROCEDURE CABG, | | | | | APPROACH |
| APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720FZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720G6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720GZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720TG PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720TZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PROVIDED TO THE PROCEDURE (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH | | | | | · |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720G6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720G2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z7 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z2 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH D | | | | | APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720GZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720T6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720TZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZC PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, DEPN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH PREVIOUS CARDIAC PROCEDURE (CABG, PTCA, Stent) DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH | | | | | · |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720T6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720TZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZC PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | | | | | OPEN APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720TZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720Z6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | | | | | APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720Z6 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | , , , , , | | | | OPEN APPROACH |
| Previous cardiac procedure (CABG, PTCA, Stent) 02720ZZ PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, OPEN APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | | | | | |
| Previous cardiac procedure (CABG, PTCA, Stent) 272346 PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | | | | | , |
| PERCUTANEOUS APPROACH Previous cardiac procedure (CABG, PTCA, Stent) 027234Z PX 10 DILATION OF CORONARY ARTERY, THREE ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS | | | | | |
| | | | | | PERCUTANEOUS APPROACH |
| | Previous cardiac procedure (CABG, PTCA, Stent) | 027234Z | PX | 10 | |


| CHEMPAL PARKED NO LET THROUGH CEREBAN ATTENT CHEMPAL PARKED NO LET T | Ischemic stroke | 163.311 | DX | 10 | CEREBRAL INFARCTION DUE TO THROMBOSIS OF RIGHT MIDDLE CEREBRAL ARTERY |
|---|---|---|---|---|---|
| Inchamic cronice | | | | | |
| Inchemic stroke | | | | | |
| Inchemic stroke IS-3.32 | | | | | |
| Schemic stroke 16.3.321 | | | | | |
| Schemic Eroke 16.3.322 | | | | | |
| Inchemic stroke IS.3.232 | | | | | |
| Inchemic stroke 16.3.32 | | | | | |
| Inchemic stroke 16.3.33 | | | | | |
| Inchemic stroke 16.3.312 | | | | | |
| Ischemic stroke ISA-332 | | | | | |
| Inchemic stroke III | | | | | |
| Ischemic stroke ISA 339 | | | | | |
| Ischemic stroke 63.34 | | | | | |
| Inchemic stroke 16.3.412 DX | | | | | |
| Ischemic stroke | | | | | |
| Ischemic stroke ISS 3.43 | | | | | |
| Ischemic stroke ISA 3.49 DX | | | | | |
| Ischemic stroke 63.4 | | | | | |
| Ischemic stroke 163.4 | | | | | |
| Ischemic stroke ISA 40 | | | | | |
| Ischemic stroke ISA-41 | | | | | |
| Ischemic stroke | | | | | |
| Ischemic stroke 163.412 | | | | | |
| Ischemic stroke Ischanic strok | | | | | |
| Ischemic stroke 163.419 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED MIDDLE CEREBRAL ARTERY Ischemic stroke 163.421 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RATERIOR CEREBRAL ARTERY Ischemic stroke 163.422 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.423 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.429 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DISTRICING CEREBRAL ARTERY Ischemic stroke 163.432 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF PRICE CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILLYTERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBLAL ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBLAL ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBRAL ARTERY Ischemic stroke 163.540 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBRAL ARTERY Ischemic stroke 163.540 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBRAL ARTERY Ischemic stroke 163.551 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBRAL ARTERY Ischemic stroke 16 | | | | | |
| Ischemic stroke 163.42 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.421 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.422 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.423 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.430 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.432 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.439 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELEBRAL ARTERY Ischemic stroke 163.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DIASPECIFIED CEREBLAR ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DIASPECIFIED CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF STRONGS OF ELEBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED CELLISON OR STRONGS OF ELEBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIE | | | | | |
| Ischemic stroke 163.422 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF RIGHT ANTERIOR CERBRAL ARTERY Ischemic stroke 163.423 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF LEFT ANTERIOR CERBRAL ARTERY Ischemic stroke 163.429 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, ANTERIOR CERBRAL ARTERY Ischemic stroke 163.431 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, ANTERIOR CERBRAL ARTERY Ischemic stroke 163.431 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF DEMOSITION CERBRAL ARTERY Ischemic stroke 163.432 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF PROSTRION CERBRAL ARTERY Ischemic stroke 163.433 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CERBRAL ARTERY Ischemic stroke 163.433 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.439 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.441 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.442 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.443 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.443 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, POSTERIOR CERBRAL ARTERY Ischemic stroke 163.449 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA, CERBELLAR ARTERY Ischemic stroke 163.459 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA CERBELLAR ARTERY Ischemic stroke 163.50 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA CERBELLAR ARTERY Ischemic stroke 163.50 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA CERBELLAR ARTERY Ischemic stroke 163.51 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA CERBELLAR ARTERY Ischemic stroke 163.51 DX 10 CERBRAL INFARCTION DUE TO EMBOLISM OF BIATERIA CERBELLAR ARTERY Ischemic stroke 163.51 DX 10 CERBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF MIDDLE CERBRAL ARTERY Ischemic stroke 163.51 DX 10 CERBRAL INFARCTION | | | | | |
| Ischemic stroke ISA. 4.22 DX | | | | | |
| Ischemic stroke 163.423 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL ANTERIOR CEREBRAL ARTERIES Ischemic stroke 163.43 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.439 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELLAR ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELLAR ARTERY Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELLAR ARTERY Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELLAR ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELLAR ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELAR ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELAR ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIET CEREBELAR ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF MIDDLE CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR S | | | | | |
| Ischemic stroke ISA.43 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke ISA.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.432 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LET POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LETF POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.439 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBLAR ARTERY Ischemic stroke ISA.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBLAR ARTERY Ischemic stroke ISA.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ERBELLAR ARTERY Ischemic stroke ISA.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ELET CEREBLAR ARTERY Ischemic stroke ISA.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LIATERAL CEREBELLAR ARTERY Ischemic stroke ISA.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DILATERAL CEREBELLAR ARTERY Ischemic stroke ISA.459 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DILATERAL CEREBELLAR ARTERY Ischemic stroke ISA.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DILATERAL CEREBRAL ARTERY Ischemic stroke ISA.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DILATERAL CEREBRAL ARTERY Ischemic stroke ISA.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke ISA.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke ISA.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULISION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke ISA.521 DX 10 CEREBRAL | | | | | |
| Ischemic stroke ISA.43 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.431 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ROSH POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.432 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke ISA.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBRAL ARTERY Ischemic stroke ISA.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBLLAR ARTERY Ischemic stroke ISA.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBLAR ARTERY Ischemic stroke ISA.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERY Ischemic stroke ISA.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERY Ischemic stroke ISA.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBRAL ARTERY Ischemic stroke ISA.59 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBRAL ARTERY Ischemic stroke ISA.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULSION OR STROSIS OF LINGHED CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULSION OR STROSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke ISA.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULSION OR STROSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke ISA.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCULSION OR STROSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke ISA.522 DX 10 CEREBRAL IN | | | | | |
| Ischemic stroke Ischemic strok | | | | | |
| Ischemic stroke I63.432 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LEFT POSTERIOR CEREBRAL ARTERY Ischemic stroke I63.439 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERY Ischemic stroke I63.444 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED POSTERIOR CEREBRAL ARTERY Ischemic stroke I63.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBELLAR ARTERY Ischemic stroke I63.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBELLAR ARTERY Ischemic stroke I63.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBELLAR ARTERY Ischemic stroke I63.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERY Ischemic stroke I63.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DITAR CEREBRAL ARTERY Ischemic stroke I63.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke I63.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF INDECERBERAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HITERIOR CEREBRAL ARTERY Ischemic stroke I63.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR | | | | | |
| Ischemic stroke 163.433 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL POSTERIOR CEREBRAL ARTERIES Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED POSTERIOR CEREBRAL ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBELLAR ARTERY Ischemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ERITE ELERBELLAR ARTERY Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF ERITE ELERBELLAR ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERY Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERY Ischemic stroke 163.499 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF DILATERAL CEREBELLAR ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF CEREBRAL ARTERY Ischemic stroke 163.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF MIDDLE CEREBRAL ARTERY Ischemic stroke 163.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke 163.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF DILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF DILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF DILATERAL ARTERY Ischemic stroke 163.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OC | | | | | |
| Ischemic stroke I63.439 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED POSTERIOR CEREBRAL ARTERY Ischemic stroke I63.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBELLAR ARTERY Ischemic stroke I63.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF IGHT CEREBELLAR ARTERY Ischemic stroke I63.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF IGHT CEREBELLAR ARTERY Ischemic stroke I63.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF HIGH TERREBELLAR ARTERY Ischemic stroke I63.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF HIGH TERREBELLAR ARTERY Ischemic stroke I63.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF HIGH TERREBELLAR ARTERY Ischemic stroke I63.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke I63.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LORSPECIFIED CEREBRAL ARTERY Ischemic stroke I63.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH CEREBRAL ARTERY Ischemic stroke I63.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TIMIDALE CEREBRAL ARTERY Ischemic stroke I63.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TIMIDALE CEREBRAL ARTERY Ischemic stroke I63.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TIMIDALE CEREBRAL ARTERY Ischemic stroke I63.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TIMIDALE CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TIMIDALE CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TERREBIC ARTERY Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF HIGH TANTERIOR CEREBRAL ARTERY Ischemic stroke I63.522 DX 10 | | | | | |
| Ischemic stroke 163.44 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF CEREBELLAR ARTERY ISchemic stroke 163.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBELLAR ARTERY ISchemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBELLAR ARTERY ISchemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERIES ISchemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED CEREBELLAR ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OF UNSPECIFIED CEREBELLAR ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF INFERIOR CEREBRAL ARTERY ISCHEMIC STROKE 163.5 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF INFERIOR CEREBR | | | | | |
| Ischemic stroke I63.441 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF RIGHT CEREBELLAR ARTERY Ischemic stroke I63.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LEFT CEREBELLAR ARTERY Ischemic stroke I63.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LEFT CEREBELLAR ARTERY Ischemic stroke I63.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED CEREBELLAR ARTERY Ischemic stroke I63.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED CEREBELLAR ARTERY Ischemic stroke I63.50 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF OTHER CEREBRAL ARTERY Ischemic stroke I63.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF CEREBRAL ARTERY Ischemic stroke I63.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF MIDDLE CEREBRAL ARTERY Ischemic stroke I63.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF MIDDLE CEREBRAL ARTERY Ischemic stroke I63.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke I63.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke I63.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke I63.519 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF GRIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY ISCHEMIC | | | | | |
| Ischemic stroke 163.442 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF LEFT CEREBELLAR ARTERY Ischemic stroke 163.443 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF BILATERAL CEREBELLAR ARTERIES Ischemic stroke 163.449 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED CEREBBLLAR ARTERY Ischemic stroke 163.49 DX 10 CEREBRAL INFARCTION DUE TO EMBOLISM OF UNSPECIFIED CEREBRAL ARTERY Ischemic stroke 163.50 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF INSPECIFIED CEREBRAL ARTERY Ischemic stroke 163.51 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke 163.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke 163.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke 163.52 DX 10 CEREBRAL INFARCTION DUE | | | | | |
| Ischemic stroke Isshemic stroke Isshemic strok | | | | | |
| Ischemic stroke ISA.499 ISCHEMIC STROKE ISCHEMBAL INFARCTION D | | | | | |
| Ischemic stroke Ischemic s | Ischemic stroke | | | | |
| Ischemic stroke Ischemic strok | Ischemic stroke | | | | |
| Ischemic stroke Ischemic strok | Ischemic stroke | | | | |
| Ischemic stroke Ischemic strok | Ischemic stroke | | | | |
| Ischemic stroke IG3.511 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT MIDDLE CEREBRAL ARTERY Ischemic stroke IG3.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT MIDDLE CEREBRAL ARTERY Ischemic stroke IG3.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERIES Ischemic stroke IG3.519 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED MIDDLE CEREBRAL ARTERY Ischemic stroke IG3.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.529 DX 10 CEREBRAL INFARCTIO | Ischemic stroke | 163.50 | | | |
| Ischemic stroke IG3.512 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT MIDDLE CEREBRAL ARTERY Ischemic stroke IG3.513 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERIES Ischemic stroke IG3.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED MIDDLE CEREBRAL ARTERY Ischemic stroke IG3.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke IG3.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERY ISchemic stroke IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE IG3.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE IGAGE INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE IGAGE INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERY ISCHEMIC STROKE IGAGE IGAG | Ischemic stroke | | | | |
| Ischemic stroke Ischem | Ischemic stroke | 163.511 | | | |
| Ischemic stroke I63.519 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED MIDDLE CEREBRAL ARTERY Ischemic stroke I63.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERIES Ischemic stroke I63.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL ARTERIES | Ischemic stroke | 163.512 | DX | | CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT MIDDLE CEREBRAL ARTERY |
| ARTERY Ischemic stroke I63.52 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERIES Ischemic stroke I63.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL | Ischemic stroke | I63.513 | DX | 10 | CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL MIDDLE CEREBRAL ARTERIES |
| Ischemic stroke I63.521 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERIES Ischemic stroke I63.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL | Ischemic stroke | 163.519 | DX | 10 | |
| Ischemic stroke I63.522 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY Ischemic stroke I63.523 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF BILATERAL ANTERIOR CEREBRAL ARTERIES Ischemic stroke I63.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL | Ischemic stroke | 163.52 | DX | 10 | CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF ANTERIOR CEREBRAL ARTERY |
| Ischemic stroke Ischem | Ischemic stroke | 163.521 | DX | 10 | CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF RIGHT ANTERIOR CEREBRAL ARTERY |
| ARTERIES Ischemic stroke I63.529 DX 10 CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF UNSPECIFIED ANTERIOR CEREBRAL | Ischemic stroke | 163.522 | DX | 10 | CEREBRAL INFARCTION DUE TO UNSPECIFIED OCCLUSION OR STENOSIS OF LEFT ANTERIOR CEREBRAL ARTERY |
| | Ischemic stroke | 163.523 | DX | 10 | |
| | Ischemic stroke | 163.529 | DX | 10 | |


| Surgery PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular PVD diagnosis or surgery_peripheral vascular Surgery PVD diagnosis or surgery_peripheral vascular PVD diagnosis or surgery_peripheral vascular O41K0JJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO RIGHT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE, Surgery PVD diagnosis or surgery_peripheral vascular O41K0JJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE, Surgery | IAL TISSUE, OPEN TE, OPEN APPROACH E, OPEN APPROACH STITUTE, OPEN PEN APPROACH |
|---|---|
| PVD diagnosis or surgery_peripheral vascular 041K0AS PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY VEIN WITH AUTOLOGOUS ARTERI. APPROACH PVD diagnosis or surgery_peripheral vascular 041K0JH PX 10 BYPASS RIGHT FEMORAL ARTERY TO RIGHT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUT surgery PVD diagnosis or surgery_peripheral vascular 041K0JJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE, surgery | TE, OPEN APPROACH E, OPEN APPROACH SSTITUTE, OPEN PEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JH PX 10 BYPASS RIGHT FEMORAL ARTERY TO RIGHT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUT surgery PVD diagnosis or surgery_peripheral vascular 041K0JJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE, surgery | E, OPEN APPROACH SSTITUTE, OPEN PEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY WITH SYNTHETIC SUBSTITUTE, surgery | SSTITUTE, OPEN PEN APPROACH |
| | PEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JK PX 10 BYPASS RIGHT FEMORAL ARTERY TO BILATERAL FEMORAL ARTERIES WITH SYNTHETIC SUBS | |
| PVD diagnosis or surgery_peripheral vascular 041K0JL PX 10 BYPASS RIGHT FEMORAL ARTERY TO POPLITEAL ARTERY WITH SYNTHETIC SUBSTITUTE, OP surgery | EN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JM PX 10 BYPASS RIGHT FEMORAL ARTERY TO PERONEAL ARTERY WITH SYNTHETIC SUBSTITUTE, OPI surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0JN PX 10 BYPASS RIGHT FEMORAL ARTERY TO POSTERIOR TIBIAL ARTERY WITH SYNTHETIC SUBSTITUTION Surgery | UTE, OPEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JP PX 10 BYPASS RIGHT FEMORAL ARTERY TO FOOT ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN AP surgery | PPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JQ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY ARTERY WITH SYNTHETIC SUBSTIT surgery | ГUTE, OPEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0JS PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY VEIN WITH SYNTHETIC SUBSTITUT surgery | ΓΕ, OPEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0KH PX 10 BYPASS RIGHT FEMORAL ARTERY TO RIGHT FEMORAL ARTERY WITH NONAUTOLOGOUS TIS Surgery APPROACH | SSUE SUBSTITUTE, OPEN |
| PVD diagnosis or surgery_peripheral vascular 041K0KJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY WITH NONAUTOLOGOUS TISS surgery APPROACH | GUE SUBSTITUTE, OPEN |
| PVD diagnosis or surgery_peripheral vascular 041K0KK PX 10 BYPASS RIGHT FEMORAL ARTERYTO BILATERAL FEMORAL ARTERIES WITH NONAUTOLOGC OPEN APPROACH | OUS TISSUE SUBSTITUTE, |
| PVD diagnosis or surgery_peripheral vascular 041K0KL PX 10 BYPASS RIGHT FEMORAL ARTERY TO POPLITEAL ARTERY WITH NONAUTOLOGOUS TISSUE S APPROACH | SUBSTITUTE, OPEN |
| PVD diagnosis or surgery_peripheral vascular 041K0KM PX 10 BYPASS RIGHT FEMORAL ARTERY TO PERONEAL ARTERY WITH NONAUTOLOGOUS TISSUE S APPROACH | SUBSTITUTE, OPEN |
| PVD diagnosis or surgery_peripheral vascular 041K0KN PX 10 BYPASS RIGHT FEMORAL ARTERY TO POSTERIOR TIBIAL ARTERY WITH NONAUTOLOGOUS T<br>surgery OPEN APPROACH | TISSUE SUBSTITUTE, |
| PVD diagnosis or surgery_peripheral vascular 041K0KP PX 10 BYPASS RIGHT FEMORAL ARTERY TO FOOT ARTERY WITH NONAUTOLOGOUS TISSUE SUBST surgery | TITUTE, OPEN APPROACH |
| PVD diagnosis or surgery_peripheral vascular 041K0KQ PX 10 BYPASS RIGHT FEMORAL ARTERYTO LOWER EXTREMITY ARTERY WITH NONAUTOLOGOUS surgery OPEN APPROACH | TISSUE SUBSTITUTE, |
| PVD diagnosis or surgery_peripheral vascular 041K0KS PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY VEIN WITH NONAUTOLOGOUS TIS surgery APPROACH | SSUE SUBSTITUTE, OPEN |
| PVD diagnosis or surgery_peripheral vascular 041K0ZH PX 10 BYPASS RIGHT FEMORAL ARTERY TO RIGHT FEMORAL ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZJ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LEFT FEMORAL ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZK PX 10 BYPASS RIGHT FEMORAL ARTERY TO BILATERAL FEMORAL ARTERIES, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZL PX 10 BYPASS RIGHT FEMORAL ARTERY TO POPLITEAL ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZM PX 10 BYPASS RIGHT FEMORAL ARTERY TO PERONEAL ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZN PX 10 BYPASS RIGHT FEMORAL ARTERY TO POSTERIOR TIBIAL ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZP PX 10 BYPASS RIGHT FEMORAL ARTERY TO FOOT ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZQ PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY ARTERY, OPEN APPROACH surgery | |
| PVD diagnosis or surgery_peripheral vascular 041K0ZS PX 10 BYPASS RIGHT FEMORAL ARTERY TO LOWER EXTREMITY VEIN, OPEN APPROACH surgery | |


| NSAIDs | PHENYLEPHRINE RX<br>HCL/KETOROLAC<br>TROMETHAMINE | Generic |
|---|---|---|
| NCAID- | | Ci- |
| NSAIDs | PIROXICAM RX | Generic |
| NSAIDs | PIROXICAM/DIETA RX | Generic |
| | RY | |
| | SUPPLEMENT, MIS | |
| | C. CB.11 | |
| NSAIDs | ROFECOXIB RX | Generic |
| NSAIDs | ROPIVACAINE RX | Generic |
| | HCL/CLONIDINE | |
| | HCL/KETOROLAC | |
| | TROMETHAMINE | |
| NSAIDs | | Gonoria |
| NSAIDs | ROPIVACAINE RX | Generic |
| | HCL/EPINEPHRINE | |
| | /CLONIDINE | |
| | HCL/KETOROLAC | |
| | TROMETH | |
| NSAIDs | ROPIVACAINE/KET RX | Generic |
| NOMIO 3 | | Generic |
| | OROLAC/KETAMIN | |
| | E | |
| NSAIDs | SALICYLIC RX | Generic |
| | ACID/IBUPROFEN/ | |
| | CIMETIDINE | |
| NSAIDs | SALIVA RX | Generic |
| ואטעוקא | | Generic |
| | COLLECTION | |
| | DEVICE/IBUPROFE | |
| | N | |
| NSAIDs | SULINDAC RX | Generic |
| NSAIDs | SUMATRIPTAN RX | Generic |
| INDUIDS | | Generic |
| | SUCCINATE/NAPR | |
| | OXEN SODIUM | |
| NSAIDs | TOLMETIN RX | Generic |
| | SODIUM | |
| NSAIDs | TRAMADOL RX | Generic |
| | HCL/CELECOXIB | Generic |
| NCAID | | 6 |
| NSAIDs | TROPICAMIDE/PR RX | Generic |
| | OPARACAINE/PHE | |
| | NYLEPHRINE/KETO | |
| | ROLAC IN WATER | |
| NCAID- | VALDECOVID DV | C |
| NSAIDs | VALDECOXIB RX | Generic |
| Oral corticosteroids | BETAMETHASONE RX | Generic |
| Oral corticosteroids | CORTISONE RX | Generic |
| | ACETATE | |
| Oral corticosteroids | DEXAMETHASONE RX | Generic |
| Oral corticosteroids | DEXAMETHASONE RX | Generic |
| | ACETATE | |
| Oral corticosteroids | DEXAMETHASONE RX | Generic |
| | ISONICOTINATE | |
| Oral corticosteroids | DEXAMETHASONE RX | Generic |
| or ar cor ticosterorus | | Generic |
| | PHOSPHATE | |
| Oral corticosteroids | DEXAMETHASONE RX | Generic |
| | SODIUM | |
| | PHOSPHATE | |
| Oral corticosteroids | DEXAMETHASONE, RX | Generic |
| 5. 5. 501 (1003)(1010) | | Generic |
| Onel continue to the | MICRONIZED | |
| Oral corticosteroids | FLUDROCORTISON RX | Generic |
| | E ACETATE | |

| Oral corticosteroids | HYDROCORTISONE R | х | Generic | Oral |
|---|---|---|---|---|
| Oral corticosteroids | HYDROCORTISONE RY | x | Generic | Oral |
| Oral corticosteroids | HYDROCORTISONE RY | x | Generic | Oral |
| Oral corticosteroids | HYDROCORTISONE RY | х | Generic | Oral |
| Oral corticosteroids | HYDROCORTISONE RY | x | Generic | Oral |
| Oral corticosteroids | HYDROCORTISONE RY<br>SOD PHOSPHATE | x | Generic | Oral |
| Oral corticosteroids | HYDROCORTISONE RY | x | Generic | Oral |
| Oral corticosteroids | METHYLPREDNISO RX | x | Generic | Oral |
| Oral corticosteroids | METHYLPREDNISO RX<br>LONE ACETATE | x | Generic | Oral |
| Oral corticosteroids | METHYLPREDNISO RY<br>LONE ACETATE,<br>MICRONIZED | X | Generic | Oral |
| Oral corticosteroids | METHYLPREDNISO RY<br>LONE SODIUM<br>SUCCINATE | x | Generic | Oral |
| Oral corticosteroids | METHYLPREDNISO RY<br>LONE,<br>MICRONIZED | X | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RX | X | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RX | x | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RY<br>ACETATE,<br>MICRONIZED | X | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RX<br>ACETATE/BROMFE<br>NAC SODIUM | x | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RX<br>SODIUM<br>PHOSPHATE | x | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE RY<br>SODIUM<br>PHOSPHATE/BRO<br>MFENAC SODIUM | X | Generic | Oral |
| Oral corticosteroids | PREDNISOLONE, RX | x | Generic | Oral |
| Oral corticosteroids | PREDNISONE RX | X | Generic | Oral |
| Oral corticosteroids | PREDNISONE RX<br>MICRONIZED | X | Generic | Oral |
| Oral corticosteroids | TRIAMCINOLONE RX | X | Generic | Oral |
| Biphosphonates | ALENDRONATE RX<br>SODIUM | x | Generic | |
| Biphosphonates | ALENDRONATE R) SODIUM/CHOLEC ALCIFEROL (VITAMIN D3) | x | Generic | |
| Biphosphonates | RISEDRONATE R | x | Generic | |

SODIUM


| Endocrinologist visit | 1959 | Provider category code |
|-----------------------|------------|---------------------------|
| Endocrinologist visit | 2860 | Provider category code |
| Endocrinologist visit | 3589 | Provider category |
| Endocrinologist visit | 5775 | code<br>Provider category |
| Endocrinologist visit | 5853 | code<br>Provider category |
| Endocrinologist visit | 207RE0101X | code<br>NUCC Taxonomy |
| Endocrinologist visit | 207RE0101X | Code 1<br>NUCC Taxonomy |
| Cardiologist visit | 0400 | Code 2 Provider category |
| Cardiologist visit | 0401 | code Provider category |
| | 0402 | code |
| Cardiologist visit | | Provider category code |
| Cardiologist visit | 0403 | Provider category code |
| Cardiologist visit | 0404 | Provider category code |
| Cardiologist visit | 0405 | Provider category code |
| Cardiologist visit | 0407 | Provider category code |
| Cardiologist visit | 0408 | Provider category code |
| Cardiologist visit | 0409 | Provider category |
| Cardiologist visit | 0410 | code<br>Provider category |
| Cardiologist visit | 0411 | code<br>Provider category |
| Cardiologist visit | 0412 | code<br>Provider category |
| Cardiologist visit | 0416 | code<br>Provider category |
| Cardiologist visit | 1108 | code Provider category |
| - | 1123 | code |
| Cardiologist visit | | Provider category<br>code |
| Cardiologist visit | 1135 | Provider category code |
| Cardiologist visit | 1162 | Provider category code |
| Cardiologist visit | 1212 | Provider category code |
| Cardiologist visit | 1582 | Provider category code |
| Cardiologist visit | 1629 | Provider category code |
| Cardiologist visit | 1728 | Provider category code |
| Cardiologist visit | 1856 | Provider category |
| Cardiologist visit | 1947 | code<br>Provider category |
| | | code |

| Cardiologist visit | 2653 | Provider category code |
|---|---|---|
| Cardiologist visit | 2810 | Provider category code |
| Cardiologist visit | 3073 | Provider category code |
| Cardiologist visit | 3137 | Provider category code |
| Cardiologist visit | 3249 | Provider category code |
| Cardiologist visit | 3534 | Provider category code |
| Cardiologist visit | 4113 | Provider category code |
| Cardiologist visit | 4163 | Provider category code |
| Cardiologist visit | 4622 | Provider category code |
| Cardiologist visit | 4644 | Provider category code |
| Cardiologist visit | 5726 | Provider category code |
| Cardiologist visit | 5742 | Provider category code |
| Cardiologist visit | 5761 | Provider category code |
| Cardiologist visit | 5771 | Provider category code |
| Cardiologist visit | 6593 | Provider category code |
| Cardiologist visit | 6616 | Provider category code |
| Cardiologist visit | 6887 | Provider category code |
| Cardiologist visit | 7034 | Provider category code |
| Cardiologist visit | 7749 | Provider category code |
| Cardiologist visit | 207RC0000X | NUCC Taxonomy<br>Code 1 |
| Cardiologist visit | 207RC0000X | NUCC Taxonomy<br>Code 2 |
| Internal medicine/family medicine visit | 0334 | Provider category code |
| Internal medicine/family medicine visit | 0335 | Provider category code |
| Internal medicine/family medicine visit | 0336 | Provider category code |
| Internal medicine/family medicine visit | 0337 | Provider category code |
| Internal medicine/family medicine visit | 0338 | Provider category code |
| Internal medicine/family medicine visit | 0339 | Provider category code |
| Internal medicine/family medicine visit | 0340 | Provider category code |
| Internal medicine/family medicine visit | 0341 | Provider category code |
| Internal medicine/family medicine visit | 0342 | Provider category code |

| Internal medicine/family medicine visit | 1133 | Provider category code |
|-----------------------------------------|------|------------------------|
| Internal medicine/family medicine visit | 1419 | Provider category code |
| Internal medicine/family medicine visit | 1673 | Provider category code |
| Internal medicine/family medicine visit | 1697 | Provider category code |
| Internal medicine/family medicine visit | 1860 | Provider category code |
| Internal medicine/family medicine visit | 1864 | Provider category code |
| Internal medicine/family medicine visit | 2050 | Provider category code |
| Internal medicine/family medicine visit | 2280 | Provider category code |
| Internal medicine/family medicine visit | 2302 | Provider category code |
| Internal medicine/family medicine visit | 2313 | Provider category code |
| Internal medicine/family medicine visit | 2314 | Provider category code |
| Internal medicine/family medicine visit | 2373 | Provider category code |
| Internal medicine/family medicine visit | 2610 | Provider category code |
| Internal medicine/family medicine visit | 2842 | Provider category code |
| Internal medicine/family medicine visit | 3268 | Provider category code |
| Internal medicine/family medicine visit | 3755 | Provider category code |
| Internal medicine/family medicine visit | 4641 | Provider category code |
| Internal medicine/family medicine visit | 4876 | Provider category code |
| Internal medicine/family medicine visit | 5724 | Provider category code |
| Internal medicine/family medicine visit | 5736 | Provider category code |
| Internal medicine/family medicine visit | 5829 | Provider category code |
| Internal medicine/family medicine visit | 5991 | Provider category code |
| Internal medicine/family medicine visit | 5998 | Provider category code |
| Internal medicine/family medicine visit | 0308 | Provider category code |
| Internal medicine/family medicine visit | 0311 | Provider category code |
| Internal medicine/family medicine visit | 0312 | Provider category code |
| Internal medicine/family medicine visit | 0313 | Provider category code |
| Internal medicine/family medicine visit | 0314 | Provider category code |
| Internal medicine/family medicine visit | 0316 | Provider category code |
| Internal medicine/family medicine visit | 0317 | Provider category code |

| Internal medicine/family medicine visit | 0318 | Provider category code |
|---|---|---|
| Internal medicine/family medicine visit | 0319 | Provider category code |
| Internal medicine/family medicine visit | 0326 | Provider category code |
| Internal medicine/family medicine visit | 0327 | Provider category |
| Internal medicine/family medicine visit | 0329 | code<br>Provider category |
| Internal medicine/family medicine visit | 0330 | code<br>Provider category |
| Internal medicine/family medicine visit | 0331 | code<br>Provider category |
| Internal medicine/family medicine visit | 0332 | code<br>Provider category<br>code |
| Internal medicine/family medicine visit | 0333 | Provider category |
| Internal medicine/family medicine visit | 1046 | code<br>Provider category |
| Internal medicine/family medicine visit | 1113 | code<br>Provider category |
| Internal medicine/family medicine visit | 1127 | code<br>Provider category |
| Internal medicine/family medicine visit | 1643 | code<br>Provider category |
| Internal medicine/family medicine visit | 1646 | code<br>Provider category |
| Internal medicine/family medicine visit | 1694 | code<br>Provider category |
| Internal medicine/family medicine visit | 1721 | code<br>Provider category |
| Internal medicine/family medicine visit | 1785 | code<br>Provider category |
| Internal medicine/family medicine visit | 1832 | code<br>Provider category |
| Internal medicine/family medicine visit | 1865 | code<br>Provider category |
| Internal medicine/family medicine visit | 1927 | code<br>Provider category |
| Internal medicine/family medicine visit | 2068 | code<br>Provider category |
| Internal medicine/family medicine visit | 2189 | code<br>Provider category |
| Internal medicine/family medicine visit | 2219 | code<br>Provider category |
| Internal medicine/family medicine visit | 2233 | code<br>Provider category |
| | 2286 | code Provider category |
| Internal medicine/family medicine visit | | code |
| Internal medicine/family medicine visit | 2340 | Provider category code |
| Internal medicine/family medicine visit | 2354 | Provider category code |
| Internal medicine/family medicine visit | 2378 | Provider category code |
| Internal medicine/family medicine visit | 2403 | Provider category code |
| Internal medicine/family medicine visit | 2574 | Provider category code |

| Internal medicine/family medicine visit | 2614 | Provider category code |
|---|---|---|
| Internal medicine/family medicine visit | 2615 | Provider category code |
| Internal medicine/family medicine visit | 2628 | Provider category code |
| Internal medicine/family medicine visit | 2644 | Provider category code |
| Internal medicine/family medicine visit | 2790 | Provider category code |
| Internal medicine/family medicine visit | 2835 | Provider category code |
| Internal medicine/family medicine visit | 2978 | Provider category code |
| Internal medicine/family medicine visit | 2996 | Provider category code |
| Internal medicine/family medicine visit | 3122 | Provider category code |
| Internal medicine/family medicine visit | 3777 | Provider category code |
| Internal medicine/family medicine visit | 3787 | Provider category code |
| Internal medicine/family medicine visit | 4362 | Provider category code |
| Internal medicine/family medicine visit | 4645 | Provider category code |
| Internal medicine/family medicine visit | 4648 | Provider category code |
| Internal medicine/family medicine visit | 5063 | Provider category code |
| Internal medicine/family medicine visit | 5683 | Provider category code |
| Internal medicine/family medicine visit | 5696 | Provider category code |
| Internal medicine/family medicine visit | 5706 | Provider category code |
| Internal medicine/family medicine visit | 5732 | Provider category code |
| Internal medicine/family medicine visit | 5774 | Provider category code |
| Internal medicine/family medicine visit | 5781 | Provider category code |
| Internal medicine/family medicine visit | 5994 | Provider category code |
| Internal medicine/family medicine visit | 6000 | Provider category code |
| Internal medicine/family medicine visit | 7017 | Provider category code |
| Internal medicine/family medicine visit | 7592 | Provider category code |
| Internal medicine/family medicine visit | 7777 | Provider category code |
| Internal medicine/family medicine visit | 7792 | Provider category code |
| Internal medicine/family medicine visit | 207Q00000X | NUCC Taxonomy<br>Code 1 |
| Internal medicine/family medicine visit | 207QA0000X | NUCC Taxonomy<br>Code 1 |
| Internal medicine/family medicine visit | 207QA0401X | NUCC Taxonomy<br>Code 1 |

